CLINICAL TRIAL: NCT02564042
Title: Study 203120: A Randomized, Blinded, Vehicle-Controlled, Dose-Finding Study of GSK2894512 Cream for the Treatment of Plaque Psoriasis
Brief Title: A Dose-Finding Study of GSK2894512 Cream in Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 203120
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Psoriasis
Keywords: Double blind; Dose-finding; Vehicle-Controlled; GSK2894512; Plaque Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — tapinarof

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- GSK2894512 1% cream twice daily (Experimental): Subjects will apply a thin layer of GSK2894512 1% (10 milligram per gram [mg/g]) topical cream twice daily (morning and evening) for 12 weeks, to all psoriasis lesions (except on the scalp).
  Interventions: Drug: GSK2894512 1% Cream
- GSK2894512 1% cream once daily (Experimental): Subjects will apply a thin layer of GSK2894512 1% (10 mg/g) topical cream once daily (evening) for 12 weeks, to all psoriasis lesions (except on the scalp).
  Interventions: Drug: GSK2894512 1% Cream
- GSK2894512 0.5% cream twice daily (Experimental): Subjects will apply a thin layer of GSK2894512 0.5% (5 mg/g) topical cream twice daily (morning and evening) for 12 weeks, to all psoriasis lesions (except on the scalp).
  Interventions: Drug: GSK2894512 0.5% Cream
- GSK2894512 0.5% cream once daily (Experimental): Subjects will apply a thin layer of GSK2894512 0.5% (5 mg/g) topical cream once daily (evening) for 12 weeks, to all psoriasis lesions (except on the scalp).
  Interventions: Drug: GSK2894512 0.5% Cream
- Vehicle cream twice daily (Placebo Comparator): Subjects will apply a thin layer of vehicle topical cream twice daily (morning and evening) for 12 weeks, to all psoriasis lesions (except on the scalp).
  Interventions: Drug: Vehicle cream
- Vehicle cream once daily (Placebo Comparator): Subjects will apply a thin layer of vehicle topical cream once daily (evening) for 12 weeks, to all psoriasis lesions (except on the scalp).
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: GSK2894512 1% Cream — 1.0% (10 mg/g) GSK2894512 will be supplied as white to off-white cream to be applied topically
  Arms: GSK2894512 1% cream once daily; GSK2894512 1% cream twice daily
Drug: GSK2894512 0.5% Cream — 0.5% (5 mg/g) GSK2894512 will be supplied as white to off-white cream to be applied topically
  Arms: GSK2894512 0.5% cream once daily; GSK2894512 0.5% cream twice daily
Drug: Vehicle cream — White to off-white vehicle cream base to be applied topically
  Arms: Vehicle cream once daily; Vehicle cream twice daily

SUMMARY:
This study will evaluate the efficacy and safety of two concentrations (0.5 percent [%] and 1%) and two application frequencies (once a day and twice a day) of GSK2894512 cream for the topical treatment in subjects with plaque psoriasis. Results from this study will be considered when selecting the most appropriate concentration of GSK2894512 cream and dosing frequency in future clinical safety and efficacy studies. This is a multicenter (United States, Canada, and Japan), randomized, double-blind (sponsor-unblind), vehicle-controlled, 6-arm, parallel-group, dose-finding study. Two concentrations of GSK2894512 cream (0.5% and 1%) and a vehicle control cream will be equally randomized and evaluated following application to all psoriasis lesions (except on the scalp) once daily (evening) or twice daily (morning and evening) for 12 weeks. This study will consist of 3 periods: up to 4 weeks screening, 12 weeks double-blind treatment, and 4 weeks post-treatment follow-up. The total duration of subject participation will be approximately 16 to 20 weeks. Approximately 270 adult males and females subjects with plaque psoriasis will be screened in order to have at least 228 randomized subjects (38 subjects for each of the 6 treatment groups) and approximately 204 evaluable subjects overall. Approximately 30 subjects will be randomized in Japan to achieve at least 24 evaluable Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Confirmed clinical diagnosis of chronic stable plaque psoriasis for >=6 months.
* Body surface area involvement >=1% and <=15%, excluding scalp, at Screening and Baseline.
* A PGA of psoriasis score >=2 at Baseline.
* One target plaque located on the trunk or proximal parts of extremities (excluding knees, elbows, and intertriginous areas) that is at least 3 (centimetre) cm х 3 cm in size at Screening and Baseline with a severity representative of the subject's overall disease.
* A female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin test), not lactating, and at least one of the following conditions applies: Non-reproductive potential defined as: 1) Pre-menopausal females with one of the following procedures documented: tubal ligation; hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; hysterectomy; bilateral oophorectomy. 2) Post-menopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone and estradiol levels consistent with menopause and falling into the central laboratory's postmenopausal reference range is confirmatory). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt are required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment; Reproductive potential and agrees to follow one of the options listed in the modified list of highly effective methods for avoiding pregnancy in females of reproductive potential from 30 days prior to the first dose of study medication and until (at least five terminal half-lives OR until any continuing pharmacologic effect has ended, whichever is longer) after the last dose of study medication and completion of the follow-up visit.

Exclusion Criteria:

* Any sign of infection of any of the psoriatic lesions.
* A history or ongoing serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, may interfere with the subject's completion of the study.
* Known hypersensitivity to the study treatment excipients, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates participation.
* Current or chronic history of liver disease, known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones), presence of hepatitis B surface antigen, or positive hepatitis C antibody test result within 3 months of screening.
* Liver function tests: alanine aminotransferase >=2x upper limit of normal (ULN); alkaline phosphatase and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* QTc >=450 milliseconds (msec) or QTc >=480 msec for subjects with bundle branch block.

NOTES: The QTc is the QT interval corrected for heart rate according to Fridericia's formula (QTcF), with machine over-read. The QTc should be based on a single ECG obtained over a brief recording period. If QTc is outside of the threshold value, triplicate ECGs may be performed with the QTc values averaged.

* Ultraviolet (UV) light therapy or prolonged exposure to natural or artificial sources of UV radiation (eg, sunlight or tanning booth) within 4 weeks prior to the baseline visit and/or intention to have such exposure during the study, which is thought by the investigator to potentially impact the subject's psoriasis.
* Used any of the following treatments within the indicated washout period before the baseline visit: 1) 12 weeks or 5 half-lives (whichever is longer) - biologic agents (eg, 24 weeks for alefacept, 12 weeks for etanercept, 15 weeks for ustekinumab); 2) 12 weeks - oral retinoids (eg, acitretin or isotretinoin); 3) 8 weeks - cyclosporin, interferon, methotrexate, other systemic immunosuppressive or immunomodulating agents, or psoralen plus UVA light treatment; 4) 4 weeks - systemic corticosteroids or adrenocorticotropic hormone analogs; 5) 2 weeks - immunizations; drugs known to possibly worsen psoriasis, such as beta-blockers (eg, propranolol), lithium, iodides, angiotensin-converting enzyme inhibitors, and indomethacin, unless on a stable dose for >12 weeks; 6) 2 weeks - topical treatments: corticosteroids, immunomodulators, anthralin (dithranol), Vitamin D derivatives, retinoids, or coal tar (used on the body).
* Participated in a clinical study and received an investigational product within the following time period prior to the baseline visit: 4 weeks, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of alcohol or other substance abuse within the last 2 years.
* Participated in a previous study using GSK2894512 (or WBI-1001).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2015-11-23; Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (36):
- United States (18):
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, North Logan, Connecticut
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Plainfield, Indiana
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Fort Gratiot Township, Michigan
  - GSK Investigational Site, High Point, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Johnston, Rhode Island
  - GSK Investigational Site, Goodlettsville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Webster, Texas
  - GSK Investigational Site, Seattle, Washington
- Canada (12):
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Markham, Ontario
  - GSK Investigational Site, North Bay, Ontario
  - GSK Investigational Site, Oakville, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Peterborough, Ontario
  - GSK Investigational Site, Richmond Hill, Ontario
  - GSK Investigational Site, Waterloo, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- Japan (6):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind, dose-finding study of GSK2894512 in adult participants with psoriasis. The study consisted of 3 periods: 4 weeks screening, 12 weeks double-blind treatment, and 4 weeks post-treatment follow-up. The total duration of study for a participant was 16-20 weeks.
Pre-assignment Details: A total of 290 participants were screened of which 63 failed screening and 227 participants were randomized into the study. Participants in the treatment phase were randomized to receive GSK2894512 cream (0.5 or 1 percent) or vehicle control once daily (QD) or twice daily (BID).
Groups:
- GSK2894512 1% BID: The participants were topically administered GSK2894512 1% (10 milligrams per gram [mg/g]) cream applied BID approximately 12 hours apart at the same time each day for 12 weeks. The cream was applied as a thin layer to all psoriasis lesions except on the scalp.
- GSK2894512 1% QD: The participants were topically administered GSK2894512 1% (10 mg/g) cream applied QD approximately the same time each day for 12 weeks. The cream was applied as a thin layer to all psoriasis lesions except on the scalp.
- GSK2894512 0.5% BID: The participants were topically administered GSK2894512 0.5% (5 mg/g) cream applied BID approximately 12 hours apart at the same time each day for 12 weeks. The cream was applied as a thin layer to all psoriasis lesions except on the scalp.
- GSK2894512 0.5% QD: The participants were topically administered GSK2894512 0.5% (5 mg/g) cream applied QD approximately the same time each day for 12 weeks. The cream was applied as a thin layer to all psoriasis lesions except on the scalp.
- Vehicle BID: The participants were topically administered vehicle applied BID approximately 12 hours apart at the same time each day for 12 weeks. The cream was applied as a thin layer to all psoriasis lesions except on the scalp.
- Vehicle QD: The participants were topically administered vehicle applied QD approximately at the same time each day for 12 weeks. The cream was applied as a thin layer to all psoriasis lesions except on the scalp.
Period: Overall Study
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Started | 38 | 38 | 38 | 38 | 37 | 38
Completed | 27 | 30 | 32 | 35 | 26 | 24
Not Completed | 11 | 8 | 6 | 3 | 11 | 14
Not completed — Adverse Event | 4 | 4 | 3 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 3 | 2 | 2 | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD | Total
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38 | 227
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.9 (11.93) | 48.5 (10.56) | 49.6 (10.93) | 48.7 (9.72) | 46.7 (12.62) | 46.4 (10.16) | 47.6 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 14 | 13 | 14 | 9 | 74
  Male | 26 | 26 | 24 | 25 | 23 | 29 | 153
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race, Customized: American Indian (Amer Ind)/Alaska Native (Ala Nat) | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Race, Customized: Asian/South East Asian Descent/Japanese Descent | 10 | 9 | 8 | 6 | 9 | 6 | 48
  Race, Customized: Black/African American (Afr Amer) | 1 | 2 | 3 | 1 | 3 | 0 | 10
  Race, Customized: White/Caucasian | 26 | 27 | 26 | 30 | 25 | 32 | 166
  Race, Customized: Amer Ind/Ala Nat & Black/Afr Amer &White/Caucasian | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Race, Customized: Black/Afr Amer & White/Caucasian | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Have a Physician Global Assessment (PGA) Score of 0 or 1 at Week 12 and a Minimum 2-grade Improvement in PGA Score From Baseline to Week 12
Description: The PGA is a clinical tool for assessing the current state/severity of a participant's psoriasis. It is a static 5-point morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema, plaque thickness, and scaling as guidelines. Each assessment was made as a visual 'average' of the severity of all treated areas at the time of the assessment. The scores ranged from 0 to 4 where 0 = Clear, 1 = Almost Clear, 2 = Mild, 3 = Moderate and 4=Severe. The percentage of responders that is, participants who achieved a PGA score of 0 or 1 and a minimum 2-grade improvement from Baseline were summarized. Baseline was defined as the latest assessment prior to the first dose. The analysis was performed on modified intent-to-treat (mITT) Population which comprised of all randomized participants except those enrolled at center ID 220008.
Time Frame: Baseline and up to Week 12
Population: mITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 23 | 25 | 26 | 28 | 19 | 20
Percentage of participants | 65 | 56 | 46 | 36 | 11 | 5
Statistical Analysis 1: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Proportion difference = 54.7, 95% CI 2-sided [25.9 to 76.6] — Difference between GSK2894512 1% BID and Vehicle BID has been presented
Statistical Analysis 2: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Proportion difference = 51.0, 95% CI 2-sided [22.2 to 73.2] — Difference between GSK2894512 1% QD and Vehicle QD has been presented
Statistical Analysis 3: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Proportion difference = 35.6, 95% CI 2-sided [6.3 to 60.5] — Difference between GSK2894512 0.5% BID and Vehicle BID has been presented
Statistical Analysis 4: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Proportion difference = 30.7, 95% CI 2-sided [1.6 to 55.9] — Difference between GSK2894512 0.5% QD and Vehicle QD has been presented

2. Secondary Outcome: Percentage of Participants With >=75 Percent Improvement in Psoriasis Area and Severity Index (PASI) From Baseline to Each Study Visit
Description: The PASI is a standard clinical tool for assessing the severity of psoriasis based on severity of erythema, thickness and scale, as well as the extent of body surface area (BSA) affected with psoriasis. The 3 clinical signs were graded on a 5 point scale (0 to 4) and the % BSA affected was scored on a 7-point scale (0 to 6) for each of the 4 specified body regions (head, upper extremities, trunk and lower extremities). The individual scores were multiplied by a weighted factor for each body region. The sum of these scores gave the overall PASI score. Higher scores indicated more severe disease. The percentage of participants with >=75% improvement in PASI from Baseline were summarized. Baseline was defined as the latest assessment prior to the first dose. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 16
Population: mITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 34 | 35 | 32 | 32 | 30 | 33
Percentage of participants
  Week 1, n=32, 35, 31, 32, 28, 32: number analyzed (Participants) | 32 | 35 | 31 | 32 | 28 | 32
  Week 1, n=32, 35, 31, 32, 28, 32 | 0 | 3 | 0 | 0 | 0 | 0
  Week 2, n=32, 33, 30, 32, 24, 30: number analyzed (Participants) | 32 | 33 | 30 | 32 | 24 | 30
  Week 2, n=32, 33, 30, 32, 24, 30 | 6 | 15 | 3 | 3 | 0 | 0
  Week 4, n=28, 31, 29, 32, 22, 26: number analyzed (Participants) | 28 | 31 | 29 | 32 | 22 | 26
  Week 4, n=28, 31, 29, 32, 22, 26 | 32 | 26 | 14 | 6 | 5 | 0
  Week 8, n=26, 27, 27, 32, 20, 20: number analyzed (Participants) | 26 | 27 | 27 | 32 | 20 | 20
  Week 8, n=26, 27, 27, 32, 20, 20 | 50 | 37 | 37 | 34 | 5 | 0
  Week 12, n=23, 25, 26, 28, 19, 20: number analyzed (Participants) | 23 | 25 | 26 | 28 | 19 | 20
  Week 12, n=23, 25, 26, 28, 19, 20 | 65 | 56 | 46 | 46 | 16 | 5
  Week 14, n=23, 26, 24, 27, 19, 19: number analyzed (Participants) | 23 | 26 | 24 | 27 | 19 | 19
  Week 14, n=23, 26, 24, 27, 19, 19 | 65 | 65 | 46 | 48 | 16 | 5
  Week 16, n=24, 26, 26, 28, 19, 19: number analyzed (Participants) | 24 | 26 | 26 | 28 | 19 | 19
  Week 16, n=24, 26, 26, 28, 19, 19 | 63 | 58 | 46 | 54 | 11 | 5
  Early withdrawal (EW), n=10, 7, 4, 2, 10, 9: number analyzed (Participants) | 10 | 7 | 4 | 2 | 10 | 9
  Early withdrawal (EW), n=10, 7, 4, 2, 10, 9 | 10 | 43 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Proportion difference = 2.9, 95% CI 2-sided [-21.0 to 26.6] — Difference between GSK2894512 1% QD and Vehicle QD at Week 1 has been presented
Statistical Analysis 2: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Proportion difference = 6.3, 95% CI [-20.5 to 32.4] — Difference between GSK2894512 1% BID and Vehicle BID at Week 2 has been presented
Statistical Analysis 3: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Proportion difference = 15.2, 95% CI 2-sided [-9.6 to 39.1] — Difference between GSK2894512 1% QD and Vehicle QD at Week 2 has been presented
Statistical Analysis 4: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Proportion difference = 3.3, 95% CI 2-sided [-23.6 to 29.9] — Difference between GSK2894512 0.5% BID and Vehicle BID at Week 2 has been presented
Statistical Analysis 5: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Proportion difference = 3.1, 95% CI 2-sided [-22.2 to 28.1] — Difference between GSK2894512 0.5% QD and Vehicle QD at Week 2 has been presented
Statistical Analysis 6: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Proportion difference = 27.6, 95% CI 2-sided [-0.5 to 52.4] — Difference between GSK2894512 1% BID and Vehicle BID at Week 4 has been presented
Statistical Analysis 7: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Proportion difference = 25.8, 95% CI 2-sided [-0.4 to 49.3] — Difference between GSK2894512 1% QD and Vehicle QD at Week 4 has been presented
Statistical Analysis 8: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Proportion difference = 9.2, 95% CI 2-sided [-18.4 to 35.7] — Difference between GSK2894512 0.5% BID and Vehicle BID at Week 4 has been presented
Statistical Analysis 9: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Proportion difference = 6.3, 95% CI 2-sided [-19.7 to 31.7] — Difference between GSK2894512 0.5% QD and Vehicle QD at Week 4 has been presented
Statistical Analysis 10: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Proportion difference = 45.0, 95% CI 2-sided [16.6 to 68.4] — Difference between GSK2894512 1% BID and Vehicle BID at Week 8 has been presented
Statistical Analysis 11: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Proportion difference = 37.0, 95% CI 2-sided [8.7 to 61.3] — Difference between GSK2894512 1% QD and Vehicle QD at Week 8 has been presented
Statistical Analysis 12: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Proportion difference = 32.0, 95% CI 2-sided [3.5 to 57.2] — Difference between GSK2894512 0.5% BID and Vehicle BID at Week 8 has been presented
Statistical Analysis 13: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Proportion difference = 34.4, 95% CI 2-sided [6.3 to 58.7] — Difference between GSK2894512 0.5% QD and Vehicle QD at Week 8 has been presented
Statistical Analysis 14: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Proportion difference = 49.4, 95% CI 2-sided [20.1 to 72.4] — Difference between GSK2894512 1% BID and Vehicle BID at Week 12 has been presented
Statistical Analysis 15: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Proportion difference = 51.0, 95% CI 2-sided [22.2 to 73.2] — Difference between GSK2894512 1% QD and Vehicle QD at Week 12 has been presented
Statistical Analysis 16: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Proportion difference = 30.4, 95% CI 2-sided [1.0 to 56.1] — Difference between GSK2894512 0.5% BID and Vehicle BID at Week 12 has been presented
Statistical Analysis 17: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Proportion difference = 41.4, 95% CI 2-sided [12.7 to 65.0] — Difference between GSK2894512 0.5% QD and Vehicle QD at Week 12 has been presented
Statistical Analysis 18: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Proportion difference = 49.4, 95% CI 2-sided [20.1 to 72.4] — Difference between GSK2894512 1% BID and Vehicle BID at Week 14 has been presented
Statistical Analysis 19: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Proportion difference = 60.1, 95% CI 2-sided [33.2 to 80.1] — Difference between GSK2894512 1% QD and Vehicle QD at Week 14 has been presented
Statistical Analysis 20: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Proportion difference = 30.0, 95% CI 2-sided [0.2 to 56.5] — Difference between GSK2894512 0.5% BID and Vehicle BID at Week 14 has been presented
Statistical Analysis 21: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Proportion difference = 42.9, 95% CI 2-sided [14.4 to 66.5] — Difference between GSK2894512 0.5% QD and Vehicle QD at Week 14 has been presented
Statistical Analysis 22: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Proportion difference = 52.0, 95% CI 2-sided [23.2 to 74.4] — Difference between GSK2894512 1% BID and Vehicle BID at Week 16 has been presented
Statistical Analysis 23: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Proportion difference = 52.4, 95% CI 2-sided [24.4 to 74.0] — Difference between GSK2894512 1% QD and Vehicle QD at Week 16 has been presented
Statistical Analysis 24: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Proportion difference = 35.6, 95% CI 2-sided [6.3 to 60.5] — Difference between GSK2894512 0.5% BID and Vehicle BID at Week 16 has been presented
Statistical Analysis 25: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Proportion difference = 48.3, 95% CI 2-sided [19.7 to 71.1] — Difference between GSK2894512 0.5% QD and Vehicle QD at Week 16 has been presented
Statistical Analysis 26: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Proportion difference = 10.0, 95% CI 2-sided [-36.9 to 53.9] — Difference between GSK2894512 1% BID and Vehicle BID at EW has been presented
Statistical Analysis 27: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Proportion difference = 42.9, 95% CI 2-sided [-6.3 to 81.6] — Difference between GSK2894512 1% QD and Vehicle QD at EW has been presented

3. Secondary Outcome: Percentage of Participants With a Minimum 2 Grade Improvement in PGA Score From Baseline to Each Study Visit
Description: The PGA is a clinical tool for assessing the current state/severity of a participant's psoriasis. It is a static 5-point morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema, plaque thickness, and scaling as guidelines. Each assessment was made as a visual 'average' of the severity of all treated areas at the time of the assessment. The scores ranged from 0 to 4 where 0 = Clear, 1 = Almost Clear, 2 = Mild, 3 = Moderate and 4=Severe. The percentage of participants who achieved a minimum 2-grade improvement from Baseline for each study visit were summarized. Baseline was defined as the latest assessment prior to the first dose. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 16
Population: mITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 34 | 35 | 32 | 32 | 30 | 33
Percentage of participants
  Week 1, n=32, 35, 31, 32, 28, 32: number analyzed (Participants) | 32 | 35 | 31 | 32 | 28 | 32
  Week 1, n=32, 35, 31, 32, 28, 32 | 0 | 0 | 6 | 0 | 4 | 0
  Week 2, n=32, 33, 30, 32, 24, 30: number analyzed (Participants) | 32 | 33 | 30 | 32 | 24 | 30
  Week 2, n=32, 33, 30, 32, 24, 30 | 13 | 12 | 13 | 6 | 0 | 0
  Week 4, n=28, 31, 29, 32, 22, 26: number analyzed (Participants) | 28 | 31 | 29 | 32 | 22 | 26
  Week 4, n=28, 31, 29, 32, 22, 26 | 21 | 23 | 24 | 13 | 5 | 0
  Week 8, n=26, 27, 27, 32, 20, 20: number analyzed (Participants) | 26 | 27 | 27 | 32 | 20 | 20
  Week 8, n=26, 27, 27, 32, 20, 20 | 46 | 37 | 41 | 41 | 0 | 0
  Week 12, n=23, 25, 26, 28, 19, 20: number analyzed (Participants) | 23 | 25 | 26 | 28 | 19 | 20
  Week 12, n=23, 25, 26, 28, 19, 20 | 65 | 56 | 50 | 36 | 11 | 5
  Week 14, n=23, 26, 24, 27, 19, 19: number analyzed (Participants) | 23 | 26 | 24 | 27 | 19 | 19
  Week 14, n=23, 26, 24, 27, 19, 19 | 61 | 62 | 38 | 37 | 5 | 0
  Week 16, n=24, 26, 26, 28, 19, 19: number analyzed (Participants) | 24 | 26 | 26 | 28 | 19 | 19
  Week 16, n=24, 26, 26, 28, 19, 19 | 58 | 54 | 38 | 36 | 5 | 0
  EW, n=10, 7, 4, 2, 10, 9: number analyzed (Participants) | 10 | 7 | 4 | 2 | 10 | 9
  EW, n=10, 7, 4, 2, 10, 9 | 20 | 43 | 25 | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants With a PGA Score of 0 or 1 at Each Study Visit
Description: The PGA is a clinical tool for assessing the current state/severity of a participant's psoriasis. It is a static 5-point morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema, plaque thickness, and scaling as guidelines. Each assessment was made as a visual 'average' of the severity of all treated areas at the time of the assessment. The scores ranged from 0 to 4 where 0 = Clear, 1 = Almost Clear, 2 = Mild, 3 = Moderate and 4=Severe. The percentage of participants who achieved a PGA score of 0 or 1 from Baseline at each study visit was summarized. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Up to Week 16
Population: mITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 34 | 35 | 32 | 32 | 30 | 33
Percentage of participants
  Week 1, n=32, 35, 31, 32, 28, 32: number analyzed (Participants) | 32 | 35 | 31 | 32 | 28 | 32
  Week 1, n=32, 35, 31, 32, 28, 32 | 0 | 9 | 3 | 0 | 4 | 0
  Week 2, n=32, 33, 30, 32, 24, 30: number analyzed (Participants) | 32 | 33 | 30 | 32 | 24 | 30
  Week 2, n=32, 33, 30, 32, 24, 30 | 16 | 18 | 10 | 6 | 0 | 0
  Week 4, n=28, 31, 29, 32, 22, 26: number analyzed (Participants) | 28 | 31 | 29 | 32 | 22 | 26
  Week 4, n=28, 31, 29, 32, 22, 26 | 21 | 42 | 24 | 16 | 5 | 4
  Week 8, n=26, 27, 27, 32, 20, 20: number analyzed (Participants) | 26 | 27 | 27 | 32 | 20 | 20
  Week 8, n=26, 27, 27, 32, 20, 20 | 54 | 56 | 44 | 41 | 0 | 5
  Week 12, n=23, 25, 26, 28, 19, 20: number analyzed (Participants) | 23 | 25 | 26 | 28 | 19 | 20
  Week 12, n=23, 25, 26, 28, 19, 20 | 70 | 72 | 54 | 39 | 11 | 10
  Week 14, n=23, 26, 24, 27, 19, 19: number analyzed (Participants) | 23 | 26 | 24 | 27 | 19 | 19
  Week 14, n=23, 26, 24, 27, 19, 19 | 61 | 69 | 42 | 41 | 5 | 5
  Week 16, n=24, 26, 26, 28, 19, 19: number analyzed (Participants) | 24 | 26 | 26 | 28 | 19 | 19
  Week 16, n=24, 26, 26, 28, 19, 19 | 58 | 65 | 50 | 43 | 5 | 5
  EW, n=10, 7, 4, 2, 10, 9: number analyzed (Participants) | 10 | 7 | 4 | 2 | 10 | 9
  EW, n=10, 7, 4, 2, 10, 9 | 10 | 57 | 25 | 0 | 0 | 0

5. Secondary Outcome: Mean Change in Percent of BSA Affected With Psoriasis From Baseline to Each Study Visit
Description: The extent of BSA affected by psoriasis is a general indicator of disease severity and was measured throughout the study. The extent of BSA to which study treatment was applied was also recorded. For the purpose of approximate clinical estimation, the total palmar surface of the palm plus 5 digits was assumed to be approximately equivalent to 1 percent BSA. Assessment of BSA affected with psoriasis was performed separately for four body surface regions: the head, the upper extremities, the trunk and the lower extremities, corresponding to 10, 20, 30 and 40 percent of the total body area, respectively. The mean change in percent BSA affected from Baseline was summarized for each study visit. Baseline was defined as the latest assessment prior to the first dose and change from Baseline was defined as the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 16
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Percentage of BSA
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 34 | 35 | 32 | 32 | 30 | 33
Percentage of BSA
  Week 1, n=32, 35, 31, 32, 28, 32: number analyzed (Participants) | 32 | 35 | 31 | 32 | 28 | 32
  Week 1, n=32, 35, 31, 32, 28, 32 | -0.53 (1.136) | -0.30 (0.990) | -0.35 (0.774) | 0.02 (0.773) | -0.05 (0.510) | 0.01 (0.277)
  Week 2, n=32, 33, 30, 32, 24, 30: number analyzed (Participants) | 32 | 33 | 30 | 32 | 24 | 30
  Week 2, n=32, 33, 30, 32, 24, 30 | -1.06 (1.496) | -0.75 (1.789) | -0.79 (1.350) | -0.51 (1.157) | -0.18 (0.657) | -0.13 (1.159)
  Week 4, n=28, 31, 29, 32, 22, 26: number analyzed (Participants) | 28 | 31 | 29 | 32 | 22 | 26
  Week 4, n=28, 31, 29, 32, 22, 26 | -2.14 (3.275) | -2.13 (2.529) | -1.93 (2.951) | -0.80 (1.468) | -0.60 (1.332) | -0.17 (1.432)
  Week 8, n=26, 27, 27, 32, 20, 20: number analyzed (Participants) | 26 | 27 | 27 | 32 | 20 | 20
  Week 8, n=26, 27, 27, 32, 20, 20 | -3.37 (3.590) | -3.60 (3.220) | -3.51 (3.756) | -1.77 (2.800) | -1.05 (1.823) | -0.65 (1.435)
  Week 12, n=23, 25, 26, 28, 19, 20: number analyzed (Participants) | 23 | 25 | 26 | 28 | 19 | 20
  Week 12, n=23, 25, 26, 28, 19, 20 | -4.88 (4.211) | -4.28 (3.508) | -4.29 (3.882) | -3.59 (3.931) | -1.57 (2.380) | -0.98 (3.335)
  Week 14, n=23, 26, 24, 27, 19, 19: number analyzed (Participants) | 23 | 26 | 24 | 27 | 19 | 19
  Week 14, n=23, 26, 24, 27, 19, 19 | -5.01 (4.108) | -4.63 (3.548) | -4.26 (4.172) | -3.59 (4.201) | -1.33 (2.475) | -0.58 (3.634)
  Week 16, n=24, 26, 26, 28, 19, 19: number analyzed (Participants) | 24 | 26 | 26 | 28 | 19 | 19
  Week 16, n=24, 26, 26, 28, 19, 19 | -5.30 (4.468) | -4.47 (3.833) | -4.34 (4.299) | -3.56 (4.716) | -1.18 (2.490) | -1.10 (3.627)
  EW, n=10, 7, 4, 2, 10, 9: number analyzed (Participants) | 10 | 7 | 4 | 2 | 10 | 9
  EW, n=10, 7, 4, 2, 10, 9 | -1.92 (2.218) | -2.31 (3.465) | 0.25 (1.893) | 1.25 (9.546) | 0.74 (1.536) | 1.17 (2.094)

6. Secondary Outcome: Mean Change in PASI Score From Baseline to Each Study Visit
Description: The PASI is a standard clinical tool for assessing the severity of psoriasis based on severity of erythema, thickness and scale, as well as the extent of BSA affected with psoriasis. The 3 clinical signs were graded on a 5 point scale (0=None to 4=Severe) and the percent of BSA affected is scored on a 7-point scale (0=0% involvement to 6=90-100%) for each of 4 specified body regions (head, upper extremities, trunk and lower extremities). The individual scores were multiplied by a weighted factor for each body region. The sum of these scores gave the overall PASI score. PASI score ranged from 0=no psoriasis to 72=worse psoriasis. The mean change in PASI score from Baseline was summarized for each study visit. Baseline was the latest assessment prior to the first dose and change from Baseline was defined as the value at post dose visit minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 16
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 34 | 35 | 32 | 32 | 30 | 33
Scores on a scale
  Week 1, n=32, 35, 31, 32, 28, 32: number analyzed (Participants) | 32 | 35 | 31 | 32 | 28 | 32
  Week 1, n=32, 35, 31, 32, 28, 32 | -2.22 (2.795) | -1.73 (2.374) | -1.11 (2.083) | -1.33 (1.807) | -0.85 (1.203) | -0.28 (1.165)
  Week 2, n=32, 33, 30, 32, 24, 30: number analyzed (Participants) | 32 | 33 | 30 | 32 | 24 | 30
  Week 2, n=32, 33, 30, 32, 24, 30 | -4.10 (3.756) | -3.07 (3.016) | -2.39 (3.118) | -2.49 (2.316) | -1.78 (2.826) | -0.61 (1.644)
  Week 4, n=28, 31, 29, 32, 22, 26: number analyzed (Participants) | 28 | 31 | 29 | 32 | 22 | 26
  Week 4, n=28, 31, 29, 32, 22, 26 | -6.07 (5.051) | -4.45 (3.072) | -3.83 (3.827) | -3.31 (2.796) | -2.88 (3.308) | -1.08 (2.026)
  Week 8, n=26, 27, 27, 32, 20, 20: number analyzed (Participants) | 26 | 27 | 27 | 32 | 20 | 20
  Week 8, n=26, 27, 27, 32, 20, 20 | -7.52 (5.612) | -5.77 (3.556) | -5.79 (5.055) | -4.58 (3.902) | -2.82 (4.081) | -1.34 (2.288)
  Week 12, n=23, 25, 26, 28, 19, 20: number analyzed (Participants) | 23 | 25 | 26 | 28 | 19 | 20
  Week 12, n=23, 25, 26, 28, 19, 20 | -8.70 (5.617) | -6.62 (3.709) | -6.30 (5.138) | -5.41 (4.424) | -2.77 (4.291) | -1.54 (2.970)
  Week 14, n=23, 26, 24, 27, 19, 19: number analyzed (Participants) | 23 | 26 | 24 | 27 | 19 | 19
  Week 14, n=23, 26, 24, 27, 19, 19 | -8.61 (5.328) | -6.65 (3.973) | -5.67 (5.100) | -5.28 (4.422) | -2.60 (4.491) | -1.29 (3.280)
  Week 16, n=24, 26, 26, 28, 19, 19: number analyzed (Participants) | 24 | 26 | 26 | 28 | 19 | 19
  Week 16, n=24, 26, 26, 28, 19, 19 | -8.46 (5.432) | -6.63 (4.067) | -5.65 (5.646) | -5.13 (4.712) | -2.41 (4.285) | -1.09 (3.914)
  EW, n=10, 7, 4, 2, 10, 9: number analyzed (Participants) | 10 | 7 | 4 | 2 | 10 | 9
  EW, n=10, 7, 4, 2, 10, 9 | -3.70 (3.391) | -4.00 (3.636) | -1.18 (1.167) | 1.50 (8.627) | -0.06 (2.784) | 0.12 (2.742)

7. Secondary Outcome: PGA Scores at Each Study Visit
Description: The PGA is a clinical tool for assessing the current state/severity of a participant's psoriasis. It is a static 5-point morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema, plaque thickness, and scaling as guidelines. Each assessment was made as a visual 'average' of the severity of all treated areas at the time of the assessment. The scores ranged from 0 to 4 where 0 = Clear, 1 = Almost Clear, 2 = Mild, 3 = Moderate and 4=Severe. The mean of PGA scores at each study visit was summarized. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Up to Week 16
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 34 | 35 | 32 | 32 | 30 | 33
Scores on a scale
  Baseline, n=34, 35, 32, 32, 30, 33 | 2.9 (0.42) | 2.7 (0.51) | 3.0 (0.54) | 2.9 (0.39) | 3.0 (0.26) | 2.8 (0.44)
  Week 1, n=32, 35, 31, 32, 28, 32: number analyzed (Participants) | 32 | 35 | 31 | 32 | 28 | 32
  Week 1, n=32, 35, 31, 32, 28, 32 | 2.7 (0.59) | 2.4 (0.65) | 2.7 (0.65) | 2.6 (0.56) | 2.9 (0.52) | 2.8 (0.51)
  Week 2, n=32, 33, 30, 32, 24, 30: number analyzed (Participants) | 32 | 33 | 30 | 32 | 24 | 30
  Week 2, n=32, 33, 30, 32, 24, 30 | 2.3 (0.77) | 2.2 (0.71) | 2.4 (0.67) | 2.5 (0.62) | 2.6 (0.50) | 2.6 (0.49)
  Week 4, n=28, 31, 29, 32, 22, 26: number analyzed (Participants) | 28 | 31 | 29 | 32 | 22 | 26
  Week 4, n=28, 31, 29, 32, 22, 26 | 2.0 (0.67) | 1.6 (0.71) | 2.1 (0.77) | 2.1 (0.78) | 2.4 (0.59) | 2.6 (0.64)
  Week 8, n=26, 27, 27, 32, 20, 20: number analyzed (Participants) | 26 | 27 | 27 | 32 | 20 | 20
  Week 8, n=26, 27, 27, 32, 20, 20 | 1.5 (0.86) | 1.4 (0.80) | 1.6 (0.75) | 1.7 (0.85) | 2.5 (0.51) | 2.5 (0.61)
  Week 12, n=23, 25, 26, 28, 19, 20: number analyzed (Participants) | 23 | 25 | 26 | 28 | 19 | 20
  Week 12, n=23, 25, 26, 28, 19, 20 | 1.1 (0.92) | 1.1 (0.81) | 1.3 (1.01) | 1.6 (0.78) | 2.4 (0.69) | 2.5 (0.69)
  Week 14, n=23, 26, 24, 27, 19, 19: number analyzed (Participants) | 23 | 26 | 24 | 27 | 19 | 19
  Week 14, n=23, 26, 24, 27, 19, 19 | 1.3 (1.01) | 1.1 (0.99) | 1.6 (0.88) | 1.7 (0.94) | 2.5 (0.61) | 2.5 (0.61)
  Week 16, n=24, 26, 26, 28, 19, 19: number analyzed (Participants) | 24 | 26 | 26 | 28 | 19 | 19
  Week 16, n=24, 26, 26, 28, 19, 19 | 1.3 (1.08) | 1.2 (1.01) | 1.5 (0.90) | 1.7 (1.06) | 2.5 (0.61) | 2.6 (0.69)
  EW, n=10, 7, 4, 2, 10, 9: number analyzed (Participants) | 10 | 7 | 4 | 2 | 10 | 9
  EW, n=10, 7, 4, 2, 10, 9 | 2.5 (1.08) | 1.6 (1.40) | 2.0 (1.41) | 2.5 (0.71) | 3.1 (0.57) | 3.1 (0.60)

8. Secondary Outcome: Mean Change in PGA Score From Baseline to Each Study Visit
Description: The PGA is a clinical tool for assessing the current state/severity of a participant's psoriasis. It is a static 5-point morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema, plaque thickness, and scaling as guidelines. Each assessment was made as a visual 'average' of the severity of all treated areas at the time of the assessment. The scores ranged from 0 to 4 where 0 = Clear, 1 = Almost Clear, 2 = Mild, 3 = Moderate and 4=Severe. The mean change in PGA scores from Baseline was summarized for each study visit. Baseline was defined as the latest assessment prior to the first dose and change from Baseline was defined as the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 16
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 34 | 35 | 32 | 32 | 30 | 33
Scores on a scale
  Week 1, n=32, 35, 31, 32, 28, 32: number analyzed (Participants) | 32 | 35 | 31 | 32 | 28 | 32
  Week 1, n=32, 35, 31, 32, 28, 32 | -0.3 (0.44) | -0.3 (0.48) | -0.3 (0.69) | -0.3 (0.47) | -0.1 (0.52) | -0.1 (0.30)
  Week 2, n=32, 33, 30, 32, 24, 30: number analyzed (Participants) | 32 | 33 | 30 | 32 | 24 | 30
  Week 2, n=32, 33, 30, 32, 24, 30 | -0.7 (0.75) | -0.6 (0.70) | -0.6 (0.77) | -0.4 (0.62) | -0.4 (0.49) | -0.2 (0.50)
  Week 4, n=28, 31, 29, 32, 22, 26: number analyzed (Participants) | 28 | 31 | 29 | 32 | 22 | 26
  Week 4, n=28, 31, 29, 32, 22, 26 | -1.0 (0.69) | -1.1 (0.70) | -0.9 (0.83) | -0.8 (0.78) | -0.5 (0.60) | -0.2 (0.51)
  Week 8, n=26, 27, 27, 32, 20, 20: number analyzed (Participants) | 26 | 27 | 27 | 32 | 20 | 20
  Week 8, n=26, 27, 27, 32, 20, 20 | -1.4 (0.90) | -1.3 (0.88) | -1.4 (0.84) | -1.2 (0.97) | -0.5 (0.60) | -0.4 (0.49)
  Week 12, n=23, 25, 26, 28, 19, 20: number analyzed (Participants) | 23 | 25 | 26 | 28 | 19 | 20
  Week 12, n=23, 25, 26, 28, 19, 20 | -1.8 (0.90) | -1.7 (1.03) | -1.7 (1.06) | -1.3 (0.81) | -0.5 (0.77) | -0.4 (0.67)
  Week 14, n=23, 26, 24, 27, 19, 19: number analyzed (Participants) | 23 | 26 | 24 | 27 | 19 | 19
  Week 14, n=23, 26, 24, 27, 19, 19 | -1.7 (0.93) | -1.6 (1.20) | -1.4 (0.88) | -1.2 (0.92) | -0.5 (0.70) | -0.4 (0.50)
  Week 16, n=24, 26, 26, 28, 19, 19: number analyzed (Participants) | 24 | 26 | 26 | 28 | 19 | 19
  Week 16, n=24, 26, 26, 28, 19, 19 | -1.6 (1.01) | -1.6 (1.24) | -1.4 (0.90) | -1.3 (1.00) | -0.4 (0.69) | -0.3 (0.56)
  EW, n=10, 7, 4, 2, 10, 9: number analyzed (Participants) | 10 | 7 | 4 | 2 | 10 | 9
  EW, n=10, 7, 4, 2, 10, 9 | -0.5 (1.18) | -1.3 (1.38) | -1.0 (1.41) | 0.0 (1.41) | 0.0 (0.47) | 0.1 (0.60)

9. Secondary Outcome: Mean Change in Individual Target Lesion Grading Scores From Baseline to Each Study Visit
Description: A single target lesion of at least 3 centimeter (cm) x 3 cm was selected at Baseline. For the selected lesion, the severity of erythema, scaling and plaque thickness (induration) was assessed by the investigator on a 5-point scale ranging from 0=none to 4=severe. The mean change in individual grading scores from Baseline was summarized for each study visit. Baseline was defined as the latest assessment prior to the first dose and change from Baseline was defined as the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 16
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 34 | 35 | 32 | 32 | 30 | 33
Scores on a scale
  Scaling; Week 1, n=32, 35, 31, 32, 28, 32: number analyzed (Participants) | 32 | 35 | 31 | 32 | 28 | 32
  Scaling; Week 1, n=32, 35, 31, 32, 28, 32 | -0.7 (0.70) | -0.7 (0.90) | -0.4 (0.76) | -0.6 (0.56) | -0.5 (0.69) | -0.3 (0.44)
  Scaling; Week 2, n=32, 33, 30, 32, 24, 30: number analyzed (Participants) | 32 | 33 | 30 | 32 | 24 | 30
  Scaling; Week 2, n=32, 33, 30, 32, 24, 30 | -0.9 (0.78) | -1.0 (1.07) | -0.9 (0.87) | -1.0 (0.84) | -1.0 (0.75) | -0.3 (0.80)
  Scaling; Week 4, n=28, 31, 29, 32, 22, 26: number analyzed (Participants) | 28 | 31 | 29 | 32 | 22 | 26
  Scaling; Week 4, n=28, 31, 29, 32, 22, 26 | -1.5 (0.88) | -1.5 (1.21) | -1.4 (0.95) | -1.4 (0.98) | -1.0 (0.84) | -0.4 (0.80)
  Scaling; Week 8, n=26, 27, 27, 32, 20, 20: number analyzed (Participants) | 26 | 27 | 27 | 32 | 20 | 20
  Scaling; Week 8, n=26, 27, 27, 32, 20, 20 | -2.0 (1.11) | -2.0 (1.19) | -1.7 (1.07) | -1.9 (1.03) | -1.2 (0.93) | -0.4 (0.81)
  Scaling; Week 12, n=23, 25, 26, 29, 19, 20: number analyzed (Participants) | 23 | 25 | 26 | 29 | 19 | 20
  Scaling; Week 12, n=23, 25, 26, 29, 19, 20 | -2.3 (0.96) | -2.4 (1.15) | -2.1 (1.07) | -2.0 (1.05) | -1.0 (1.11) | -0.7 (0.81)
  Scaling; Week 14, n=23, 26, 24, 27, 19, 19: number analyzed (Participants) | 23 | 26 | 24 | 27 | 19 | 19
  Scaling; Week 14, n=23, 26, 24, 27, 19, 19 | -2.1 (1.20) | -2.2 (1.43) | -1.7 (1.17) | -1.8 (1.37) | -0.7 (1.05) | -0.5 (0.77)
  Scaling; Week 16, n=24, 26, 26, 28, 19, 19: number analyzed (Participants) | 24 | 26 | 26 | 28 | 19 | 19
  Scaling; Week 16, n=24, 26, 26, 28, 19, 19 | -2.1 (1.19) | -2.2 (1.24) | -1.6 (1.45) | -1.8 (1.29) | -0.6 (1.07) | -0.3 (0.67)
  Scaling; EW, n=10, 7, 4, 2, 10, 9: number analyzed (Participants) | 10 | 7 | 4 | 2 | 10 | 9
  Scaling; EW, n=10, 7, 4, 2, 10, 9 | -1.5 (1.27) | -1.6 (1.27) | -1.3 (1.50) | -0.5 (0.71) | -0.5 (0.97) | 0.0 (0.71)
  Erythema; Week 1, n=32, 35, 31, 32, 28, 32: number analyzed (Participants) | 32 | 35 | 31 | 32 | 28 | 32
  Erythema; Week 1, n=32, 35, 31, 32, 28, 32 | -0.4 (0.66) | -0.5 (0.78) | -0.3 (0.64) | -0.4 (0.50) | -0.2 (0.48) | -0.1 (0.39)
  Erythema; Week 2, n=32, 33, 30, 32, 24, 30: number analyzed (Participants) | 32 | 33 | 30 | 32 | 24 | 30
  Erythema; Week 2, n=32, 33, 30, 32, 24, 30 | -0.8 (0.83) | -1.1 (0.97) | -0.7 (0.94) | -0.8 (0.74) | -0.3 (0.75) | -0.2 (0.48)
  Erythema; Week 4, n=28, 31, 29, 32, 22, 26: number analyzed (Participants) | 28 | 31 | 29 | 32 | 22 | 26
  Erythema; Week 4, n=28, 31, 29, 32, 22, 26 | -1.3 (0.90) | -1.5 (0.89) | -1.3 (0.85) | -1.1 (0.80) | -0.6 (0.85) | -0.4 (0.64)
  Erythema; Week 8, n=26, 27, 27, 32, 20, 20: number analyzed (Participants) | 26 | 27 | 27 | 32 | 20 | 20
  Erythema; Week 8, n=26, 27, 27, 32, 20, 20 | -1.8 (1.10) | -2.0 (1.04) | -1.9 (0.95) | -1.5 (0.92) | -0.8 (0.85) | -0.5 (0.76)
  Erythema; Week 12, n=23, 25, 26, 29, 19, 20: number analyzed (Participants) | 23 | 25 | 26 | 29 | 19 | 20
  Erythema; Week 12, n=23, 25, 26, 29, 19, 20 | -2.3 (1.10) | -2.5 (1.08) | -2.2 (1.01) | -1.9 (1.13) | -0.5 (1.07) | -0.8 (0.97)
  Erythema; Week 14, n=23, 26, 24, 27, 19, 19: number analyzed (Participants) | 23 | 26 | 24 | 27 | 19 | 19
  Erythema; Week 14, n=23, 26, 24, 27, 19, 19 | -2.1 (1.28) | -2.2 (1.21) | -1.9 (0.95) | -1.7 (1.27) | -0.6 (1.12) | -0.9 (0.91)
  Erythema; Week 16, n=24, 26, 26, 28, 19, 19: number analyzed (Participants) | 24 | 26 | 26 | 28 | 19 | 19
  Erythema; Week 16, n=24, 26, 26, 28, 19, 19 | -2.1 (1.23) | -2.3 (1.09) | -1.8 (1.10) | -2.0 (1.26) | -0.6 (0.96) | -0.5 (0.90)
  Erythema; EW, n=10, 7, 4, 2, 10, 9: number analyzed (Participants) | 10 | 7 | 4 | 2 | 10 | 9
  Erythema; EW, n=10, 7, 4, 2, 10, 9 | -1.3 (1.06) | -1.4 (1.40) | -0.8 (1.50) | 0.0 (1.41) | -0.5 (0.97) | -0.1 (0.60)
  Plaque thickness; Week 1, n=32,35,31,32,28,32: number analyzed (Participants) | 32 | 35 | 31 | 32 | 28 | 32
  Plaque thickness; Week 1, n=32,35,31,32,28,32 | -0.5 (0.67) | -0.5 (0.82) | -0.4 (0.56) | -0.3 (0.60) | -0.4 (0.50) | -0.2 (0.45)
  Plaque thickness; Week 2, n=32,33,30,32,24,30: number analyzed (Participants) | 32 | 33 | 30 | 32 | 24 | 30
  Plaque thickness; Week 2, n=32,33,30,32,24,30 | -0.9 (0.84) | -0.9 (1.01) | -0.9 (0.94) | -0.8 (0.80) | -0.7 (0.76) | -0.3 (0.66)
  Plaque thickness; Week 4, n=28,31,29,32,22,26: number analyzed (Participants) | 28 | 31 | 29 | 32 | 22 | 26
  Plaque thickness; Week 4, n=28,31,29,32,22,26 | -1.4 (1.03) | -1.5 (1.26) | -1.3 (1.00) | -1.2 (0.93) | -1.0 (0.65) | -0.4 (0.64)
  Plaque thickness; Week 8, n=26,27,27,32,20,20: number analyzed (Participants) | 26 | 27 | 27 | 32 | 20 | 20
  Plaque thickness; Week 8, n=26,27,27,32,20,20 | -1.8 (1.17) | -1.8 (1.15) | -1.8 (1.09) | -1.7 (1.12) | -0.9 (0.88) | -0.5 (0.60)
  Plaque thickness; Week 12, n=23,25,26,29,19,20: number analyzed (Participants) | 23 | 25 | 26 | 29 | 19 | 20
  Plaque thickness; Week 12, n=23,25,26,29,19,20 | -2.3 (0.93) | -2.1 (1.19) | -1.9 (1.20) | -1.9 (1.13) | -1.0 (0.94) | -0.7 (0.80)
  Plaque thickness; Week 14, n=23,26,24,27,19,19: number analyzed (Participants) | 23 | 26 | 24 | 27 | 19 | 19
  Plaque thickness; Week 14, n=23,26,24,27,19,19 | -2.1 (1.16) | -2.1 (1.20) | -1.8 (1.19) | -1.7 (1.32) | -0.9 (1.13) | -0.7 (0.87)
  Plaque thickness; Week 16, n=24,26 26,28,19,19: number analyzed (Participants) | 24 | 26 | 26 | 28 | 19 | 19
  Plaque thickness; Week 16, n=24,26 26,28,19,19 | -2.1 (1.19) | -2.1 (1.32) | -1.6 (1.39) | -1.8 (1.31) | -0.7 (1.10) | -0.4 (0.69)
  Plaque thickness; EW, n=10,7,4,2,10,9: number analyzed (Participants) | 10 | 7 | 4 | 2 | 10 | 9
  Plaque thickness; EW, n=10,7,4,2,10,9 | -1.3 (1.06) | -1.9 (1.21) | -1.0 (1.41) | 0.0 (0.00) | -0.6 (1.07) | 0.4 (0.73)

10. Secondary Outcome: Mean Change in Weekly Average Itch/Pruritus Numeric Rating Scale (NRS) From Baseline to Each Study Visit
Description: The participant reported itch severity was obtained from the response of the participants to the itch NRS item in the psoriasis symptom diary (PSD). PSD was developed to assess daily self-reports of psoriasis symptoms and the functional impact related to the underlying pathophysiology of the disease. The participants answered questions related to the severity and impact of the signs and symptoms daily using a 11 point NRS with scores ranging from 0 (absent) to 10 (worst imaginable). Mean change in itch/pruritis NRS from Baseline to each study visit was presented. Baseline was defined as the latest assessment prior to the first dose and change from Baseline was defined as the post dose weekly average value minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 16
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 34 | 35 | 32 | 32 | 30 | 33
Scores on a scale
  Week 1, n=28, 33, 21, 31, 21, 29: number analyzed (Participants) | 28 | 33 | 21 | 31 | 21 | 29
  Week 1, n=28, 33, 21, 31, 21, 29 | -0.66 (1.800) | -0.17 (2.007) | -1.00 (2.038) | -0.32 (1.710) | -1.31 (1.689) | -0.63 (1.612)
  Week 2, n=27, 30, 22, 32, 20, 25: number analyzed (Participants) | 27 | 30 | 22 | 32 | 20 | 25
  Week 2, n=27, 30, 22, 32, 20, 25 | -1.62 (2.334) | -0.85 (1.870) | -1.97 (2.366) | -1.24 (1.949) | -1.66 (2.444) | -1.12 (2.147)
  Week 4, n=20, 25, 21, 30, 17, 24: number analyzed (Participants) | 20 | 25 | 21 | 30 | 17 | 24
  Week 4, n=20, 25, 21, 30, 17, 24 | -2.35 (3.057) | -1.78 (2.402) | -3.13 (2.075) | -1.91 (2.723) | -1.67 (2.727) | -1.31 (2.338)
  Week 8, n=18, 22, 20, 29, 16, 20: number analyzed (Participants) | 18 | 22 | 20 | 29 | 16 | 20
  Week 8, n=18, 22, 20, 29, 16, 20 | -3.66 (3.248) | -1.93 (2.543) | -3.29 (2.605) | -2.06 (2.842) | -1.98 (3.239) | -1.43 (2.664)
  Week 12, n=14, 20, 21, 24, 15, 18: number analyzed (Participants) | 14 | 20 | 21 | 24 | 15 | 18
  Week 12, n=14, 20, 21, 24, 15, 18 | -3.53 (2.933) | -2.59 (2.923) | -3.65 (2.605) | -2.73 (2.922) | -2.46 (3.389) | -1.43 (2.765)
  Week 14, n=13, 14, 15, 24, 15, 13: number analyzed (Participants) | 13 | 14 | 15 | 24 | 15 | 13
  Week 14, n=13, 14, 15, 24, 15, 13 | -3.56 (2.698) | -3.52 (2.489) | -3.58 (2.296) | -2.24 (3.067) | -1.90 (2.643) | -2.19 (2.898)
  Week 16, n=10, 9, 12, 19, 13, 10: number analyzed (Participants) | 10 | 9 | 12 | 19 | 13 | 10
  Week 16, n=10, 9, 12, 19, 13, 10 | -3.67 (3.766) | -2.19 (2.695) | -3.66 (2.059) | -2.25 (2.992) | -2.36 (2.837) | -2.06 (3.225)
  EW, n=6, 3, 2, 0, 5, 5: number analyzed (Participants) | 6 | 3 | 2 | 0 | 5 | 5
  EW, n=6, 3, 2, 0, 5, 5 | -1.77 (1.647) | -0.07 (1.501) | -5.67 (6.128) |  | -1.79 (1.654) | -0.51 (1.391)

11. Secondary Outcome: Percentage of Participants Who Achieved a PGA Score of 0 or 1 and a Minimum 2 Grade Improvement From Baseline to Each Study Visit
Description: The PGA is a clinical tool for assessing the current state/severity of a participant's psoriasis. It is a static 5-point morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema, plaque thickness, and scaling as guidelines. Each assessment was made as a visual 'average' of the severity of all treated areas at the time of the assessment. The scores ranged from 0 to 4 where 0 = Clear, 1 = Almost Clear, 2 = Mild, 3 = Moderate and 4=Severe. The percentage of responders that is, participants who achieved a PGA score of 0 or 1 and a minimum 2-grade improvement from baseline were summarized. Baseline was defined as the latest assessment prior to the first dose and change from Baseline was defined as the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 16
Population: mITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 34 | 35 | 32 | 32 | 30 | 33
Percentage of participants
  Week 1, n=32, 35, 31, 32, 28, 32: number analyzed (Participants) | 32 | 35 | 31 | 32 | 28 | 32
  Week 1, n=32, 35, 31, 32, 28, 32 | 0 | 0 | 3 | 0 | 4 | 0
  Week 2, n=32, 33, 30, 32, 24, 30: number analyzed (Participants) | 32 | 33 | 30 | 32 | 24 | 30
  Week 2, n=32, 33, 30, 32, 24, 30 | 9 | 9 | 10 | 6 | 0 | 0
  Week 4, n=28, 31, 29, 32, 22, 26: number analyzed (Participants) | 28 | 31 | 29 | 32 | 22 | 26
  Week 4, n=28, 31, 29, 32, 22, 26 | 14 | 19 | 17 | 13 | 5 | 0
  Week 8, n=26, 27, 27, 32, 20, 20: number analyzed (Participants) | 26 | 27 | 27 | 32 | 20 | 20
  Week 8, n=26, 27, 27, 32, 20, 20 | 42 | 37 | 33 | 41 | 0 | 0
  Week 12, n=23, 25, 26, 28, 19, 20: number analyzed (Participants) | 23 | 25 | 26 | 28 | 19 | 20
  Week 12, n=23, 25, 26, 28, 19, 20 | 65 | 56 | 46 | 36 | 11 | 5
  Week 14, n=23, 26, 24, 27, 19, 19: number analyzed (Participants) | 23 | 26 | 24 | 27 | 19 | 19
  Week 14, n=23, 26, 24, 27, 19, 19 | 57 | 62 | 29 | 37 | 5 | 0
  Week 16, n=24, 26, 26, 28, 19, 19: number analyzed (Participants) | 24 | 26 | 26 | 28 | 19 | 19
  Week 16, n=24, 26, 26, 28, 19, 19 | 58 | 54 | 35 | 36 | 5 | 0
  EW, n=10, 7, 4, 2, 10, 9: number analyzed (Participants) | 10 | 7 | 4 | 2 | 10 | 9
  EW, n=10, 7, 4, 2, 10, 9 | 10 | 43 | 25 | 0 | 0 | 0
Statistical Analysis 1: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Proportion difference = -3.6, 95% CI 2-sided [-28.8 to 21.9] — Difference between GSK2894512 1% BID and Vehicle BID at Week 1 has been presented
Statistical Analysis 2: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Proportion difference = -0.3, 95% CI 2-sided [-25.4 to 25.1] — Difference between GSK2894512 0.5% BID and Vehicle BID at Week 1 has been presented
Statistical Analysis 3: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Proportion difference = 9.4, 95% CI 2-sided [-17.5 to 35.3] — Difference between GSK2894512 1% BID and Vehicle BID at Week 2 has been presented
Statistical Analysis 4: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Proportion difference = 9.1, 95% CI 2-sided [-15.4 to 33.3] — Difference between GSK2894512 1% QD and Vehicle QD at Week 2 has been presented
Statistical Analysis 5: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Proportion difference = 10.0, 95% CI 2-sided [-17.1 to 36.1] — Difference between GSK2894512 0.5% BID and Vehicle BID at Week 2 has been presented
Statistical Analysis 6: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Proportion difference = 6.3, 95% CI 2-sided [-19.3 to 31.0] — Difference between GSK2894512 0.5% QD and Vehicle QD at Week 2 has been presented
Statistical Analysis 7: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Proportion difference = 9.7, 95% CI 2-sided [-18.2 to 36.7] — Difference between GSK2894512 1% BID and Vehicle BID at Week 4 has been presented
Statistical Analysis 8: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Proportion difference = 19.4, 95% CI 2-sided [-6.9 to 43.6] — Difference between GSK2894512 1% QD and Vehicle QD at Week 4 has been presented
Statistical Analysis 9: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Proportion difference = 12.7, 95% CI 2-sided [-15.1 to 38.9] — Difference between GSK2894512 0.5% BID and Vehicle BID at Week 4 has been presented
Statistical Analysis 10: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Proportion difference = 12.5, 95% CI 2-sided [-13.6 to 37.4] — Difference between GSK2894512 0.5% QD and Vehicle QD at Week 4 has been presented
Statistical Analysis 11: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Proportion difference = 42.3, 95% CI 2-sided [13.8 to 66.0] — Difference between GSK2894512 1% BID and Vehicle BID at Week 8 has been presented
Statistical Analysis 12: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Proportion difference = 37.0, 95% CI 2-sided [8.7 to 61.3] — Difference between GSK2894512 1% QD and Vehicle QD at Week 8 has been presented
Statistical Analysis 13: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Proportion difference = 33.3, 95% CI 2-sided [4.8 to 58.2] — Difference between GSK2894512 0.5% BID and Vehicle BID at Week 8 has been presented
Statistical Analysis 14: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Proportion difference = 40.6, 95% CI 2-sided [12.8 to 63.9] — Difference between GSK2894512 0.5% QD and Vehicle QD at Week 8 has been presented
Statistical Analysis 15: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Proportion difference = 54.7, 95% CI 2-sided [25.9 to 76.6] — Difference between GSK2894512 1% BID and Vehicle BID at Week 12 has been presented
Statistical Analysis 16: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Proportion difference = 51.0, 95% CI 2-sided [22.2 to 73.2] — Difference between GSK2894512 1% QD and Vehicle QD at Week 12 has been presented
Statistical Analysis 17: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Proportion difference = 35.6, 95% CI 2-sided [6.3 to 60.5] — Difference between GSK2894512 0.5% BID and Vehicle BID at Week 12 has been presented
Statistical Analysis 18: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Proportion difference = 30.7, 95% CI 2-sided [1.6 to 55.9] — Difference between GSK2894512 0.5% QD and Vehicle QD at Week 12 has been presented
Statistical Analysis 19: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Proportion difference = 51.3, 95% CI 2-sided [22.0 to 74.0] — Difference between GSK2894512 1% BID and Vehicle BID at Week 14 has been presented
Statistical Analysis 20: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Proportion difference = 61.5, 95% CI 2-sided [34.6 to 81.0] — Difference between GSK2894512 1% QD and Vehicle QD at Week 14 has been presented
Statistical Analysis 21: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Proportion difference = 23.9, 95% CI 2-sided [-6.1 to 51.0] — Difference between GSK2894512 0.5% BID and Vehicle BID at Week 14 has been presented
Statistical Analysis 22: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Proportion difference = 37.0, 95% CI 2-sided [7.8 to 61.6] — Difference between GSK2894512 0.5% QD and Vehicle QD at Week 14 has been presented
Statistical Analysis 23: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Proportion difference = 53.1, 95% CI 2-sided [24.7 to 75.6] — Difference between GSK2894512 1% BID and Vehicle BID at Week 16 has been presented
Statistical Analysis 24: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Proportion difference = 53.8, 95% CI 2-sided [25.8 to 75.5] — Difference between GSK2894512 1% QD and Vehicle QD at Week 16 has been presented
Statistical Analysis 25: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Proportion difference = 29.4, 95% CI 2-sided [-0.3 to 55.0] — Difference between GSK2894512 0.5% BID and Vehicle BID at Week 16 has been presented
Statistical Analysis 26: Comparison: GSK2894512 0.5% QD vs Vehicle QD; Test type: Other; Proportion difference = 35.7, 95% CI 2-sided [6.5 to 60.2] — Difference between GSK2894512 0.5% QD and Vehicle QD at Week 16 has been presented
Statistical Analysis 27: Comparison: GSK2894512 1% BID vs Vehicle BID; Test type: Other; Proportion difference = 10.0, 95% CI 2-sided [-36.9 to 53.9] — Difference between GSK2894512 1% BID and Vehicle BID at EW has been presented
Statistical Analysis 28: Comparison: GSK2894512 1% QD vs Vehicle QD; Test type: Other; Proportion difference = 42.9, 95% CI 2-sided [-6.3 to 81.6] — Difference between GSK2894512 1% QD and Vehicle QD at EW has been presented
Statistical Analysis 29: Comparison: GSK2894512 0.5% BID vs Vehicle BID; Test type: Other; Proportion difference = 25.0, 95% CI 2-sided [-35.7 to 80.6] — Difference between GSK2894512 0.5% BID and Vehicle BID at EW has been presented

12. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE is defined as any untoward medical occurrence in a participant under clinical investigation, temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/ birth defect, other situations and is associated with liver injury or impaired liver function. A TEAE is defined as an AE which occurred on or after study treatment start date and on or before the last visit. Number of participants with AEs and SAEs were presented. The analysis was performed on safety Population which comprised of all participants who received at least one dose of study treatment.
Time Frame: Up to Week 16
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
Participants
  TEAEs | 26 | 20 | 22 | 17 | 9 | 10
  serious TEAEs | 1 | 3 | 3 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Reported Local Tolerability Scores
Description: The assessment of the presence and degree of burning/stinging and itching at the application site following application of the study treatment was done at each specified study visit using a 5 point tolerability scale. The scores ranged from 0 to 4 where 0=None and 4=Strong/Severe. The score represented an average across all application sites. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Up to Week 14
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
Participants
  Week 1, none, n=36, 38, 37,38, 35, 37: number analyzed (Participants) | 36 | 38 | 37 | 38 | 35 | 37
  Week 1, none, n=36, 38, 37,38, 35, 37 | 19 | 17 | 18 | 26 | 19 | 26
  Week 1, slight, n=36, 38, 37,38, 35, 37: number analyzed (Participants) | 36 | 38 | 37 | 38 | 35 | 37
  Week 1, slight, n=36, 38, 37,38, 35, 37 | 4 | 8 | 7 | 1 | 6 | 8
  Week 1, mild, n=36, 38, 37,38, 35, 37: number analyzed (Participants) | 36 | 38 | 37 | 38 | 35 | 37
  Week 1, mild, n=36, 38, 37,38, 35, 37 | 8 | 9 | 5 | 8 | 6 | 2
  Week 1, moderate, n=36, 38, 37,38, 35, 37: number analyzed (Participants) | 36 | 38 | 37 | 38 | 35 | 37
  Week 1, moderate, n=36, 38, 37,38, 35, 37 | 4 | 4 | 6 | 3 | 2 | 1
  Week 1, strong/severe, n=36, 38, 37,38, 35, 37: number analyzed (Participants) | 36 | 38 | 37 | 38 | 35 | 37
  Week 1, strong/severe, n=36, 38, 37,38, 35, 37 | 1 | 0 | 1 | 0 | 2 | 0
  Week 2, none, n=36, 36, 36,38, 31, 35: number analyzed (Participants) | 36 | 36 | 36 | 38 | 31 | 35
  Week 2, none, n=36, 36, 36,38, 31, 35 | 24 | 28 | 20 | 31 | 23 | 26
  Week 2, slight, n=36, 36, 36,38, 31, 35: number analyzed (Participants) | 36 | 36 | 36 | 38 | 31 | 35
  Week 2, slight, n=36, 36, 36,38, 31, 35 | 4 | 4 | 7 | 4 | 4 | 5
  Week 2, mild, n=36, 36, 36,38, 31, 35: number analyzed (Participants) | 36 | 36 | 36 | 38 | 31 | 35
  Week 2, mild, n=36, 36, 36,38, 31, 35 | 7 | 4 | 3 | 2 | 1 | 4
  Week 2, moderate, n=36, 36, 36,38, 31, 35: number analyzed (Participants) | 36 | 36 | 36 | 38 | 31 | 35
  Week 2, moderate, n=36, 36, 36,38, 31, 35 | 1 | 0 | 6 | 1 | 1 | 0
  Week 2, strong/severe, n=36, 36, 36,38, 31, 35: number analyzed (Participants) | 36 | 36 | 36 | 38 | 31 | 35
  Week 2, strong/severe, n=36, 36, 36,38, 31, 35 | 0 | 0 | 0 | 0 | 2 | 0
  Week 4, none, n=32, 34, 35,38, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 38 | 29 | 31
  Week 4, none, n=32, 34, 35,38, 29, 31 | 19 | 24 | 23 | 32 | 21 | 26
  Week 4, slight, n=32, 34, 35,38, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 38 | 29 | 31
  Week 4, slight, n=32, 34, 35,38, 29, 31 | 7 | 5 | 4 | 2 | 3 | 3
  Week 4, mild, n=32, 34, 35,38, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 38 | 29 | 31
  Week 4, mild, n=32, 34, 35,38, 29, 31 | 4 | 4 | 5 | 3 | 3 | 1
  Week 4, moderate, n=32, 34, 35,38, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 38 | 29 | 31
  Week 4, moderate, n=32, 34, 35,38, 29, 31 | 2 | 1 | 3 | 1 | 1 | 1
  Week 4, strong/severe, n=32, 34, 35,38, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 38 | 29 | 31
  Week 4, strong/severe, n=32, 34, 35,38, 29, 31 | 0 | 0 | 0 | 0 | 1 | 0
  Week 8, none, n=30, 31, 33,38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  Week 8, none, n=30, 31, 33,38, 27, 26 | 24 | 24 | 24 | 33 | 24 | 22
  Week 8, slight, n=30, 31, 33,38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  Week 8, slight, n=30, 31, 33,38, 27, 26 | 4 | 7 | 5 | 3 | 3 | 2
  Week 8, mild, n=30, 31, 33,38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  Week 8, mild, n=30, 31, 33,38, 27, 26 | 1 | 0 | 3 | 1 | 0 | 0
  Week 8, moderate, n=30, 31, 33,38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  Week 8, moderate, n=30, 31, 33,38, 27, 26 | 1 | 0 | 1 | 1 | 0 | 2
  Week 8, strong/severe, n=30, 31, 33,38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  Week 8, strong/severe, n=30, 31, 33,38, 27, 26 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12, none, n=27, 29, 32,35, 26, 25: number analyzed (Participants) | 27 | 29 | 32 | 35 | 26 | 25
  Week 12, none, n=27, 29, 32,35, 26, 25 | 20 | 24 | 25 | 31 | 24 | 23
  Week 12, slight, n=27, 29, 32,35, 26, 25: number analyzed (Participants) | 27 | 29 | 32 | 35 | 26 | 25
  Week 12, slight, n=27, 29, 32,35, 26, 25 | 4 | 2 | 3 | 3 | 2 | 1
  Week 12, mild, n=27, 29, 32,35, 26, 25: number analyzed (Participants) | 27 | 29 | 32 | 35 | 26 | 25
  Week 12, mild, n=27, 29, 32,35, 26, 25 | 2 | 3 | 3 | 1 | 0 | 0
  Week 12, moderate, n=27, 29, 32,35, 26, 25: number analyzed (Participants) | 27 | 29 | 32 | 35 | 26 | 25
  Week 12, moderate, n=27, 29, 32,35, 26, 25 | 1 | 0 | 1 | 0 | 0 | 1
  Week 12, strong/severe, n=27, 29, 32,35, 26, 25: number analyzed (Participants) | 27 | 29 | 32 | 35 | 26 | 25
  Week 12, strong/severe, n=27, 29, 32,35, 26, 25 | 0 | 0 | 0 | 0 | 0 | 0
  Week 14, none, n=27, 30, 33, 33, 27, 24: number analyzed (Participants) | 27 | 30 | 33 | 33 | 27 | 24
  Week 14, none, n=27, 30, 33, 33, 27, 24 | 24 | 25 | 25 | 31 | 25 | 23
  Week 14, slight, n=27, 30, 33, 33, 27, 24: number analyzed (Participants) | 27 | 30 | 33 | 33 | 27 | 24
  Week 14, slight, n=27, 30, 33, 33, 27, 24 | 1 | 3 | 3 | 2 | 1 | 0
  Week 14, mild, n=27, 30, 33, 33, 27, 24: number analyzed (Participants) | 27 | 30 | 33 | 33 | 27 | 24
  Week 14, mild, n=27, 30, 33, 33, 27, 24 | 1 | 1 | 3 | 0 | 1 | 0
  Week 14, moderate, n=27, 30, 33, 33, 27, 24: number analyzed (Participants) | 27 | 30 | 33 | 33 | 27 | 24
  Week 14, moderate, n=27, 30, 33, 33, 27, 24 | 1 | 1 | 2 | 0 | 0 | 1
  Week 14, strong/severe, n=27, 30, 33, 33, 27, 24: number analyzed (Participants) | 27 | 30 | 33 | 33 | 27 | 24
  Week 14, strong/severe, n=27, 30, 33, 33, 27, 24 | 0 | 0 | 0 | 0 | 0 | 0
  EW, none, n=9, 7, 4, 2, 10, 9: number analyzed (Participants) | 9 | 7 | 4 | 2 | 10 | 9
  EW, none, n=9, 7, 4, 2, 10, 9 | 4 | 2 | 0 | 2 | 4 | 8
  EW, slight, n=9, 7, 4, 2, 10, 9: number analyzed (Participants) | 9 | 7 | 4 | 2 | 10 | 9
  EW, slight, n=9, 7, 4, 2, 10, 9 | 1 | 2 | 1 | 0 | 2 | 0
  EW, mild, n=9, 7, 4, 2, 10, 9: number analyzed (Participants) | 9 | 7 | 4 | 2 | 10 | 9
  EW, mild, n=9, 7, 4, 2, 10, 9 | 0 | 0 | 2 | 0 | 2 | 0
  EW, moderate, n=9, 7, 4, 2, 10, 9: number analyzed (Participants) | 9 | 7 | 4 | 2 | 10 | 9
  EW, moderate, n=9, 7, 4, 2, 10, 9 | 2 | 1 | 0 | 0 | 1 | 1
  EW, strong/severe, n=9,7,4, 2, 10, 9: number analyzed (Participants) | 9 | 7 | 4 | 2 | 10 | 9
  EW, strong/severe, n=9,7,4, 2, 10, 9 | 2 | 2 | 1 | 0 | 1 | 0

14. Secondary Outcome: Change From Baseline in Albumin and Protein Level
Description: Blood samples were collected for the evaluation of change in albumin and protein levels from Baseline throughout the study. Baseline was defined as the latest assessment (including unscheduled visits) prior to the first dose and change from Baseline was defined as the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: grams/liter (g/L)
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
grams/liter (g/L)
  Albumin, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  Albumin, Week 2, n=35, 36, 35, 37, 29, 34 | -0.9 (2.11) | -1.1 (2.70) | -0.9 (2.83) | -1.1 (2.33) | -0.9 (3.37) | -0.6 (2.76)
  Albumin, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  Albumin, Week 4, n=32, 34, 33, 37, 29, 30 | -1.3 (2.10) | -1.2 (2.52) | -1.0 (3.57) | -0.4 (1.99) | -0.8 (3.53) | -0.2 (3.23)
  Albumin, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  Albumin, Week 8, n=30, 31, 32, 37, 27, 26 | -1.0 (1.65) | -0.6 (2.33) | -1.0 (3.33) | -1.0 (2.49) | -0.6 (3.19) | -1.0 (2.36)
  Albumin, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  Albumin, Week 12, n=27, 30, 32, 36, 26, 24 | -0.8 (2.19) | -0.5 (3.31) | -1.3 (3.39) | -1.2 (1.67) | -0.6 (3.14) | -1.1 (2.85)
  Albumin, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  Albumin, Week 14, n=29, 31, 33, 34, 27, 24 | -1.3 (2.74) | -1.1 (2.72) | -1.5 (2.71) | -1.1 (2.81) | -1.6 (4.24) | -2.0 (2.40)
  Albumin, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Albumin, EW, n=10, 6, 3, 2, 10, 9 | -0.3 (2.06) | -1.7 (2.50) | 0.0 (3.46) | -3.5 (3.54) | -0.8 (1.99) | -0.2 (2.54)
  Protein, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  Protein, Week 2, n=35, 36, 35, 37, 29, 34 | -1.1 (3.84) | -2.5 (3.95) | -1.3 (4.25) | -1.5 (3.07) | -1.8 (4.21) | -1.0 (4.25)
  Protein, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  Protein, Week 4, n=32, 34, 33, 37, 29, 30 | -2.3 (3.23) | -2.9 (3.41) | -0.9 (4.94) | -0.7 (3.37) | -1.9 (4.99) | -0.3 (4.70)
  Protein, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  Protein, Week 8, n=30, 31, 32, 37, 27, 26 | -2.1 (3.28) | -1.7 (3.74) | -1.9 (4.88) | -1.3 (3.89) | -1.5 (4.42) | -1.4 (3.30)
  Protein, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  Protein, Week 12, n=27, 30, 32, 36, 26, 24 | -1.3 (2.73) | -2.5 (3.72) | -2.4 (4.23) | -1.7 (3.27) | -1.8 (4.05) | -1.5 (3.84)
  Protein, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  Protein, Week 14, n=29, 31, 33, 34, 27, 24 | -2.1 (3.06) | -2.9 (3.61) | -2.4 (4.34) | -1.9 (4.01) | -3.0 (4.32) | -2.6 (2.81)
  Protein, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Protein, EW, n=10, 6, 3, 2, 10, 9 | -0.8 (2.66) | -3.5 (3.83) | -3.0 (5.00) | -3.5 (2.12) | -1.2 (3.52) | -0.2 (3.42)

15. Secondary Outcome: Change From Baseline in Alkaline Phosphatase (Alk Phos), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), and Gamma Glutamyl Transferase (GGT) Levels.
Description: Blood samples were collected for the evaluation of change in levels of alk phos, ALT, AST and GGT from Baseline throughout the study. Baseline was defined as the latest assessment (including unscheduled visits) prior to the first dose and change from Baseline was defined as the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International Units (IU)/L
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
International Units (IU)/L
  Alk. Phos, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  Alk. Phos, Week 2, n=35, 36, 35, 37, 29, 34 | -0.6 (10.83) | -0.9 (8.44) | -0.7 (13.47) | -2.9 (10.93) | 0.7 (18.06) | -2.1 (7.02)
  Alk. Phos, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  Alk. Phos, Week 4, n=32, 34, 33, 37, 29, 30 | -0.2 (20.50) | -0.6 (7.03) | 0.1 (13.51) | 0.4 (11.33) | -0.0 (14.42) | -2.9 (8.69)
  Alk. Phos, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  Alk. Phos, Week 8, n=30, 31, 32, 37, 27, 26 | -4.1 (17.59) | -1.2 (11.06) | -0.1 (9.53) | -3.9 (9.54) | 0.0 (12.56) | 2.3 (11.25)
  Alk. Phos, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  Alk. Phos, Week 12, n=27, 30, 32, 36, 26, 24 | -5.7 (18.74) | -3.1 (10.45) | -1.7 (9.29) | -2.3 (8.30) | -1.7 (15.72) | 1.2 (13.29)
  Alk. Phos, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  Alk. Phos, Week 14, n=29, 31, 33, 34, 27, 24 | -2.3 (15.62) | -4.1 (10.56) | -3.1 (12.34) | -4.9 (13.20) | -2.4 (16.98) | -2.8 (13.62)
  Alk. Phos, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Alk. Phos, EW, n=10, 6, 3, 2, 10, 9 | -3.7 (7.27) | 2.7 (10.95) | 7.7 (16.80) | -13.5 (6.36) | -3.4 (10.51) | -1.8 (9.13)
  ALT, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  ALT, Week 2, n=35, 36, 35, 37, 29, 34 | -2.1 (7.98) | -2.6 (7.95) | -2.3 (6.18) | -2.9 (9.75) | -2.7 (13.45) | -1.3 (4.54)
  ALT, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  ALT, Week 4, n=32, 34, 33, 37, 29, 30 | 0.3 (22.68) | -2.7 (5.99) | -3.7 (13.21) | -2.9 (9.91) | -2.4 (11.83) | 2.3 (9.10)
  ALT, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  ALT, Week 8, n=30, 31, 32, 37, 27, 26 | -1.5 (10.37) | -3.9 (12.47) | 0.1 (11.68) | -4.4 (10.88) | 0.3 (14.28) | -0.4 (10.21)
  ALT, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  ALT, Week 12, n=27, 30, 32, 36, 26, 24 | -1.8 (15.35) | -2.2 (8.25) | -0.1 (13.72) | -5.4 (9.54) | -2.6 (14.93) | 1.5 (20.39)
  ALT, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  ALT, Week 14, n=29, 31, 33, 34, 27, 24 | -3.8 (17.42) | -3.5 (10.37) | -1.8 (12.99) | -6.5 (10.33) | -1.4 (19.63) | -1.7 (9.27)
  ALT, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  ALT, EW, n=10, 6, 3, 2, 10, 9 | -1.1 (5.02) | -2.2 (7.31) | 5.0 (16.64) | -5.0 (7.07) | -8.2 (12.16) | -1.3 (5.52)
  AST, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  AST, Week 2, n=35, 36, 35, 37, 29, 34 | -0.6 (4.91) | -1.2 (5.09) | 0.5 (3.71) | -1.8 (11.91) | -2.3 (10.76) | -1.0 (5.70)
  AST, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  AST, Week 4, n=32, 34, 33, 37, 29, 30 | 0.2 (9.76) | -1.9 (3.21) | -1.0 (5.22) | -3.1 (11.61) | -1.9 (9.05) | 0.5 (6.66)
  AST, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  AST, Week 8, n=30, 31, 32, 37, 27, 26 | -1.0 (4.22) | -2.2 (6.32) | 2.6 (11.60) | -4.2 (11.50) | -0.3 (10.52) | -1.7 (8.47)
  AST, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  AST, Week 12, n=27, 30, 32, 36, 26, 24 | 0.6 (9.09) | -2.2 (7.49) | 1.9 (8.89) | -4.1 (9.90) | -1.6 (12.75) | -0.3 (8.45)
  AST, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  AST, Week 14, n=29, 31, 33, 34, 27, 24 | -0.4 (7.55) | -2.7 (8.76) | 0.7 (8.39) | -5.1 (11.36) | -1.3 (13.40) | -1.0 (6.92)
  AST, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  AST, EW, n=10, 6, 3, 2, 10, 9 | -1.0 (4.24) | 5.2 (15.84) | 1.7 (9.07) | -1.0 (4.24) | -3.7 (7.73) | -0.3 (7.48)
  GGT, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  GGT, Week 2, n=35, 36, 35, 37, 29, 34 | -1.0 (6.63) | -2.1 (8.38) | -0.4 (17.64) | -1.6 (14.39) | -3.1 (15.17) | -4.5 (9.92)
  GGT, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  GGT, Week 4, n=32, 34, 33, 37, 29, 30 | 8.5 (56.71) | -3.5 (17.84) | -4.6 (22.06) | 0.3 (15.40) | -2.5 (18.08) | -2.1 (11.77)
  GGT, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  GGT, Week 8, n=30, 31, 32, 37, 27, 26 | 1.9 (20.56) | -7.6 (32.91) | -1.2 (21.11) | -3.2 (20.11) | -3.1 (23.93) | -0.4 (13.61)
  GGT, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  GGT, Week 12, n=27, 30, 32, 36, 26, 24 | -0.1 (24.48) | -2.4 (12.78) | 2.1 (20.03) | -5.9 (12.56) | -3.7 (30.64) | 3.3 (23.10)
  GGT, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  GGT, Week 14, n=29, 31, 33, 34, 27, 24 | -1.9 (16.31) | -2.5 (11.69) | -0.1 (16.58) | -5.9 (17.67) | -0.5 (38.93) | -1.3 (11.15)
  GGT, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  GGT, EW, n=10, 6, 3, 2, 10, 9 | -2.0 (6.25) | -5.3 (7.42) | -2.0 (6.56) | -2.5 (7.78) | -2.6 (4.65) | -10.1 (25.73)

16. Secondary Outcome: Change From Baseline in Direct Bilirubin (Bil), Bilirubin (Bil), Creatinine and Urate.
Description: Blood samples were collected for the evaluation of change in levels of direct bil, bil, creatinine and urate from Baseline throughout the study. Baseline was defined as the latest assessment (including unscheduled visits) prior to the first dose and change from Baseline was defined as the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: micromoles (µmol)/L
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
micromoles (µmol)/L
  Direct bil, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  Direct bil, Week 2, n=35, 36, 35, 37, 29, 34 | -0.2 (0.81) | -0.4 (1.36) | 0.0 (1.08) | -0.1 (1.24) | -0.1 (1.51) | 0.0 (0.85)
  Direct bil, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  Direct bil, Week 4, n=32, 34, 33, 37, 29, 30 | -0.3 (0.67) | -0.5 (1.50) | -0.1 (1.17) | -0.2 (0.99) | -0.1 (1.36) | -0.1 (1.17)
  Direct bil, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  Direct bil, Week 8, n=30, 31, 32, 37, 27, 26 | -0.4 (0.97) | -0.3 (1.24) | -0.2 (0.93) | -0.2 (1.03) | -0.1 (1.35) | -0.5 (1.33)
  Direct bil, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  Direct bil, Week 12, n=27, 30, 32, 36, 26, 24 | -0.2 (0.64) | -0.3 (1.26) | -0.2 (1.18) | -0.4 (1.15) | 0.0 (1.26) | -0.1 (1.10)
  Direct bil, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  Direct bil, Week 14, n=29, 31, 33, 34, 27, 24 | 0.1 (1.19) | -0.3 (1.28) | -0.1 (1.06) | -0.1 (1.04) | 0.1 (1.52) | -0.2 (0.82)
  Direct bil, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Direct bil, EW, n=10, 6, 3, 2, 10, 9 | 0.2 (1.14) | 0.0 (0.00) | 0.0 (0.00) | 2.0 (0.00) | -0.4 (1.26) | -0.2 (1.20)
  Bil, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  Bil, Week 2, n=35, 36, 35, 37, 29, 34 | -0.7 (3.03) | -1.4 (3.24) | -0.6 (2.98) | -0.3 (2.56) | -0.3 (4.40) | 0.8 (4.15)
  Bil, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  Bil, Week 4, n=32, 34, 33, 37, 29, 30 | -0.4 (3.50) | -1.2 (3.42) | 0.4 (4.34) | -0.6 (2.87) | -0.6 (4.84) | 1.7 (4.29)
  Bil, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  Bil, Week 8, n=30, 31, 32, 37, 27, 26 | -0.3 (2.86) | 0.1 (2.73) | -0.8 (2.48) | -0.3 (3.06) | -0.9 (4.27) | 0.2 (3.81)
  Bil, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  Bil, Week 12, n=27, 30, 32, 36, 26, 24 | -0.2 (2.10) | -0.7 (2.70) | -0.9 (3.13) | -0.4 (3.13) | -0.4 (4.93) | 0.6 (4.02)
  Bil, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  Bil, Week 14, n=29, 31, 33, 34, 27, 24 | 0.6 (3.70) | -0.7 (4.34) | -0.9 (2.74) | -0.5 (3.56) | -0.8 (4.84) | 0.5 (2.96)
  Bil, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Bil, EW, n=10, 6, 3, 2, 10, 9 | -0.8 (2.53) | 0.0 (2.19) | 2.7 (3.06) | -1.0 (1.41) | 0.4 (3.10) | -0.2 (3.23)
  Creatinine, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  Creatinine, Week 2, n=35, 36, 35, 37, 29, 34 | -0.26 (7.565) | 0.86 (9.588) | 1.14 (7.202) | 0.27 (9.708) | -1.65 (5.812) | 1.22 (6.632)
  Creatinine, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  Creatinine, Week 4, n=32, 34, 33, 37, 29, 30 | -2.27 (6.493) | 0.12 (8.469) | 0.97 (7.802) | 1.81 (7.510) | -2.38 (6.095) | 1.57 (10.282)
  Creatinine, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  Creatinine, Week 8, n=30, 31, 32, 37, 27, 26 | -0.09 (6.792) | 0.55 (7.030) | 0.48 (7.086) | 2.82 (11.713) | -2.89 (7.566) | 1.40 (8.515)
  Creatinine, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  Creatinine, Week 12, n=27, 30, 32, 36, 26, 24 | 2.39 (7.526) | 0.14 (6.543) | 0.34 (6.852) | 0.37 (11.501) | -4.35 (10.528) | 1.49 (7.718)
  Creatinine, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  Creatinine, Week 14, n=29, 31, 33, 34, 27, 24 | 1.74 (5.748) | 1.67 (7.316) | 3.41 (7.309) | 1.67 (14.096) | -2.33 (9.715) | 3.06 (8.970)
  Creatinine, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Creatinine, EW, n=10, 6, 3, 2, 10, 9 | -0.80 (8.570) | -5.02 (9.374) | 21.77 (31.832) | -1.80 (0.000) | -1.58 (6.009) | -2.36 (5.544)
  Urate, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  Urate, Week 2, n=35, 36, 35, 37, 29, 34 | -6.0 (55.26) | -7.8 (40.29) | 15.4 (41.96) | 6.2 (61.07) | -8.3 (62.91) | -0.3 (62.06)
  Urate, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  Urate, Week 4, n=32, 34, 33, 37, 29, 30 | -12.5 (34.36) | -7.9 (43.82) | 11.2 (48.01) | 5.7 (49.36) | -10.7 (54.11) | 2.7 (52.06)
  Urate, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  Urate, Week 8, n=30, 31, 32, 37, 27, 26 | -5.0 (37.30) | -8.7 (37.13) | -3.8 (32.30) | -0.3 (45.43) | -6.3 (73.54) | -4.2 (75.80)
  Urate, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  Urate, Week 12, n=27, 30, 32, 36, 26, 24 | -6.3 (28.44) | 5.7 (34.51) | 1.6 (35.21) | -1.7 (55.01) | 0.4 (88.79) | 15.4 (66.27)
  Urate, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  Urate, Week 14, n=29, 31, 33, 34, 27, 24 | 3.1 (41.15) | 19.4 (71.04) | 16.4 (48.98) | -5.9 (54.72) | -14.1 (59.37) | -2.5 (65.62)
  Urate, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Urate, EW, n=10, 6, 3, 2, 10, 9 | -2.0 (35.21) | -38.3 (31.89) | 76.7 (98.15) | -10.0 (14.14) | -13.0 (33.68) | -13.3 (52.92)

17. Secondary Outcome: Change From Baseline in Calcium, Chloride, Carbon Dioxide (CO2), Glucose, Potassium, Sodium and Urea Levels
Description: Blood samples were collected for the evaluation of change in levels of calcium, chloride, CO2, glucose, potassium, sodium, and urea from Baseline throughout the study. Baseline was defined as the latest assessment (including unscheduled visits) prior to the first dose and change from Baseline was defined as the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: millimoles (mmol)/L
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
millimoles (mmol)/L
  Calcium, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  Calcium, Week 2, n=35, 36, 35, 37, 29, 34 | -0.036 (0.1241) | -0.036 (0.0935) | -0.041 (0.1411) | -0.036 (0.0967) | -0.048 (0.1239) | -0.006 (0.0887)
  Calcium, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  Calcium, Week 4, n=32, 34, 33, 37, 29, 30 | -0.037 (0.1003) | -0.045 (0.0788) | -0.033 (0.1306) | -0.014 (0.0899) | -0.036 (0.1451) | 0.003 (0.0830)
  Calcium, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  Calcium, Week 8, n=30, 31, 32, 37, 27, 26 | -0.034 (0.1205) | -0.015 (0.0853) | -0.036 (0.0951) | -0.010 (0.1000) | -0.039 (0.1131) | -0.017 (0.0948)
  Calcium, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  Calcium, Week 12, n=27, 30, 32, 36, 26, 24 | -0.019 (0.0910) | -0.013 (0.0934) | -0.034 (0.0845) | -0.021 (0.1129) | -0.032 (0.0988) | 0.011 (0.1127)
  Calcium, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  Calcium, Week 14, n=29, 31, 33, 34, 27, 24 | -0.028 (0.0912) | -0.030 (0.1067) | -0.029 (0.0930) | -0.025 (0.0935) | -0.045 (0.1270) | -0.020 (0.1052)
  Calcium, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Calcium, EW, n=10, 6, 3, 2, 10, 9 | -0.024 (0.0717) | -0.020 (0.0632) | 0.007 (0.1286) | -0.030 (0.0990) | -0.014 (0.0366) | 0.004 (0.0691)
  Chloride, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  Chloride, Week 2, n=35, 36, 35, 37, 29, 34 | -0.1 (2.30) | 0.3 (2.00) | -0.3 (1.98) | 0.1 (2.05) | 0.3 (2.44) | -0.0 (2.29)
  Chloride, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  Chloride, Week 4, n=32, 34, 33, 37, 29, 30 | -0.1 (1.66) | 0.5 (1.97) | -0.4 (2.56) | -0.5 (1.83) | 0.1 (2.62) | -0.7 (2.74)
  Chloride, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  Chloride, Week 8, n=30, 31, 32, 37, 27, 26 | 0.3 (1.73) | 0.6 (1.89) | -0.3 (2.02) | 0.3 (2.03) | -0.1 (2.13) | -0.3 (3.07)
  Chloride, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  Chloride, Week 12, n=27, 30, 32, 36, 26, 24 | -0.4 (2.62) | 0.7 (2.00) | 0.1 (2.29) | -0.2 (2.35) | 0.7 (2.37) | -0.7 (2.80)
  Chloride, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  Chloride, Week 14, n=29, 31, 33, 34, 27, 24 | 0.4 (2.24) | 0.5 (2.23) | -0.3 (2.31) | 0.5 (2.30) | -0.3 (2.84) | 0.2 (2.55)
  Chloride, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Chloride, EW, n=10, 6, 3, 2, 10, 9 | -0.8 (3.19) | -1.5 (0.84) | -1.0 (2.00) | 1.0 (1.41) | 0.0 (2.31) | -1.9 (2.98)
  CO2, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  CO2, Week 2, n=35, 36, 35, 37, 29, 34 | -1.6 (2.13) | -1.1 (2.48) | -1.2 (2.64) | -1.2 (1.96) | -0.6 (2.37) | -0.9 (2.04)
  CO2, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  CO2, Week 4, n=32, 34, 33, 37, 29, 30 | -1.0 (2.21) | -1.4 (2.57) | -2.0 (2.81) | -0.8 (2.12) | -0.5 (1.99) | -1.5 (2.50)
  CO2, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  CO2, Week 8, n=30, 31, 32, 37, 27, 26 | -1.6 (2.19) | -1.5 (2.49) | -1.3 (1.89) | -1.0 (2.25) | -1.0 (1.85) | -1.5 (2.47)
  CO2, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  CO2, Week 12, n=27, 30, 32, 36, 26, 24 | -1.0 (1.58) | -1.1 (1.87) | -1.2 (2.55) | -1.1 (2.31) | -0.9 (2.66) | -1.1 (2.23)
  CO2, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  CO2, Week 14, n=29, 31, 33, 34, 27, 24 | -0.7 (2.02) | -0.7 (2.55) | -1.0 (2.38) | -1.1 (2.32) | -0.3 (2.31) | -1.2 (2.19)
  CO2, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  CO2, EW, n=10, 6, 3, 2, 10, 9 | -1.7 (1.57) | 0.5 (1.52) | 0.0 (3.46) | 0.0 (1.41) | -0.6 (1.65) | -0.1 (1.27)
  Glucose, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  Glucose, Week 2, n=35, 36, 35, 37, 29, 34 | 0.35 (1.147) | 0.59 (1.445) | -0.09 (1.852) | 0.05 (1.864) | -0.01 (1.168) | 0.28 (1.398)
  Glucose, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  Glucose, Week 4, n=32, 34, 33, 37, 29, 30 | 0.84 (1.750) | 0.53 (1.656) | 0.40 (3.059) | 0.42 (2.842) | 0.01 (1.299) | 0.73 (2.436)
  Glucose, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  Glucose, Week 8, n=30, 31, 32, 37, 27, 26 | 0.32 (1.571) | 0.29 (1.340) | 0.63 (2.604) | 0.35 (1.376) | 0.18 (1.505) | 0.55 (2.392)
  Glucose, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  Glucose, Week 12, n=27, 30, 32, 36, 26, 24 | 0.26 (2.223) | -0.33 (1.099) | 0.42 (2.704) | -0.02 (1.977) | -0.24 (0.966) | 0.45 (1.703)
  Glucose, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  Glucose, Week 14, n=29, 31, 33, 34, 27, 24 | 0.03 (1.708) | 0.15 (1.628) | 0.79 (2.608) | 0.12 (2.224) | -0.02 (2.104) | 0.13 (1.696)
  Glucose, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Glucose, EW, n=10, 6, 3, 2, 10, 9 | 0.00 (1.524) | 0.58 (2.185) | 0.43 (1.361) | -0.25 (0.212) | 0.35 (0.357) | 0.37 (1.665)
  Potassium, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  Potassium, Week 2, n=35, 36, 35, 37, 29, 34 | 0.07 (0.412) | 0.03 (0.322) | 0.10 (0.450) | 0.12 (0.349) | 0.20 (0.408) | -0.00 (0.306)
  Potassium, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  Potassium, Week 4, n=32, 34, 33, 37, 29, 30 | 0.07 (0.382) | 0.09 (0.370) | 0.05 (0.281) | -0.01 (0.307) | 0.13 (0.480) | 0.01 (0.380)
  Potassium, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  Potassium, Week 8, n=30, 31, 32, 37, 27, 26 | 0.10 (0.365) | 0.09 (0.576) | 0.06 (0.312) | -0.04 (0.302) | 0.05 (0.377) | 0.10 (0.600)
  Potassium, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  Potassium, Week 12, n=27, 30, 32, 36, 26, 24 | -0.07 (0.321) | 0.02 (0.228) | 0.13 (0.395) | 0.00 (0.359) | 0.02 (0.376) | 0.02 (0.298)
  Potassium, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  Potassium, Week 14, n=29, 31, 33, 34, 27, 24 | -0.01 (0.274) | 0.02 (0.268) | 0.05 (0.361) | -0.06 (0.319) | -0.01 (0.372) | 0.01 (0.372)
  Potassium, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Potassium, EW, n=10, 6, 3, 2, 10, 9 | -0.05 (0.217) | -0.02 (0.605) | 0.23 (0.493) | 0.35 (0.071) | -0.15 (0.357) | -0.08 (0.291)
  Sodium, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  Sodium, Week 2, n=35, 36, 35, 37, 29, 34 | -0.7 (2.19) | -0.2 (2.04) | -0.2 (2.13) | -0.6 (2.09) | -0.0 (2.21) | -0.5 (1.94)
  Sodium, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  Sodium, Week 4, n=32, 34, 33, 37, 29, 30 | -0.6 (1.52) | -0.1 (1.81) | -1.1 (2.28) | -0.8 (2.07) | 0.1 (2.47) | -1.2 (2.06)
  Sodium, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  Sodium, Week 8, n=30, 31, 32, 37, 27, 26 | -0.3 (1.86) | -0.2 (1.93) | -0.9 (2.01) | -0.2 (2.25) | -1.1 (2.21) | -0.8 (2.43)
  Sodium, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  Sodium, Week 12, n=27, 30, 32, 36, 26, 24 | -0.6 (2.75) | 0.1 (1.93) | -0.3 (2.43) | -0.5 (1.90) | -0.2 (2.60) | -1.2 (2.08)
  Sodium, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  Sodium, Week 14, n=29, 31, 33, 34, 27, 24 | -0.3 (2.17) | -0.2 (1.51) | -0.6 (2.18) | -0.7 (2.29) | -0.8 (2.33) | -1.0 (2.30)
  Sodium, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Sodium, EW, n=10, 6, 3, 2, 10, 9 | -1.4 (2.17) | -0.5 (1.52) | -1.0 (2.65) | 1.0 (1.41) | -0.8 (2.15) | -2.0 (2.06)
  Urea, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  Urea, Week 2, n=35, 36, 35, 37, 29, 34 | 0.17 (1.317) | 0.44 (2.242) | 0.06 (1.193) | 0.38 (1.187) | -0.09 (1.044) | 0.10 (1.347)
  Urea, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  Urea, Week 4, n=32, 34, 33, 37, 29, 30 | -0.23 (0.907) | 0.41 (1.469) | 0.05 (1.195) | 0.36 (0.991) | -0.19 (1.198) | 0.28 (1.501)
  Urea, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  Urea, Week 8, n=30, 31, 32, 37, 27, 26 | -0.07 (1.158) | -0.13 (1.049) | -0.45 (1.310) | 0.32 (0.876) | -0.22 (1.022) | -0.13 (1.179)
  Urea, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  Urea, Week 12, n=27, 30, 32, 36, 26, 24 | -0.17 (0.888) | 0.28 (1.201) | -0.27 (1.344) | 0.43 (1.220) | -0.19 (0.861) | -0.15 (1.485)
  Urea, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  Urea, Week 14, n=29, 31, 33, 34, 27, 24 | -0.10 (1.105) | 0.55 (1.485) | -0.08 (1.442) | 0.07 (1.303) | 0.35 (1.199) | -0.15 (1.272)
  Urea, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Urea, EW, n=10, 6, 3, 2, 10, 9 | 0.25 (1.007) | -0.83 (0.983) | 1.83 (3.884) | 0.00 (1.414) | -0.05 (1.012) | 0.28 (1.460)

18. Secondary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets and Leukocyte Count
Description: Blood samples were collected for the evaluation of change in levels of basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelets and leukocyte count from Baseline throughout the study. Baseline was defined as the latest assessment (including unscheduled visits) prior to the first dose and change from Baseline was defined as the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Giga unit/liter (GI/L)
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
Giga unit/liter (GI/L)
  Basophils, Week 2, n=35, 35, 36, 37, 29, 35: number analyzed (Participants) | 35 | 35 | 36 | 37 | 29 | 35
  Basophils, Week 2, n=35, 35, 36, 37, 29, 35 | 0.004 (0.0213) | -0.005 (0.0167) | -0.005 (0.0178) | 0.006 (0.0243) | 0.003 (0.0248) | 0.003 (0.0172)
  Basophils, Week 4, n=31, 34, 35, 37, 29, 31: number analyzed (Participants) | 31 | 34 | 35 | 37 | 29 | 31
  Basophils, Week 4, n=31, 34, 35, 37, 29, 31 | 0.003 (0.0176) | -0.002 (0.0285) | -0.002 (0.0166) | -0.003 (0.0184) | 0.002 (0.0175) | -0.000 (0.0143)
  Basophils, Week 8, n=30, 30, 32, 37, 27, 26: number analyzed (Participants) | 30 | 30 | 32 | 37 | 27 | 26
  Basophils, Week 8, n=30, 30, 32, 37, 27, 26 | -0.001 (0.0167) | -0.001 (0.0181) | -0.004 (0.0150) | -0.002 (0.0195) | 0.002 (0.0233) | -0.008 (0.0145)
  Basophils, Week 12, n=27, 30, 31, 36, 26, 25: number analyzed (Participants) | 27 | 30 | 31 | 36 | 26 | 25
  Basophils, Week 12, n=27, 30, 31, 36, 26, 25 | -0.003 (0.0151) | 0.004 (0.0233) | -0.007 (0.0170) | 0.000 (0.0161) | 0.006 (0.0250) | -0.003 (0.0151)
  Basophils, Week 14, n=29, 30, 33, 34, 27, 23: number analyzed (Participants) | 29 | 30 | 33 | 34 | 27 | 23
  Basophils, Week 14, n=29, 30, 33, 34, 27, 23 | -0.003 (0.0176) | -0.003 (0.0184) | -0.003 (0.0188) | 0.002 (0.0250) | -0.001 (0.0188) | -0.001 (0.0216)
  Basophils, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Basophils, EW, n=10, 6, 3, 2, 10, 9 | -0.001 (0.0179) | -0.017 (0.0294) | -0.010 (0.0100) | 0.000 (0.000) | -0.005 (0.0151) | 0.012 (0.0217)
  Eosinophils, Week 2, n=35, 35, 36, 37, 29, 35: number analyzed (Participants) | 35 | 35 | 36 | 37 | 29 | 35
  Eosinophils, Week 2, n=35, 35, 36, 37, 29, 35 | 0.021 (0.1157) | 0.043 (0.1356) | -0.017 (0.1857) | 0.011 (0.0972) | -0.021 (0.1363) | -0.015 (0.1295)
  Eosinophils, Week 4, n=31, 34, 35, 37, 29, 31: number analyzed (Participants) | 31 | 34 | 35 | 37 | 29 | 31
  Eosinophils, Week 4, n=31, 34, 35, 37, 29, 31 | 0.019 (0.1380) | 0.034 (0.1371) | -0.005 (0.1554) | 0.005 (0.0954) | -0.019 (0.1205) | -0.005 (0.1522)
  Eosinophils, Week 8, n=30, 30, 32, 37, 27, 26: number analyzed (Participants) | 30 | 30 | 32 | 37 | 27 | 26
  Eosinophils, Week 8, n=30, 30, 32, 37, 27, 26 | 0.012 (0.1134) | 0.024 (0.1015) | -0.008 (0.1495) | 0.037 (0.1001) | -0.008 (0.1142) | -0.048 (0.1258)
  Eosinophils, Week 12, n=27, 30, 31, 36, 26, 25: number analyzed (Participants) | 27 | 30 | 31 | 36 | 26 | 25
  Eosinophils, Week 12, n=27, 30, 31, 36, 26, 25 | 0.047 (0.2302) | 0.000 (0.1002) | -0.032 (0.1714) | 0.026 (0.0934) | 0.001 (0.1375) | -0.027 (0.1322)
  Eosinophils, Week 14, n=29, 30, 33, 34, 27, 23: number analyzed (Participants) | 29 | 30 | 33 | 34 | 27 | 23
  Eosinophils, Week 14, n=29, 30, 33, 34, 27, 23 | 0.033 (0.1084) | 0.004 (0.0979) | -0.011 (0.2186) | 0.002 (0.1053) | 0.004 (0.1469) | -0.053 (0.1867)
  Eosinophils, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Eosinophils, EW, n=10, 6, 3, 2, 10, 9 | 0.029 (0.0841) | 0.090 (0.1563) | -0.233 (0.3955) | 0.095 (0.0071) | 0.053 (0.2675) | -0.047 (0.1775)
  Lymphocytes, Week 2, n=35, 35, 36, 37, 29, 35: number analyzed (Participants) | 35 | 35 | 36 | 37 | 29 | 35
  Lymphocytes, Week 2, n=35, 35, 36, 37, 29, 35 | 0.100 (0.4690) | -0.002 (0.3827) | 0.097 (0.3995) | 0.145 (0.3966) | -0.138 (0.4764) | -0.018 (0.4774)
  Lymphocytes, Week 4, n=31, 34, 35, 37, 29, 31: number analyzed (Participants) | 31 | 34 | 35 | 37 | 29 | 31
  Lymphocytes, Week 4, n=31, 34, 35, 37, 29, 31 | -0.083 (0.6201) | -0.044 (0.4101) | 0.041 (0.3875) | 0.228 (0.5664) | -0.142 (0.4421) | -0.077 (0.4524)
  Lymphocytes, Week 8, n=30, 30, 32, 37, 27, 26: number analyzed (Participants) | 30 | 30 | 32 | 37 | 27 | 26
  Lymphocytes, Week 8, n=30, 30, 32, 37, 27, 26 | 0.048 (0.5656) | -0.009 (0.3778) | -0.048 (0.4379) | 0.075 (0.5255) | -0.110 (0.6406) | 0.032 (0.4913)
  Lymphocytes, Week 12, n=27, 30, 31, 36, 26, 25: number analyzed (Participants) | 27 | 30 | 31 | 36 | 26 | 25
  Lymphocytes, Week 12, n=27, 30, 31, 36, 26, 25 | 0.050 (0.6354) | 0.052 (0.4589) | 0.120 (0.5800) | 0.148 (0.4774) | -0.110 (0.6003) | -0.145 (0.4177)
  Lymphocytes, Week 14, n=29, 30, 33, 34, 27, 23: number analyzed (Participants) | 29 | 30 | 33 | 34 | 27 | 23
  Lymphocytes, Week 14, n=29, 30, 33, 34, 27, 23 | 0.261 (0.9065) | 0.021 (0.6397) | 0.075 (0.5712) | 0.174 (0.7327) | -0.031 (0.6712) | 0.109 (0.4985)
  Lymphocytes, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Lymphocytes, EW, n=10, 6, 3, 2, 10, 9 | -0.164 (0.6069) | -0.078 (0.3542) | -0.113 (0.3502) | -0.185 (0.1061) | 0.032 (0.2862) | 0.246 (0.4375)
  Monocytes, Week 2, n=35, 35, 36, 37, 29, 35: number analyzed (Participants) | 35 | 35 | 36 | 37 | 29 | 35
  Monocytes, Week 2, n=35, 35, 36, 37, 29, 35 | 0.029 (0.1833) | -0.061 (0.1055) | 0.012 (0.1314) | -0.035 (0.1117) | -0.007 (0.1583) | -0.013 (0.1083)
  Monocytes, Week 4, n=31, 34, 35, 37, 29, 31: number analyzed (Participants) | 31 | 34 | 35 | 37 | 29 | 31
  Monocytes, Week 4, n=31, 34, 35, 37, 29, 31 | -0.017 (0.1241) | -0.014 (0.1706) | -0.014 (0.1226) | -0.049 (0.1119) | -0.032 (0.1972) | -0.011 (0.1464)
  Monocytes, Week 8, n=30, 30, 32, 37, 27, 26: number analyzed (Participants) | 30 | 30 | 32 | 37 | 27 | 26
  Monocytes, Week 8, n=30, 30, 32, 37, 27, 26 | 0.034 (0.1468) | -0.071 (0.1258) | -0.036 (0.1252) | -0.043 (0.1579) | -0.048 (0.1692) | -0.025 (0.1770)
  Monocytes, Week 12, n=27, 30, 31, 36, 26, 25: number analyzed (Participants) | 27 | 30 | 31 | 36 | 26 | 25
  Monocytes, Week 12, n=27, 30, 31, 36, 26, 25 | -0.002 (0.1173) | -0.050 (0.1036) | -0.055 (0.1399) | -0.043 (0.1578) | -0.015 (0.1964) | -0.026 (0.1323)
  Monocytes, Week 14, n=29, 30, 33, 34, 27, 23: number analyzed (Participants) | 29 | 30 | 33 | 34 | 27 | 23
  Monocytes, Week 14, n=29, 30, 33, 34, 27, 23 | 0.031 (0.1418) | -0.009 (0.1341) | -0.057 (0.1378) | -0.054 (0.1609) | -0.025 (0.2130) | -0.017 (0.1202)
  Monocytes, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Monocytes, EW, n=10, 6, 3, 2, 10, 9 | 0.046 (0.1959) | -0.015 (0.1299) | -0.243 (0.2593) | -0.045 (0.1061) | 0.006 (0.1179) | -0.084 (0.2625)
  Neutrophils, Week 2, n=35, 35, 36, 37, 29, 35: number analyzed (Participants) | 35 | 35 | 36 | 37 | 29 | 35
  Neutrophils, Week 2, n=35, 35, 36, 37, 29, 35 | 0.355 (1.7248) | 0.310 (1.3852) | 0.341 (1.3914) | 0.009 (1.3107) | -0.058 (1.8094) | 0.107 (1.1007)
  Neutrophils, Week 4, n=31, 34, 35, 37, 29, 31: number analyzed (Participants) | 31 | 34 | 35 | 37 | 29 | 31
  Neutrophils, Week 4, n=31, 34, 35, 37, 29, 31 | 0.215 (1.5812) | 0.139 (1.6995) | 0.291 (1.2083) | 0.267 (1.3310) | 0.049 (1.7831) | 0.059 (1.0011)
  Neutrophils, Week 8, n=30, 30, 32, 37, 27, 26: number analyzed (Participants) | 30 | 30 | 32 | 37 | 27 | 26
  Neutrophils, Week 8, n=30, 30, 32, 37, 27, 26 | 0.402 (1.1117) | 0.140 (1.1014) | -0.049 (1.4021) | -0.075 (1.4243) | -0.181 (1.4359) | 0.285 (1.3332)
  Neutrophils, Week 12, n=27, 30, 31, 36, 26, 25: number analyzed (Participants) | 27 | 30 | 31 | 36 | 26 | 25
  Neutrophils, Week 12, n=27, 30, 31, 36, 26, 25 | 0.277 (1.0785) | 0.099 (1.3124) | -0.015 (1.4752) | -0.008 (1.4329) | 0.043 (1.3470) | 0.008 (1.0432)
  Neutrophils, Week 14, n=29, 30, 33, 34, 27, 23: number analyzed (Participants) | 29 | 30 | 33 | 34 | 27 | 23
  Neutrophils, Week 14, n=29, 30, 33, 34, 27, 23 | 0.158 (1.0726) | 0.519 (1.4793) | -0.053 (1.0828) | -0.225 (1.5059) | 0.267 (2.2299) | -0.052 (0.8640)
  Neutrophils, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Neutrophils, EW, n=10, 6, 3, 2, 10, 9 | 0.307 (1.1539) | -0.305 (1.3530) | 2.727 (3.3561) | -0.735 (0.2899) | -0.285 (1.2029) | -0.019 (0.9601)
  Platelets, Week 2, n=35, 35, 36, 37, 29, 35: number analyzed (Participants) | 35 | 35 | 36 | 37 | 29 | 35
  Platelets, Week 2, n=35, 35, 36, 37, 29, 35 | -0.3 (36.30) | 5.4 (40.50) | 2.3 (26.06) | -5.6 (47.57) | 0.5 (29.07) | -6.1 (23.70)
  Platelets, Week 4, n=32, 34, 35, 37, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 37 | 29 | 31
  Platelets, Week 4, n=32, 34, 35, 37, 29, 31 | -12.3 (39.49) | -4.1 (26.64) | 1.9 (26.97) | -1.0 (38.16) | 2.6 (26.00) | -0.7 (28.81)
  Platelets, Week 8, n=30, 31, 32, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 38 | 27 | 26
  Platelets, Week 8, n=30, 31, 32, 38, 27, 26 | -6.8 (34.57) | -1.0 (23.87) | -1.8 (25.81) | -11.5 (50.01) | 0.2 (28.94) | -1.5 (23.61)
  Platelets, Week 12, n=27, 30, 31, 36, 26, 25: number analyzed (Participants) | 27 | 30 | 31 | 36 | 26 | 25
  Platelets, Week 12, n=27, 30, 31, 36, 26, 25 | -10.3 (35.25) | -7.9 (24.25) | -4.9 (26.54) | -15.7 (38.39) | -5.5 (38.31) | -8.9 (26.72)
  Platelets, Week 14, n=29, 30, 33, 34, 27, 23: number analyzed (Participants) | 29 | 30 | 33 | 34 | 27 | 23
  Platelets, Week 14, n=29, 30, 33, 34, 27, 23 | -2.9 (18.68) | -9.6 (29.12) | -2.9 (20.21) | -18.5 (41.03) | -1.7 (37.21) | 1.2 (18.69)
  Platelets, EW, n=10, 5, 3, 2, 9, 9: number analyzed (Participants) | 10 | 5 | 3 | 2 | 9 | 9
  Platelets, EW, n=10, 5, 3, 2, 9, 9 | -2.1 (27.63) | -7.6 (13.89) | 37.0 (37.80) | -30.5 (48.79) | 1.6 (22.36) | 23.1 (25.21)
  Leukocytes, Week 2, n=35, 35, 36, 37, 29, 35: number analyzed (Participants) | 35 | 35 | 36 | 37 | 29 | 35
  Leukocytes, Week 2, n=35, 35, 36, 37, 29, 35 | 0.50 (1.834) | 0.28 (1.381) | 0.42 (1.686) | 0.12 (1.391) | -0.21 (1.892) | 0.08 (1.166)
  Leukocytes, Week 4, n=31, 34, 35, 37, 29, 31: number analyzed (Participants) | 31 | 34 | 35 | 37 | 29 | 31
  Leukocytes, Week 4, n=31, 34, 35, 37, 29, 31 | 0.13 (1.972) | 0.12 (1.748) | 0.31 (1.374) | 0.44 (1.398) | -0.14 (1.798) | -0.03 (1.059)
  Leukocytes, Week 8, n=30, 30, 32, 37, 27, 26: number analyzed (Participants) | 30 | 30 | 32 | 37 | 27 | 26
  Leukocytes, Week 8, n=30, 30, 32, 37, 27, 26 | 0.49 (1.272) | 0.08 (1.167) | -0.14 (1.516) | -0.02 (1.604) | -0.35 (1.392) | 0.23 (1.527)
  Leukocytes, Week 12, n=27, 30, 31, 36, 26, 25: number analyzed (Participants) | 27 | 30 | 31 | 36 | 26 | 25
  Leukocytes, Week 12, n=27, 30, 31, 36, 26, 25 | 0.36 (1.439) | 0.12 (1.359) | 0.02 (1.460) | 0.10 (1.538) | -0.07 (1.301) | -0.19 (1.221)
  Leukocytes, Week 14, n=29, 30, 33, 34, 27, 23: number analyzed (Participants) | 29 | 30 | 33 | 34 | 27 | 23
  Leukocytes, Week 14, n=29, 30, 33, 34, 27, 23 | 0.47 (1.472) | 0.54 (1.757) | -0.05 (1.256) | -0.11 (1.380) | 0.22 (2.172) | -0.00 (1.207)
  Leukocytes, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Leukocytes, EW, n=10, 6, 3, 2, 10, 9 | 0.21 (1.066) | -0.35 (1.395) | 2.13 (2.940) | -0.85 (0.354) | -0.21 (1.260) | 0.10 (0.505)

19. Secondary Outcome: Change From Baseline in Hematocrit Levels
Description: Blood samples were collected for the evaluation of change in hematocrit levels from Baseline throughout the study. Baseline was defined as the latest assessment (including unscheduled visits) prior to the first dose and change from Baseline was defined as the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
Proportion of red blood cells in blood
  Week 2, n=35, 35, 36, 37, 29, 35: number analyzed (Participants) | 35 | 35 | 36 | 37 | 29 | 35
  Week 2, n=35, 35, 36, 37, 29, 35 | 0.0029 (0.0198) | -0.0036 (0.0243) | -0.0002 (0.0251) | -0.0038 (0.0193) | -0.0063 (0.0243) | 0.0011 (0.0217)
  Week 4, n=32, 34, 35, 37, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 37 | 29 | 31
  Week 4, n=32, 34, 35, 37, 29, 31 | 0.0007 (0.0227) | -0.0049 (0.0238) | 0.0058 (0.0283) | -0.0008 (0.0269) | 0.0028 (0.0291) | 0.0054 (0.0239)
  Week 8, n=30, 31, 32, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 38 | 27 | 26
  Week 8, n=30, 31, 32, 38, 27, 26 | 0.0020 (0.0273) | 0.0047 (0.0274) | -0.0004 (0.0288) | -0.0036 (0.0342) | 0.0084 (0.0284) | 0.0092 (0.0319)
  Week 12, n=27, 30, 31, 36, 26, 25: number analyzed (Participants) | 27 | 30 | 31 | 36 | 26 | 25
  Week 12, n=27, 30, 31, 36, 26, 25 | 0.0045 (0.0238) | 0.0059 (0.0275) | 0.0059 (0.0235) | -0.0013 (0.0202) | 0.0045 (0.0225) | 0.0084 (0.0286)
  Week 14, n=29, 30, 33, 34, 27, 23: number analyzed (Participants) | 29 | 30 | 33 | 34 | 27 | 23
  Week 14, n=29, 30, 33, 34, 27, 23 | 0.0017 (0.0259) | -0.0010 (0.0274) | 0.0021 (0.0288) | -0.0120 (0.0348) | -0.0021 (0.0336) | 0.0035 (0.0186)
  EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  EW, n=10, 6, 3, 2, 10, 9 | 0.0014 (0.0185) | -0.0273 (0.0221) | -0.0093 (0.0134) | -0.0050 (0.0014) | -0.0017 (0.0161) | 0.0014 (0.0268)

20. Secondary Outcome: Change From Baseline in Hemoglobin (Hgb) Level and Erythrocyte Mean Corpuscular Hgb Concentration (MCHC)
Description: Blood samples were collected for the evaluation of change in Hgb levels and MCHC from Baseline throughout the study. Baseline was defined as the latest assessment (including unscheduled visits) prior to the first dose and change from Baseline was defined as the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
G/L
  Hgb, Week 2, n=35, 35, 36, 37, 29, 35: number analyzed (Participants) | 35 | 35 | 36 | 37 | 29 | 35
  Hgb, Week 2, n=35, 35, 36, 37, 29, 35 | 0.3 (5.84) | -1.6 (6.98) | -1.4 (7.51) | -0.6 (6.29) | -1.3 (7.79) | 0.1 (6.18)
  Hgb, Week 4, n=32, 34, 35, 37, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 37 | 29 | 31
  Hgb, Week 4, n=32, 34, 35, 37, 29, 31 | -1.0 (6.02) | -2.5 (5.86) | 0.3 (8.74) | -0.1 (8.82) | -0.7 (8.77) | 1.0 (5.68)
  Hgb, Week 8, n=30, 31, 32, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 38 | 27 | 26
  Hgb, Week 8, n=30, 31, 32, 38, 27, 26 | -1.8 (6.18) | 0.1 (6.78) | -2.8 (9.06) | -2.1 (9.17) | 1.0 (8.82) | 1.2 (7.73)
  Hgb, Week 12, n=27, 30, 31, 36, 26, 25: number analyzed (Participants) | 27 | 30 | 31 | 36 | 26 | 25
  Hgb, Week 12, n=27, 30, 31, 36, 26, 25 | -1.3 (5.74) | -0.8 (6.86) | -1.9 (8.76) | -2.4 (5.94) | -1.0 (7.65) | 0.2 (6.27)
  Hgb, Week 14, n=29, 30, 33, 34, 27, 23: number analyzed (Participants) | 29 | 30 | 33 | 34 | 27 | 23
  Hgb, Week 14, n=29, 30, 33, 34, 27, 23 | -1.9 (7.85) | -2.7 (7.54) | -2.6 (8.64) | -5.0 (10.24) | -2.8 (8.82) | -1.6 (5.94)
  Hgb, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Hgb, EW, n=10, 6, 3, 2, 10, 9 | 0.0 (7.26) | -7.8 (8.73) | -5.7 (3.79) | -1.5 (0.71) | -2.3 (4.99) | -0.1 (6.13)
  MCHC, Week 2, n=35, 35, 36, 37, 29, 35: number analyzed (Participants) | 35 | 35 | 36 | 37 | 29 | 35
  MCHC, Week 2, n=35, 35, 36, 37, 29, 35 | -1.5 (8.77) | -1.3 (9.44) | -3.0 (10.32) | 1.0 (7.15) | 0.9 (7.99) | -0.5 (7.10)
  MCHC, Week 4, n=32, 34, 35, 37, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 37 | 29 | 31
  MCHC, Week 4, n=32, 34, 35, 37, 29, 31 | -3.1 (11.45) | -2.1 (9.88) | -3.6 (10.60) | 0.4 (8.36) | -3.8 (9.19) | -1.6 (10.02)
  MCHC, Week 8, n=30, 31, 32, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 38 | 27 | 26
  MCHC, Week 8, n=30, 31, 32, 38, 27, 26 | -5.4 (11.25) | -3.2 (12.76) | -5.9 (13.41) | -2.3 (11.29) | -4.4 (10.65) | -3.8 (11.40)
  MCHC, Week 12, n=27, 30, 31, 36, 26, 25: number analyzed (Participants) | 27 | 30 | 31 | 36 | 26 | 25
  MCHC, Week 12, n=27, 30, 31, 36, 26, 25 | -6.1 (12.65) | -6.1 (11.25) | -8.6 (11.49) | -4.8 (10.39) | -5.9 (10.14) | -5.0 (10.74)
  MCHC, Week 14, n=29, 30, 33, 34, 27, 23: number analyzed (Participants) | 29 | 30 | 33 | 34 | 27 | 23
  MCHC, Week 14, n=29, 30, 33, 34, 27, 23 | -5.4 (8.55) | -5.5 (9.15) | -7.4 (10.74) | -2.7 (9.40) | -5.3 (9.27) | -5.9 (9.79)
  MCHC, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  MCHC, EW, n=10, 6, 3, 2, 10, 9 | -1.1 (11.57) | 1.5 (8.50) | -6.3 (9.07) | 0.0 (0.00) | -4.1 (4.12) | -1.3 (9.10)

21. Secondary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular Hemoglobin Level
Description: Blood samples were collected for the evaluation of change in erythrocyte mean corpuscular hemoglobin level from Baseline throughout the study. Baseline was defined as the latest assessment (including unscheduled visits) prior to the first dose and change from Baseline was defined as the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Picogram (pg)
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
Picogram (pg)
  Week 2, n=35, 35, 36, 37, 29, 35: number analyzed (Participants) | 35 | 35 | 36 | 37 | 29 | 35
  Week 2, n=35, 35, 36, 37, 29, 35 | 0.10 (0.493) | 0.05 (0.408) | -0.08 (0.590) | 0.11 (0.733) | -0.10 (1.519) | -0.01 (0.605)
  Week 4, n=32, 34, 35, 37, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 37 | 29 | 31
  Week 4, n=32, 34, 35, 37, 29, 31 | 0.01 (0.562) | -0.06 (0.517) | -0.19 (0.750) | 0.08 (0.774) | -0.15 (1.257) | -0.15 (0.863)
  Week 8, n=30, 31, 32, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 38 | 27 | 26
  Week 8, n=30, 31, 32, 38, 27, 26 | 0.13 (0.608) | 0.31 (2.220) | -0.20 (0.805) | -0.04 (0.803) | -0.13 (1.286) | -0.09 (0.753)
  Week 12, n=27, 30, 31, 36, 26, 25: number analyzed (Participants) | 27 | 30 | 31 | 36 | 26 | 25
  Week 12, n=27, 30, 31, 36, 26, 25 | 0.20 (0.804) | -0.07 (0.672) | -0.15 (0.532) | -0.00 (0.837) | -0.30 (1.265) | -0.21 (0.764)
  Week 14, n=29, 30, 33, 34, 27, 23: number analyzed (Participants) | 29 | 30 | 33 | 34 | 27 | 23
  Week 14, n=29, 30, 33, 34, 27, 23 | 0.39 (0.671) | 0.02 (0.406) | -0.19 (0.685) | 0.07 (0.785) | -0.23 (1.396) | 0.01 (0.557)
  EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  EW, n=10, 6, 3, 2, 10, 9 | 0.10 (0.371) | 0.15 (0.734) | -0.50 (0.520) | 0.05 (0.071) | -0.02 (0.181) | -0.12 (0.533)

22. Secondary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular Volume
Description: Blood samples were collected for the evaluation of change in erythrocyte mean corpuscular volume from Baseline throughout the study. Baseline was defined as the latest assessment (including unscheduled visits) prior to the first dose and change from Baseline was defined as the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Femtoliter (fL)
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
Femtoliter (fL)
  Week 2, n=35, 35, 36, 37, 29, 35: number analyzed (Participants) | 35 | 35 | 36 | 37 | 29 | 35
  Week 2, n=35, 35, 36, 37, 29, 35 | 0.7 (2.38) | 0.6 (2.07) | 0.6 (2.39) | 0.1 (2.11) | -0.5 (4.05) | 0.2 (1.96)
  Week 4, n=32, 34, 35, 37, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 37 | 29 | 31
  Week 4, n=32, 34, 35, 37, 29, 31 | 0.8 (2.21) | 0.4 (1.94) | 0.4 (2.65) | 0.2 (2.39) | 0.7 (3.73) | 0.0 (3.10)
  Week 8, n=30, 31, 32, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 38 | 27 | 26
  Week 8, n=30, 31, 32, 38, 27, 26 | 2.0 (2.39) | 2.0 (5.05) | 1.1 (3.57) | 0.6 (3.41) | 0.9 (3.80) | 0.9 (3.10)
  Week 12, n=27, 30, 31, 36, 26, 25: number analyzed (Participants) | 27 | 30 | 31 | 36 | 26 | 25
  Week 12, n=27, 30, 31, 36, 26, 25 | 2.4 (2.27) | 1.6 (1.94) | 1.9 (3.41) | 1.4 (3.72) | 0.8 (3.98) | 0.9 (2.93)
  Week 14, n=29, 30, 33, 34, 27, 23: number analyzed (Participants) | 29 | 30 | 33 | 34 | 27 | 23
  Week 14, n=29, 30, 33, 34, 27, 23 | 2.7 (2.87) | 1.6 (2.08) | 1.5 (3.04) | 0.9 (3.27) | 0.9 (3.95) | 1.9 (2.36)
  EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  EW, n=10, 6, 3, 2, 10, 9 | 0.6 (3.41) | 0.0 (2.19) | -0.3 (0.58) | -0.5 (0.71) | 1.1 (1.60) | 0.1 (2.42)

23. Secondary Outcome: Change From Baseline in Erythrocyte Count
Description: Blood samples were collected for the evaluation of change in erythrocyte count from Baseline throughout the study. Baseline was defined as the latest assessment (including unscheduled visits) prior to the first dose and change from Baseline was defined as the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Tetra unit/L (TI/L)
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
Tetra unit/L (TI/L)
  Week 2, n=35, 35, 36, 37, 29, 35: number analyzed (Participants) | 35 | 35 | 36 | 37 | 29 | 35
  Week 2, n=35, 35, 36, 37, 29, 35 | -0.01 (0.180) | -0.06 (0.243) | -0.04 (0.315) | -0.05 (0.210) | -0.03 (0.363) | 0.01 (0.269)
  Week 4, n=32, 34, 35, 37, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 37 | 29 | 31
  Week 4, n=32, 34, 35, 37, 29, 31 | -0.03 (0.213) | -0.06 (0.220) | 0.02 (0.358) | -0.01 (0.269) | 0.01 (0.421) | 0.05 (0.294)
  Week 8, n=30, 31, 32, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 38 | 27 | 26
  Week 8, n=30, 31, 32, 38, 27, 26 | -0.09 (0.273) | -0.05 (0.468) | -0.07 (0.306) | -0.07 (0.257) | 0.06 (0.356) | 0.03 (0.317)
  Week 12, n=27, 30, 31, 36, 26, 25: number analyzed (Participants) | 27 | 30 | 31 | 36 | 26 | 25
  Week 12, n=27, 30, 31, 36, 26, 25 | -0.07 (0.237) | 0.00 (0.257) | -0.05 (0.356) | -0.08 (0.228) | 0.00 (0.328) | 0.04 (0.229)
  Week 14, n=29, 30, 33, 34, 27, 23: number analyzed (Participants) | 29 | 30 | 33 | 34 | 27 | 23
  Week 14, n=29, 30, 33, 34, 27, 23 | -0.13 (0.334) | -0.09 (0.252) | -0.07 (0.374) | -0.18 (0.343) | -0.06 (0.370) | -0.07 (0.194)
  EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  EW, n=10, 6, 3, 2, 10, 9 | -0.03 (0.250) | -0.30 (0.268) | -0.13 (0.153) | -0.10 (0.000) | -0.07 (0.200) | 0.00 (0.212)

24. Secondary Outcome: Number of Participants With Chemistry Data of Potential Clinical Importance
Description: Blood samples were collected for the evaluation of clinical chemistry parameters including alk phos, ALT, AST, bil, calcium, CO2, creatinine, glucose and potassium. The number of participants with chemistry data of potential clinical importance for the mentioned parameters was presented. Baseline was defined as the latest assessment (including unscheduled visits) prior to the first dose. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Up to Week 14
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
Participants
  Alk. Phos, Baseline, n=38, 38, 38, 38, 37, 38 | 0 | 0 | 0 | 0 | 0 | 0
  Alk. Phos, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  Alk. Phos, Week 2, n=35, 36, 35, 37, 29, 34 | 0 | 0 | 0 | 0 | 0 | 0
  Alk. Phos, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  Alk. Phos, Week 4, n=32, 34, 33, 37, 29, 30 | 0 | 0 | 1 | 0 | 0 | 0
  Alk. Phos, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  Alk. Phos, Week 8, n=30, 31, 32, 37, 27, 26 | 0 | 0 | 0 | 0 | 0 | 0
  Alk. Phos, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  Alk. Phos, Week 12, n=27, 30, 32, 36, 26, 24 | 0 | 0 | 0 | 0 | 0 | 0
  Alk. Phos, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  Alk. Phos, Week 14, n=29, 31, 33, 34, 27, 24 | 0 | 0 | 0 | 0 | 0 | 0
  Alk. Phos, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Alk. Phos, EW, n=10, 6, 3, 2, 10, 9 | 0 | 0 | 0 | 0 | 0 | 0
  Alk. Phos,post-screen(PS),n=38, 37, 37, 38, 36, 36: number analyzed (Participants) | 38 | 37 | 37 | 38 | 36 | 36
  Alk. Phos,post-screen(PS),n=38, 37, 37, 38, 36, 36 | 0 | 0 | 1 | 0 | 0 | 0
  ALT, Baseline, n=38, 38, 38, 38, 37, 38 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  ALT, Week 2, n=35, 36, 35, 37, 29, 34 | 0 | 0 | 0 | 0 | 0 | 1
  ALT, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  ALT, Week 4, n=32, 34, 33, 37, 29, 30 | 1 | 0 | 0 | 0 | 0 | 1
  ALT, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  ALT, Week 8, n=30, 31, 32, 37, 27, 26 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  ALT, Week 12, n=27, 30, 32, 36, 26, 24 | 0 | 0 | 0 | 0 | 0 | 1
  ALT, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  ALT, Week 14, n=29, 31, 33, 34, 27, 24 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  ALT, EW, n=10, 6, 3, 2, 10, 9 | 0 | 0 | 0 | 0 | 0 | 0
  ALT, PS, n=38, 37, 37, 38, 36, 36: number analyzed (Participants) | 38 | 37 | 37 | 38 | 36 | 36
  ALT, PS, n=38, 37, 37, 38, 36, 36 | 1 | 0 | 0 | 0 | 0 | 2
  AST, Baseline, n=38, 38, 38, 38, 37, 38 | 0 | 1 | 0 | 0 | 0 | 0
  AST, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  AST, Week 2, n=35, 36, 35, 37, 29, 34 | 0 | 1 | 0 | 0 | 0 | 0
  AST, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  AST, Week 4, n=32, 34, 33, 37, 29, 30 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  AST, Week 8, n=30, 31, 32, 37, 27, 26 | 0 | 1 | 0 | 0 | 0 | 0
  AST, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  AST, Week 12, n=27, 30, 32, 36, 26, 24 | 0 | 0 | 0 | 0 | 0 | 0
  AST, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  AST, Week 14, n=29, 31, 33, 34, 27, 24 | 0 | 0 | 0 | 0 | 0 | 0
  AST, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  AST, EW, n=10, 6, 3, 2, 10, 9 | 0 | 0 | 0 | 0 | 0 | 0
  AST, PS, n=38, 37, 37, 38, 36, 36: number analyzed (Participants) | 38 | 37 | 37 | 38 | 36 | 36
  AST, PS, n=38, 37, 37, 38, 36, 36 | 0 | 2 | 0 | 0 | 0 | 0
  Bil, Baseline, n=38, 38, 38, 38, 37, 38 | 0 | 0 | 0 | 0 | 0 | 1
  Bil, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  Bil, Week 2, n=35, 36, 35, 37, 29, 34 | 0 | 0 | 0 | 0 | 1 | 1
  Bil, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  Bil, Week 4, n=32, 34, 33, 37, 29, 30 | 0 | 0 | 0 | 0 | 0 | 1
  Bil, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  Bil, Week 8, n=30, 31, 32, 37, 27, 26 | 0 | 0 | 0 | 0 | 0 | 1
  Bil, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  Bil, Week 12, n=27, 30, 32, 36, 26, 24 | 0 | 0 | 0 | 0 | 0 | 1
  Bil, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  Bil, Week 14, n=29, 31, 33, 34, 27, 24 | 0 | 0 | 0 | 0 | 0 | 1
  Bil, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Bil, EW, n=10, 6, 3, 2, 10, 9 | 0 | 0 | 0 | 0 | 0 | 0
  Bil, PS, n=38, 37, 37, 38, 36, 36: number analyzed (Participants) | 38 | 37 | 37 | 38 | 36 | 36
  Bil, PS, n=38, 37, 37, 38, 36, 36 | 0 | 0 | 0 | 0 | 1 | 1
  Calcium, Baseline, n=38, 38, 38, 38, 37, 38 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  Calcium, Week 2, n=35, 36, 35, 37, 29, 34 | 0 | 0 | 1 | 0 | 0 | 0
  Calcium, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  Calcium, Week 4, n=32, 34, 33, 37, 29, 30 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  Calcium, Week 8, n=30, 31, 32, 37, 27, 26 | 0 | 0 | 1 | 0 | 0 | 0
  Calcium, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  Calcium, Week 12, n=27, 30, 32, 36, 26, 24 | 0 | 0 | 0 | 1 | 0 | 0
  Calcium, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  Calcium, Week 14, n=29, 31, 33, 34, 27, 24 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Calcium, EW, n=10, 6, 3, 2, 10, 9 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, PS, n=38, 37, 37, 38, 36, 36: number analyzed (Participants) | 38 | 37 | 37 | 38 | 36 | 36
  Calcium, PS, n=38, 37, 37, 38, 36, 36 | 0 | 0 | 2 | 1 | 0 | 0
  CO2, Baseline, n=38, 38, 38, 38, 37, 38 | 0 | 0 | 1 | 0 | 0 | 0
  CO2, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  CO2, Week 2, n=35, 36, 35, 37, 29, 34 | 1 | 0 | 4 | 1 | 0 | 0
  CO2, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  CO2, Week 4, n=32, 34, 33, 37, 29, 30 | 0 | 1 | 3 | 0 | 0 | 0
  CO2, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  CO2, Week 8, n=30, 31, 32, 37, 27, 26 | 1 | 1 | 1 | 0 | 0 | 0
  CO2, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  CO2, Week 12, n=27, 30, 32, 36, 26, 24 | 0 | 0 | 3 | 1 | 0 | 0
  CO2, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  CO2, Week 14, n=29, 31, 33, 34, 27, 24 | 0 | 0 | 1 | 1 | 0 | 0
  CO2, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  CO2, EW, n=10, 6, 3, 2, 10, 9 | 0 | 0 | 0 | 0 | 0 | 0
  CO2, PS, n=38, 37, 37, 38, 36, 36: number analyzed (Participants) | 38 | 37 | 37 | 38 | 36 | 36
  CO2, PS, n=38, 37, 37, 38, 36, 36 | 1 | 1 | 8 | 2 | 0 | 0
  Creatinine, Baseline, n=38, 38, 38, 38, 37, 38 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  Creatinine, Week 2, n=35, 36, 35, 37, 29, 34 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  Creatinine, Week 4, n=32, 34, 33, 37, 29, 30 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  Creatinine, Week 8, n=30, 31, 32, 37, 27, 26 | 0 | 0 | 0 | 1 | 0 | 0
  Creatinine, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  Creatinine, Week 12, n=27, 30, 32, 36, 26, 24 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  Creatinine, Week 14, n=29, 31, 33, 34, 27, 24 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Creatinine, EW, n=10, 6, 3, 2, 10, 9 | 0 | 0 | 1 | 0 | 0 | 0
  Creatinine, PS, n=38, 37, 37, 38, 36, 36: number analyzed (Participants) | 38 | 37 | 37 | 38 | 36 | 36
  Creatinine, PS, n=38, 37, 37, 38, 36, 36 | 0 | 0 | 1 | 1 | 0 | 0
  Glucose, Baseline, n=38, 38, 38, 38, 37, 38 | 0 | 4 | 5 | 2 | 5 | 1
  Glucose, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  Glucose, Week 2, n=35, 36, 35, 37, 29, 34 | 2 | 5 | 5 | 2 | 2 | 2
  Glucose, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  Glucose, Week 4, n=32, 34, 33, 37, 29, 30 | 4 | 4 | 4 | 3 | 5 | 3
  Glucose, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  Glucose, Week 8, n=30, 31, 32, 37, 27, 26 | 1 | 3 | 6 | 2 | 4 | 3
  Glucose, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  Glucose, Week 12, n=27, 30, 32, 36, 26, 24 | 3 | 3 | 7 | 4 | 2 | 2
  Glucose, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  Glucose, Week 14, n=29, 31, 33, 34, 27, 24 | 1 | 2 | 7 | 4 | 5 | 3
  Glucose, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Glucose, EW, n=10, 6, 3, 2, 10, 9 | 1 | 0 | 0 | 0 | 0 | 0
  Glucose, PS, n=38, 37, 37, 38, 36, 36: number analyzed (Participants) | 38 | 37 | 37 | 38 | 36 | 36
  Glucose, PS, n=38, 37, 37, 38, 36, 36 | 7 | 7 | 7 | 8 | 6 | 9
  Potassium, Baseline, n=38, 38, 38, 38, 37, 38 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, Week 2, n=35, 36, 35, 37, 29, 34: number analyzed (Participants) | 35 | 36 | 35 | 37 | 29 | 34
  Potassium, Week 2, n=35, 36, 35, 37, 29, 34 | 0 | 0 | 1 | 0 | 1 | 0
  Potassium, Week 4, n=32, 34, 33, 37, 29, 30: number analyzed (Participants) | 32 | 34 | 33 | 37 | 29 | 30
  Potassium, Week 4, n=32, 34, 33, 37, 29, 30 | 1 | 0 | 0 | 0 | 2 | 1
  Potassium, Week 8, n=30, 31, 32, 37, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 37 | 27 | 26
  Potassium, Week 8, n=30, 31, 32, 37, 27, 26 | 0 | 1 | 0 | 0 | 0 | 2
  Potassium, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  Potassium, Week 12, n=27, 30, 32, 36, 26, 24 | 0 | 0 | 1 | 0 | 0 | 0
  Potassium, Week 14, n=29, 31, 33, 34, 27, 24: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 24
  Potassium, Week 14, n=29, 31, 33, 34, 27, 24 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Potassium, EW, n=10, 6, 3, 2, 10, 9 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, PS, n=38, 37, 37, 38, 36, 36: number analyzed (Participants) | 38 | 37 | 37 | 38 | 36 | 36
  Potassium, PS, n=38, 37, 37, 38, 36, 36 | 1 | 1 | 1 | 0 | 2 | 2

25. Secondary Outcome: Number of Participants With Hematology Data of Clinical Importance
Description: Blood samples were collected for the evaluation of hematology parameters including hematocrit, Hgb, lymphocytes, neutrophils and platelets. The number of participants with clinically significant abnormal values of the mentioned hematology parameters was presented. Baseline was defined as the latest assessment (including unscheduled visits) prior to the first dose. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Up to Week 14
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
Participants
  Hematocrit,Baseline, n=38, 38, 38, 38, 37, 38 | 0 | 0 | 0 | 2 | 0 | 0
  Hematocrit, Week 2, n=35, 35, 36, 37, 29, 35: number analyzed (Participants) | 35 | 35 | 36 | 37 | 29 | 35
  Hematocrit, Week 2, n=35, 35, 36, 37, 29, 35 | 1 | 0 | 0 | 2 | 0 | 0
  Hematocrit, Week 4, n=32, 34, 35, 37, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 37 | 29 | 31
  Hematocrit, Week 4, n=32, 34, 35, 37, 29, 31 | 0 | 0 | 1 | 2 | 0 | 0
  Hematocrit, Week 8, n=30, 31, 32, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 38 | 27 | 26
  Hematocrit, Week 8, n=30, 31, 32, 38, 27, 26 | 0 | 0 | 0 | 2 | 0 | 1
  Hematocrit, Week 12, n=27, 30, 31, 36, 26, 25: number analyzed (Participants) | 27 | 30 | 31 | 36 | 26 | 25
  Hematocrit, Week 12, n=27, 30, 31, 36, 26, 25 | 0 | 0 | 0 | 2 | 0 | 0
  Hematocrit, Week 14, n=29, 30, 33, 34, 27, 23: number analyzed (Participants) | 29 | 30 | 33 | 34 | 27 | 23
  Hematocrit, Week 14, n=29, 30, 33, 34, 27, 23 | 1 | 0 | 0 | 1 | 1 | 0
  Hematocrit, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Hematocrit, EW, n=10, 6, 3, 2, 10, 9 | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit, PS, n=38, 37, 37, 38, 36, 36: number analyzed (Participants) | 38 | 37 | 37 | 38 | 36 | 36
  Hematocrit, PS, n=38, 37, 37, 38, 36, 36 | 2 | 0 | 1 | 3 | 1 | 1
  Hgb,Baseline, n=38, 38, 38, 38, 37, 38 | 0 | 0 | 0 | 0 | 0 | 0
  Hgb, Week 2, n=35, 35, 36, 37, 29, 35: number analyzed (Participants) | 35 | 35 | 36 | 37 | 29 | 35
  Hgb, Week 2, n=35, 35, 36, 37, 29, 35 | 0 | 0 | 0 | 1 | 0 | 0
  Hgb, Week 4, n=32, 34, 35, 37, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 37 | 29 | 31
  Hgb, Week 4, n=32, 34, 35, 37, 29, 31 | 0 | 0 | 0 | 1 | 0 | 0
  Hgb, Week 8, n=30, 31, 32, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 38 | 27 | 26
  Hgb, Week 8, n=30, 31, 32, 38, 27, 26 | 0 | 0 | 0 | 2 | 0 | 0
  Hgb, Week 12, n=27, 30, 31, 36, 26, 25: number analyzed (Participants) | 27 | 30 | 31 | 36 | 26 | 25
  Hgb, Week 12, n=27, 30, 31, 36, 26, 25 | 0 | 0 | 0 | 0 | 0 | 0
  Hgb, Week 14, n=29, 30, 33, 34, 27, 23: number analyzed (Participants) | 29 | 30 | 33 | 34 | 27 | 23
  Hgb, Week 14, n=29, 30, 33, 34, 27, 23 | 1 | 0 | 0 | 1 | 0 | 0
  Hgb, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Hgb, EW, n=10, 6, 3, 2, 10, 9 | 0 | 0 | 0 | 0 | 0 | 0
  Hgb, PS, n=38, 37, 37, 38, 36, 36: number analyzed (Participants) | 38 | 37 | 37 | 38 | 36 | 36
  Hgb, PS, n=38, 37, 37, 38, 36, 36 | 1 | 0 | 0 | 2 | 0 | 0
  Lymphocytes, Baseline, n=38, 38, 38, 38, 37, 38 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes, Week 2, n=35, 35, 36, 37, 29, 35: number analyzed (Participants) | 35 | 35 | 36 | 37 | 29 | 35
  Lymphocytes, Week 2, n=35, 35, 36, 37, 29, 35 | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocytes, Week 4, n=31, 34, 35, 37, 29, 31: number analyzed (Participants) | 31 | 34 | 35 | 37 | 29 | 31
  Lymphocytes, Week 4, n=31, 34, 35, 37, 29, 31 | 0 | 1 | 0 | 0 | 0 | 1
  Lymphocytes, Week 8, n=30, 30, 32, 37, 27, 26: number analyzed (Participants) | 30 | 30 | 32 | 37 | 27 | 26
  Lymphocytes, Week 8, n=30, 30, 32, 37, 27, 26 | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocytes, Week 12, n=27, 30, 31, 36, 26, 25: number analyzed (Participants) | 27 | 30 | 31 | 36 | 26 | 25
  Lymphocytes, Week 12, n=27, 30, 31, 36, 26, 25 | 0 | 0 | 0 | 0 | 1 | 0
  Lymphocytes, Week 14, n=29, 30, 33, 34, 27, 23: number analyzed (Participants) | 29 | 30 | 33 | 34 | 27 | 23
  Lymphocytes, Week 14, n=29, 30, 33, 34, 27, 23 | 0 | 1 | 0 | 0 | 0 | 0
  Lymphocytes, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Lymphocytes, EW, n=10, 6, 3, 2, 10, 9 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes, PS, n=38, 37, 37, 38, 36, 36: number analyzed (Participants) | 38 | 37 | 37 | 38 | 36 | 36
  Lymphocytes, PS, n=38, 37, 37, 38, 36, 36 | 0 | 1 | 0 | 0 | 1 | 1
  Neutrophils,Baseline, n=38, 38, 38, 38, 37, 38 | 0 | 0 | 1 | 0 | 0 | 0
  Neutrophils, Week 2, n=35, 35, 36, 37, 29, 35: number analyzed (Participants) | 35 | 35 | 36 | 37 | 29 | 35
  Neutrophils, Week 2, n=35, 35, 36, 37, 29, 35 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils, Week 4, n=31, 34, 35, 37, 29, 31: number analyzed (Participants) | 31 | 34 | 35 | 37 | 29 | 31
  Neutrophils, Week 4, n=31, 34, 35, 37, 29, 31 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils, Week 8, n=30, 30, 32, 37, 27, 26: number analyzed (Participants) | 30 | 30 | 32 | 37 | 27 | 26
  Neutrophils, Week 8, n=30, 30, 32, 37, 27, 26 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils, Week 12, n=27, 30, 31, 36, 26, 25: number analyzed (Participants) | 27 | 30 | 31 | 36 | 26 | 25
  Neutrophils, Week 12, n=27, 30, 31, 36, 26, 25 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils, Week 14, n=29, 30, 33, 34, 27, 23: number analyzed (Participants) | 29 | 30 | 33 | 34 | 27 | 23
  Neutrophils, Week 14, n=29, 30, 33, 34, 27, 23 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils, EW, n=10, 6, 3, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 3 | 2 | 10 | 9
  Neutrophils, EW, n=10, 6, 3, 2, 10, 9 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils, PS, n=38, 37, 37, 38, 36, 36: number analyzed (Participants) | 38 | 37 | 37 | 38 | 36 | 36
  Neutrophils, PS, n=38, 37, 37, 38, 36, 36 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets,Baseline, n=38, 38, 38, 38, 37, 38 | 0 | 1 | 0 | 0 | 0 | 0
  Platelets, Week 2, n=35, 35, 36, 37, 29, 35: number analyzed (Participants) | 35 | 35 | 36 | 37 | 29 | 35
  Platelets, Week 2, n=35, 35, 36, 37, 29, 35 | 0 | 1 | 0 | 0 | 0 | 0
  Platelets, Week 4, n=32, 34, 35, 37, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 37 | 29 | 31
  Platelets, Week 4, n=32, 34, 35, 37, 29, 31 | 0 | 0 | 0 | 0 | 1 | 0
  Platelets, Week 8, n=30, 31, 32, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 32 | 38 | 27 | 26
  Platelets, Week 8, n=30, 31, 32, 38, 27, 26 | 0 | 0 | 0 | 0 | 1 | 0
  Platelets, Week 12, n=27, 30, 31, 36, 26, 25: number analyzed (Participants) | 27 | 30 | 31 | 36 | 26 | 25
  Platelets, Week 12, n=27, 30, 31, 36, 26, 25 | 0 | 0 | 0 | 0 | 1 | 0
  Platelets, Week 14, n=29, 30, 33, 34, 27, 23: number analyzed (Participants) | 29 | 30 | 33 | 34 | 27 | 23
  Platelets, Week 14, n=29, 30, 33, 34, 27, 23 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets, EW, n=10, 5, 3, 2, 9, 9: number analyzed (Participants) | 10 | 5 | 3 | 2 | 9 | 9
  Platelets, EW, n=10, 5, 3, 2, 9, 9 | 0 | 1 | 0 | 0 | 0 | 0
  Platelets, PS, n=38, 37, 37, 38, 35, 36: number analyzed (Participants) | 38 | 37 | 37 | 38 | 35 | 36
  Platelets, PS, n=38, 37, 37, 38, 35, 36 | 0 | 1 | 0 | 0 | 1 | 0

26. Secondary Outcome: Change From Baseline in Immunoglobulin (Ig) A, IgG and IgM Levels
Description: Blood samples were collected for the evaluation of change in IgA, IgG and IgM levels from Baseline throughout the study. Baseline was defined as the latest assessment (including unscheduled visits) prior to the first dose and change from Baseline was defined as the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 12
Population: Safety Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
g/L
  IgA, Week 4, n=32, 34, 35, 38, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 38 | 29 | 31
  IgA, Week 4, n=32, 34, 35, 38, 29, 31 | -0.035 (0.2151) | -0.138 (0.3147) | -0.153 (0.5744) | -0.024 (0.6150) | 0.125 (0.5462) | 0.006 (0.2350)
  IgA, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  IgA, Week 8, n=30, 31, 33, 38, 27, 26 | 0.021 (0.3615) | -0.151 (0.3497) | -0.239 (0.6447) | -0.064 (0.6353) | 0.086 (0.6911) | -0.050 (0.4347)
  IgA, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  IgA, Week 12, n=27, 30, 32, 36, 26, 24 | -0.028 (0.2806) | -0.138 (0.2461) | -0.271 (0.6764) | -0.037 (1.0705) | -0.023 (0.8912) | -0.018 (0.2355)
  IgG, Week 4, n=32, 34, 35, 38, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 38 | 29 | 31
  IgG, Week 4, n=32, 34, 35, 38, 29, 31 | 0.130 (0.8150) | -0.223 (1.0422) | 0.117 (1.4003) | 0.028 (1.7157) | 0.441 (1.6655) | 0.218 (1.1025)
  IgG, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  IgG, Week 8, n=30, 31, 33, 38, 27, 26 | -0.098 (1.1559) | -0.055 (1.1243) | -0.016 (1.4066) | 0.195 (1.4330) | 0.634 (1.4913) | 0.299 (1.3855)
  IgG, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  IgG, Week 12, n=27, 30, 32, 36, 26, 24 | 0.248 (0.8937) | 0.029 (1.1145) | -0.360 (1.3683) | 0.251 (1.4115) | 0.377 (2.0539) | 0.283 (1.0979)
  IgM, Week 4, n=32, 34, 35, 38, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 38 | 29 | 31
  IgM, Week 4, n=32, 34, 35, 38, 29, 31 | -0.077 (0.1215) | -0.050 (0.0797) | -0.023 (0.3524) | -0.017 (0.1434) | -0.004 (0.1951) | -0.016 (0.1371)
  IgM, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  IgM, Week 8, n=30, 31, 33, 38, 27, 26 | -0.103 (0.1649) | -0.030 (0.1737) | -0.005 (0.4892) | -0.012 (0.1213) | -0.011 (0.1951) | -0.006 (0.1802)
  IgM, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  IgM, Week 12, n=27, 30, 32, 36, 26, 24 | -0.072 (0.0992) | -0.082 (0.1264) | -0.047 (0.5307) | -0.017 (0.1495) | -0.023 (0.2431) | -0.033 (0.1900)

27. Secondary Outcome: Number of Participants With Ig Data Outside the Reference Range
Description: Blood samples were collected for the evaluation of change in Ig levels from Baseline throughout the study. Baseline was defined as the latest assessment (including unscheduled visits) prior to the first dose. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Up to Week 12
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
Participants
  IgA, Baseline, n=38, 38, 38, 38, 37, 38 | 2 | 1 | 3 | 4 | 2 | 2
  IgA, Week 4, n=32, 34, 35, 38, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 38 | 29 | 31
  IgA, Week 4, n=32, 34, 35, 38, 29, 31 | 1 | 1 | 1 | 2 | 2 | 1
  IgA, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  IgA, Week 8, n=30, 31, 33, 38, 27, 26 | 1 | 1 | 1 | 2 | 1 | 1
  IgA, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  IgA, Week 12, n=27, 30, 32, 36, 26, 24 | 0 | 1 | 2 | 3 | 0 | 1
  IgA, PS, n=33, 34, 36, 38, 29, 31: number analyzed (Participants) | 33 | 34 | 36 | 38 | 29 | 31
  IgA, PS, n=33, 34, 36, 38, 29, 31 | 2 | 1 | 2 | 3 | 2 | 1
  IgG, Baseline, n=38, 38, 38, 38, 37, 38 | 4 | 2 | 3 | 2 | 1 | 4
  IgG, Week 4, n=32, 34, 35, 38, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 38 | 29 | 31
  IgG, Week 4, n=32, 34, 35, 38, 29, 31 | 3 | 2 | 3 | 3 | 0 | 4
  IgG, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  IgG, Week 8, n=30, 31, 33, 38, 27, 26 | 3 | 2 | 4 | 2 | 1 | 4
  IgG, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  IgG, Week 12, n=27, 30, 32, 36, 26, 24 | 2 | 1 | 4 | 4 | 1 | 2
  IgG, PS, n=33, 34, 36, 38, 29, 31: number analyzed (Participants) | 33 | 34 | 36 | 38 | 29 | 31
  IgG, PS, n=33, 34, 36, 38, 29, 31 | 3 | 2 | 5 | 4 | 1 | 4
  IgM, Baseline, n=38, 38, 38, 38, 37, 38 | 11 | 5 | 9 | 3 | 2 | 5
  IgM, Week 4, n=32, 34, 35, 38, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 38 | 29 | 31
  IgM, Week 4, n=32, 34, 35, 38, 29, 31 | 9 | 5 | 9 | 4 | 2 | 3
  IgM, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  IgM, Week 8, n=30, 31, 33, 38, 27, 26 | 9 | 6 | 8 | 4 | 2 | 4
  IgM, Week 12, n=27, 30, 32, 36, 26, 24: number analyzed (Participants) | 27 | 30 | 32 | 36 | 26 | 24
  IgM, Week 12, n=27, 30, 32, 36, 26, 24 | 8 | 5 | 8 | 3 | 2 | 2
  IgM, PS, n=33, 34, 36, 38, 29, 31: number analyzed (Participants) | 33 | 34 | 36 | 38 | 29 | 31
  IgM, PS, n=33, 34, 36, 38, 29, 31 | 11 | 6 | 10 | 5 | 3 | 4

28. Secondary Outcome: Number of Participants With Immunophenotyping Data Outside the Reference Range
Description: Blood samples were collected for the evaluation of change in levels of cluster of differentiation (CD)19, CD3, CD3 Treg flow cytometry (CD3TFLC), CD3+CD8+, CD3+CD8+ TFLC, CD3+CD4+, CD3+CD4+ TFLC, CD16+CD56+, CD3+CD4+CD25+CD127 flow cytometry (CD3+CD4+CD25+CD127), CD3+CD4+foxP3+CD25+CD127 flow cytometry (CD3+CD4+fP3+CD25+CD127) and T Cell B Cell Natural Killer Lymphocytes flow cytometry (T-B cell NKL). Baseline was defined as the latest assessment (including unscheduled visits) prior to the first dose. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Up to Week 12
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
Participants
  CD19, Baseline, n=38, 38, 38, 38, 37, 38 | 5 | 5 | 5 | 7 | 11 | 1
  CD19, Week 4, n=30, 32, 35, 38, 29, 30: number analyzed (Participants) | 30 | 32 | 35 | 38 | 29 | 30
  CD19, Week 4, n=30, 32, 35, 38, 29, 30 | 2 | 6 | 4 | 6 | 6 | 3
  CD19, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  CD19, Week 8, n=30, 31, 33, 38, 27, 26 | 4 | 5 | 6 | 6 | 5 | 2
  CD19, Week 12, n=27, 29, 32, 36, 26, 24: number analyzed (Participants) | 27 | 29 | 32 | 36 | 26 | 24
  CD19, Week 12, n=27, 29, 32, 36, 26, 24 | 2 | 4 | 4 | 4 | 6 | 1
  CD19, PS, n=33, 34, 36, 38, 29, 31: number analyzed (Participants) | 33 | 34 | 36 | 38 | 29 | 31
  CD19, PS, n=33, 34, 36, 38, 29, 31 | 5 | 7 | 8 | 7 | 9 | 4
  CD3, Baseline, n=38, 38, 38, 38, 37, 38 | 4 | 3 | 5 | 3 | 1 | 2
  CD3, Week 4, n=30, 32, 35, 38, 29, 30: number analyzed (Participants) | 30 | 32 | 35 | 38 | 29 | 30
  CD3, Week 4, n=30, 32, 35, 38, 29, 30 | 1 | 1 | 4 | 0 | 0 | 2
  CD3, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  CD3, Week 8, n=30, 31, 33, 38, 27, 26 | 2 | 1 | 4 | 2 | 1 | 2
  CD3, Week 12, n=27, 29, 32, 36, 26, 24: number analyzed (Participants) | 27 | 29 | 32 | 36 | 26 | 24
  CD3, Week 12, n=27, 29, 32, 36, 26, 24 | 1 | 2 | 3 | 2 | 2 | 0
  CD3, PS, n=33, 34, 36, 38, 29, 31: number analyzed (Participants) | 33 | 34 | 36 | 38 | 29 | 31
  CD3, PS, n=33, 34, 36, 38, 29, 31 | 3 | 4 | 8 | 3 | 2 | 3
  CD3 TFLC, Baseline, n=37,36,38, 38, 36, 38: number analyzed (Participants) | 37 | 36 | 38 | 38 | 36 | 38
  CD3 TFLC, Baseline, n=37,36,38, 38, 36, 38 | 0 | 0 | 0 | 0 | 0 | 0
  CD3 TFLC, Week 4, n=28, 30, 32, 36, 28, 26: number analyzed (Participants) | 28 | 30 | 32 | 36 | 28 | 26
  CD3 TFLC, Week 4, n=28, 30, 32, 36, 28, 26 | 0 | 1 | 0 | 0 | 0 | 0
  CD3 TFLC, Week 8, n=30, 29, 31, 34, 25, 22: number analyzed (Participants) | 30 | 29 | 31 | 34 | 25 | 22
  CD3 TFLC, Week 8, n=30, 29, 31, 34, 25, 22 | 0 | 1 | 0 | 0 | 0 | 0
  CD3 TFLC, Week 12, n=26,26,30, 34, 24, 24: number analyzed (Participants) | 26 | 26 | 30 | 34 | 24 | 24
  CD3 TFLC, Week 12, n=26,26,30, 34, 24, 24 | 0 | 1 | 0 | 0 | 0 | 0
  CD3 TFLC, PS, n=33, 33, 36, 38, 29, 31: number analyzed (Participants) | 33 | 33 | 36 | 38 | 29 | 31
  CD3 TFLC, PS, n=33, 33, 36, 38, 29, 31 | 0 | 1 | 0 | 0 | 0 | 0
  CD3+CD8+, Baseline, n=38, 38, 38, 38, 37, 38 | 0 | 4 | 2 | 3 | 3 | 5
  CD3+CD8+, Week 4, n=30, 32, 35, 38, 29, 30: number analyzed (Participants) | 30 | 32 | 35 | 38 | 29 | 30
  CD3+CD8+, Week 4, n=30, 32, 35, 38, 29, 30 | 0 | 3 | 3 | 2 | 0 | 3
  CD3+CD8+, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  CD3+CD8+, Week 8, n=30, 31, 33, 38, 27, 26 | 0 | 3 | 0 | 1 | 3 | 3
  CD3+CD8+, Week 12, n=27, 29, 32, 36, 26, 24: number analyzed (Participants) | 27 | 29 | 32 | 36 | 26 | 24
  CD3+CD8+, Week 12, n=27, 29, 32, 36, 26, 24 | 0 | 2 | 0 | 1 | 2 | 2
  CD3+CD8+, PS, n=33, 34, 36, 38, 29, 31: number analyzed (Participants) | 33 | 34 | 36 | 38 | 29 | 31
  CD3+CD8+, PS, n=33, 34, 36, 38, 29, 31 | 0 | 4 | 3 | 3 | 3 | 5
  CD3+CD8+ TFLC, Baseline, n=37, 36, 38, 38, 36, 38: number analyzed (Participants) | 37 | 36 | 38 | 38 | 36 | 38
  CD3+CD8+ TFLC, Baseline, n=37, 36, 38, 38, 36, 38 | 0 | 0 | 0 | 0 | 0 | 0
  CD3+CD8+ TFLC, Week 4, n=28, 30, 32, 36, 28, 36: number analyzed (Participants) | 28 | 30 | 32 | 36 | 28 | 36
  CD3+CD8+ TFLC, Week 4, n=28, 30, 32, 36, 28, 36 | 0 | 1 | 0 | 0 | 1 | 0
  CD3+CD8+ TFLC, Week 8, n=30, 29, 31, 34, 25, 22: number analyzed (Participants) | 30 | 29 | 31 | 34 | 25 | 22
  CD3+CD8+ TFLC, Week 8, n=30, 29, 31, 34, 25, 22 | 0 | 1 | 0 | 1 | 1 | 0
  CD3+CD8+ TFLC, Week 12, n=26, 26, 30, 34, 24, 24: number analyzed (Participants) | 26 | 26 | 30 | 34 | 24 | 24
  CD3+CD8+ TFLC, Week 12, n=26, 26, 30, 34, 24, 24 | 0 | 1 | 0 | 0 | 0 | 0
  CD3+CD8+TFLC, PS, n=33, 33,36, 38, 29, 31: number analyzed (Participants) | 33 | 33 | 36 | 38 | 29 | 31
  CD3+CD8+TFLC, PS, n=33, 33,36, 38, 29, 31 | 0 | 1 | 1 | 2 | 2 | 0
  CD3+CD4+, Baseline, n=38, 38, 38, 38, 37, 38 | 6 | 5 | 4 | 2 | 2 | 1
  CD3+CD4+, Week 4, n=30, 32, 35, 38, 29, 30: number analyzed (Participants) | 30 | 32 | 35 | 38 | 29 | 30
  CD3+CD4+, Week 4, n=30, 32, 35, 38, 29, 30 | 3 | 1 | 5 | 3 | 1 | 3
  CD3+CD4+, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  CD3+CD4+, Week 8, n=30, 31, 33, 38, 27, 26 | 3 | 3 | 3 | 2 | 2 | 1
  CD3+CD4+, Week 12, n=27, 29, 32, 36, 26, 24: number analyzed (Participants) | 27 | 29 | 32 | 36 | 26 | 24
  CD3+CD4+, Week 12, n=27, 29, 32, 36, 26, 24 | 1 | 2 | 4 | 2 | 1 | 0
  CD3+CD4+, PS, n=33, 34, 36, 38, 29, 31: number analyzed (Participants) | 33 | 34 | 36 | 38 | 29 | 31
  CD3+CD4+, PS, n=33, 34, 36, 38, 29, 31 | 5 | 6 | 8 | 5 | 5 | 3
  CD3+CD4+ TFLC, Baseline, n=37, 36, 38, 38, 36, 38: number analyzed (Participants) | 37 | 36 | 38 | 38 | 36 | 38
  CD3+CD4+ TFLC, Baseline, n=37, 36, 38, 38, 36, 38 | 0 | 0 | 0 | 0 | 0 | 0
  CD3+CD4+ TFLC, Week 4, n=28, 30, 32, 36, 28, 36: number analyzed (Participants) | 28 | 30 | 32 | 36 | 28 | 36
  CD3+CD4+ TFLC, Week 4, n=28, 30, 32, 36, 28, 36 | 0 | 1 | 0 | 0 | 0 | 0
  CD3+CD4+ TFLC, Week 8, n=30, 29, 31, 34, 25, 22: number analyzed (Participants) | 30 | 29 | 31 | 34 | 25 | 22
  CD3+CD4+ TFLC, Week 8, n=30, 29, 31, 34, 25, 22 | 0 | 1 | 0 | 0 | 0 | 0
  CD3+CD4+ TFLC, Week 12, n=26, 26, 30, 34, 24, 24: number analyzed (Participants) | 26 | 26 | 30 | 34 | 24 | 24
  CD3+CD4+ TFLC, Week 12, n=26, 26, 30, 34, 24, 24 | 0 | 1 | 0 | 0 | 0 | 0
  CD3+CD4+ TF, PS, n=33, 33, 36, 38, 29, 31: number analyzed (Participants) | 33 | 33 | 36 | 38 | 29 | 31
  CD3+CD4+ TF, PS, n=33, 33, 36, 38, 29, 31 | 0 | 1 | 0 | 0 | 0 | 0
  CD16+CD56+, Baseline, n=38, 38, 38, 38, 37, 38 | 0 | 0 | 0 | 1 | 0 | 1
  CD16+CD56+, Week 4, n=30, 32, 35, 38, 29, 30: number analyzed (Participants) | 30 | 32 | 35 | 38 | 29 | 30
  CD16+CD56+, Week 4, n=30, 32, 35, 38, 29, 30 | 1 | 0 | 0 | 0 | 0 | 1
  CD16+CD56+, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  CD16+CD56+, Week 8, n=30, 31, 33, 38, 27, 26 | 0 | 0 | 0 | 0 | 1 | 1
  CD16+CD56+, Week 12, n=27, 29, 32, 36, 26, 24: number analyzed (Participants) | 27 | 29 | 32 | 36 | 26 | 24
  CD16+CD56+, Week 12, n=27, 29, 32, 36, 26, 24 | 1 | 0 | 0 | 0 | 0 | 1
  CD16+CD56+, PS, n=33, 34, 36, 38, 29, 31: number analyzed (Participants) | 33 | 34 | 36 | 38 | 29 | 31
  CD16+CD56+, PS, n=33, 34, 36, 38, 29, 31 | 1 | 0 | 1 | 2 | 1 | 1
  CD3+CD4+CD25+CD127, Baseline, n=37,36,38,38,36,38: number analyzed (Participants) | 37 | 36 | 38 | 38 | 36 | 38
  CD3+CD4+CD25+CD127, Baseline, n=37,36,38,38,36,38 | 0 | 0 | 0 | 0 | 0 | 0
  CD3+CD4+CD25+CD127, Week 4, n=28,30,32,36,28,36: number analyzed (Participants) | 28 | 30 | 32 | 36 | 28 | 36
  CD3+CD4+CD25+CD127, Week 4, n=28,30,32,36,28,36 | 1 | 3 | 1 | 3 | 5 | 0
  CD3+CD4+CD25+CD127, Week 8, n=30,29,31,34,25,22: number analyzed (Participants) | 30 | 29 | 31 | 34 | 25 | 22
  CD3+CD4+CD25+CD127, Week 8, n=30,29,31,34,25,22 | 0 | 4 | 1 | 2 | 5 | 0
  CD3+CD4+CD25+CD127, Week 12, n=26,26,30,34,24,24: number analyzed (Participants) | 26 | 26 | 30 | 34 | 24 | 24
  CD3+CD4+CD25+CD127, Week 12, n=26,26,30,34,24,24 | 0 | 6 | 1 | 7 | 5 | 0
  CD3+CD4+CD25+CD127, PS, n=33,33,36,38,29,31: number analyzed (Participants) | 33 | 33 | 36 | 38 | 29 | 31
  CD3+CD4+CD25+CD127, PS, n=33,33,36,38,29,31 | 1 | 7 | 1 | 9 | 7 | 2
  CD3+CD4+fP3+CD25+CD127Baseline,n=37,36,38,38,36,38: number analyzed (Participants) | 37 | 36 | 38 | 38 | 36 | 38
  CD3+CD4+fP3+CD25+CD127Baseline,n=37,36,38,38,36,38 | 0 | 0 | 0 | 0 | 0 | 0
  CD3+CD4+fP3+CD25+CD127, Week 4,n=28,30,32,36,28,36: number analyzed (Participants) | 28 | 30 | 32 | 36 | 28 | 36
  CD3+CD4+fP3+CD25+CD127, Week 4,n=28,30,32,36,28,36 | 5 | 8 | 4 | 5 | 7 | 3
  CD3+CD4+fP3+CD25+CD127, Week 8,n=30,29,31,34,25,22: number analyzed (Participants) | 30 | 29 | 31 | 34 | 25 | 22
  CD3+CD4+fP3+CD25+CD127, Week 8,n=30,29,31,34,25,22 | 6 | 7 | 6 | 6 | 5 | 4
  CD3+CD4+fP3+CD25+CD127 Week 12,n=26,26,30,34,24,24: number analyzed (Participants) | 26 | 26 | 30 | 34 | 24 | 24
  CD3+CD4+fP3+CD25+CD127 Week 12,n=26,26,30,34,24,24 | 4 | 6 | 3 | 8 | 2 | 2
  CD3+CD4+fP3+CD25+CD127, PS,n=33,33,36,38,29,31: number analyzed (Participants) | 33 | 33 | 36 | 38 | 29 | 31
  CD3+CD4+fP3+CD25+CD127, PS,n=33,33,36,38,29,31 | 11 | 14 | 12 | 15 | 11 | 7
  T-B cell NKL, Baseline, n=38,38,38,38,37,38 | 1 | 1 | 0 | 1 | 1 | 0
  T-B cell NKL, Week 4, n=30,32,35,38,29,30: number analyzed (Participants) | 30 | 32 | 35 | 38 | 29 | 30
  T-B cell NKL, Week 4, n=30,32,35,38,29,30 | 0 | 1 | 1 | 0 | 0 | 1
  T-B cell NKL, Week 8, n=30,31,33,38,27,26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  T-B cell NKL, Week 8, n=30,31,33,38,27,26 | 0 | 0 | 1 | 0 | 0 | 1
  T-B cell NKL, Week 12, n=27,29,32,36,26,24: number analyzed (Participants) | 27 | 29 | 32 | 36 | 26 | 24
  T-B cell NKL, Week 12, n=27,29,32,36,26,24 | 0 | 0 | 0 | 0 | 1 | 0
  T-B cell NKL, PS, n=33,34,36,38,29,31: number analyzed (Participants) | 33 | 34 | 36 | 38 | 29 | 31
  T-B cell NKL, PS, n=33,34,36,38,29,31 | 0 | 1 | 2 | 0 | 1 | 1

29. Secondary Outcome: Change From Baseline in Immunophenotype Data
Description: Blood samples were collected for the evaluation of change from Baseline in immunophenotype levels including CD19, CD3, CD3TFLC, CD3+CD8+, CD3+CD8+ TFLC, CD3+CD4+, CD3+CD4+ TFLC, CD16+CD56+, CD3+CD4+CD25+CD127 flow cytometry (CD3+CD4+CD25+CD127), CD3+CD4+foxP3+CD25+CD127 flow cytometry (CD3+CD4+fP3+CD25+CD127) and T-B cell NKL. Baseline was defined as the latest assessment (including unscheduled visits) prior to the first dose and change from Baseline was defined as the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 12
Population: Safety Population
Measure: Mean (Standard Deviation); unit: GI/L
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
GI/L
  CD19, Week 4, n=30, 32, 35, 38, 29, 30: number analyzed (Participants) | 30 | 32 | 35 | 38 | 29 | 30
  CD19, Week 4, n=30, 32, 35, 38, 29, 30 | -0.0182 (0.1060) | 0.0318 (0.1046) | -0.0261 (0.1177) | -0.0184 (0.2460) | -0.0241 (0.3210) | -0.0109 (0.0659)
  CD19, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  CD19, Week 8, n=30, 31, 33, 38, 27, 26 | 0.0367 (0.1284) | 0.0491 (0.0984) | -0.0288 (0.0953) | -0.0464 (0.2220) | -0.0533 (0.2878) | 0.0150 (0.1099)
  CD19, Week 12, n=27, 29, 32, 36, 26, 24: number analyzed (Participants) | 27 | 29 | 32 | 36 | 26 | 24
  CD19, Week 12, n=27, 29, 32, 36, 26, 24 | 0.0059 (0.1178) | 0.0362 (0.0968) | -0.0334 (0.0968) | -0.0305 (0.2591) | -0.0443 (0.2863) | -0.0097 (0.0774)
  CD3, Week 4, n=30, 32, 35, 38, 29, 30: number analyzed (Participants) | 30 | 32 | 35 | 38 | 29 | 30
  CD3, Week 4, n=30, 32, 35, 38, 29, 30 | -0.1067 (0.3964) | 0.1044 (0.3945) | -0.0360 (0.3419) | 0.0186 (0.3417) | -0.0842 (0.2888) | -0.0584 (0.3175)
  CD3, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  CD3, Week 8, n=30, 31, 33, 38, 27, 26 | 0.0227 (0.4318) | 0.1426 (0.3650) | -0.0101 (0.3231) | -0.0053 (0.3463) | -0.1063 (0.4996) | -0.0213 (0.2936)
  CD3, Week 12, n=27, 29, 32, 36, 26, 24: number analyzed (Participants) | 27 | 29 | 32 | 36 | 26 | 24
  CD3, Week 12, n=27, 29, 32, 36, 26, 24 | -0.0511 (0.4225) | 0.1327 (0.4230) | -0.0248 (0.3140) | -0.0315 (0.3259) | -0.0822 (0.3222) | -0.0142 (0.3345)
  CD3 TFLC, Week 4, n=27, 29, 32, 36, 28, 26: number analyzed (Participants) | 27 | 29 | 32 | 36 | 28 | 26
  CD3 TFLC, Week 4, n=27, 29, 32, 36, 28, 26 | -0.0829 (0.4002) | 0.1270 (0.4233) | 0.0196 (0.3104) | 0.0320 (0.3412) | -0.0937 (0.3115) | -0.1031 (0.3504)
  CD3 TFLC, Week 8, n=29, 27, 31, 34, 25, 22: number analyzed (Participants) | 29 | 27 | 31 | 34 | 25 | 22
  CD3 TFLC, Week 8, n=29, 27, 31, 34, 25, 22 | 0.0187 (0.4749) | 0.1296 (0.3352) | -0.0158 (0.3503) | 0.0053 (0.2782) | -0.1393 (0.5368) | -0.0383 (0.3471)
  CD3 TFLC, Week 12, n=25,24,30, 34, 24, 24: number analyzed (Participants) | 25 | 24 | 30 | 34 | 24 | 24
  CD3 TFLC, Week 12, n=25,24,30, 34, 24, 24 | -0.0916 (0.4466) | 0.1494 (0.4745) | -0.0266 (0.3227) | -0.0342 (0.3157) | -0.1220 (0.3010) | -0.0280 (0.3630)
  CD3+CD8+, Week 4, n=30, 32, 35, 38, 29, 30: number analyzed (Participants) | 30 | 32 | 35 | 38 | 29 | 30
  CD3+CD8+, Week 4, n=30, 32, 35, 38, 29, 30 | -0.0297 (0.1394) | 0.0524 (0.1516) | 0.0094 (0.1279) | 0.0095 (0.1217) | -0.0009 (0.1871) | 0.0179 (0.1504)
  CD3+CD8+, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  CD3+CD8+, Week 8, n=30, 31, 33, 38, 27, 26 | 0.0001 (0.1582) | 0.0683 (0.1697) | 0.0100 (0.1006) | 0.0219 (0.1550) | -0.0189 (0.2073) | 0.0566 (0.1508)
  CD3+CD8+, Week 12, n=27, 29, 32, 36, 26, 24: number analyzed (Participants) | 27 | 29 | 32 | 36 | 26 | 24
  CD3+CD8+, Week 12, n=27, 29, 32, 36, 26, 24 | -0.0174 (0.1417) | 0.0477 (0.1642) | 0.0106 (0.1253) | 0.0151 (0.1594) | 0.0081 (0.1920) | 0.0326 (0.1690)
  CD3+CD8+ TFLC, Week 4, n=27, 29, 32, 36, 28, 26: number analyzed (Participants) | 27 | 29 | 32 | 36 | 28 | 26
  CD3+CD8+ TFLC, Week 4, n=27, 29, 32, 36, 28, 26 | -0.0203 (0.1264) | 0.0359 (0.1719) | 0.0083 (0.0980) | -0.0069 (0.1480) | -0.0107 (0.1759) | -0.0180 (0.1055)
  CD3+CD8+ TFLC, Week 8, n=29, 27, 31, 34, 25, 22: number analyzed (Participants) | 29 | 27 | 31 | 34 | 25 | 22
  CD3+CD8+ TFLC, Week 8, n=29, 27, 31, 34, 25, 22 | -0.0066 (0.1420) | 0.0375 (0.1628) | 0.0091 (0.0920) | 0.0035 (0.1194) | -0.0254 (0.2065) | 0.0139 (0.1195)
  CD3+CD8+ TFLC, Week 12, n=25, 24, 30, 34, 24, 24: number analyzed (Participants) | 25 | 24 | 30 | 34 | 24 | 24
  CD3+CD8+ TFLC, Week 12, n=25, 24, 30, 34, 24, 24 | -0.0306 (0.1284) | 0.0260 (0.1760) | -0.0042 (0.1113) | 0.0010 (0.1518) | -0.0112 (0.1493) | 0.0193 (0.1535)
  CD3+CD4+, Week 4, n=30, 32, 35, 38, 29, 30: number analyzed (Participants) | 30 | 32 | 35 | 38 | 29 | 30
  CD3+CD4+, Week 4, n=30, 32, 35, 38, 29, 30 | -0.0750 (0.2756) | 0.0525 (0.2577) | -0.0374 (0.2429) | 0.0210 (0.2475) | -0.0857 (0.1802) | -0.0775 (0.2286)
  CD3+CD4+, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  CD3+CD4+, Week 8, n=30, 31, 33, 38, 27, 26 | 0.0296 (0.3006) | 0.0758 (0.2036) | -0.0042 (0.2396) | -0.0164 (0.2338) | -0.0821 (0.3158) | -0.0715 (0.2205)
  CD3+CD4+, Week 12, n=27, 29, 32, 36, 26, 24: number analyzed (Participants) | 27 | 29 | 32 | 36 | 26 | 24
  CD3+CD4+, Week 12, n=27, 29, 32, 36, 26, 24 | -0.0228 (0.2928) | 0.0936 (0.2664) | -0.0225 (0.2149) | -0.0249 (0.2005) | -0.0798 (0.1817) | -0.0458 (0.1960)
  CD3+CD4+ TFLC, Week 4, n=27, 29, 32, 36, 28, 26: number analyzed (Participants) | 27 | 29 | 32 | 36 | 28 | 26
  CD3+CD4+ TFLC, Week 4, n=27, 29, 32, 36, 28, 26 | -0.0512 (0.2493) | 0.0764 (0.2613) | 0.0009 (0.2121) | 0.0280 (0.2521) | -0.0729 (0.1786) | -0.0621 (0.2216)
  CD3+CD4+ TFLC, Week 8, n=29, 27, 31, 34, 25, 22: number analyzed (Participants) | 29 | 27 | 31 | 34 | 25 | 22
  CD3+CD4+ TFLC, Week 8, n=29, 27, 31, 34, 25, 22 | 0.0268 (0.3134) | 0.0857 (0.1814) | -0.0075 (0.2525) | 0.0138 (0.2066) | -0.0784 (0.3136) | -0.0298 (0.2089)
  CD3+CD4+ TFLC, Week 12, n=25, 24, 30, 34, 24, 24: number analyzed (Participants) | 25 | 24 | 30 | 34 | 24 | 24
  CD3+CD4+ TFLC, Week 12, n=25, 24, 30, 34, 24, 24 | -0.0511 (0.2835) | 0.1196 (0.2891) | -0.0159 (0.2244) | 0.0044 (0.1730) | -0.0679 (0.1740) | -0.0386 (0.1832)
  CD16+CD56+, Week 4, n=30, 32, 35, 38, 29, 30: number analyzed (Participants) | 30 | 32 | 35 | 38 | 29 | 30
  CD16+CD56+, Week 4, n=30, 32, 35, 38, 29, 30 | -0.023 (0.0910) | 0.014 (0.1031) | 0.011 (0.0897) | -0.009 (0.0821) | -0.013 (0.1134) | 0.001 (0.0876)
  CD16+CD56+, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  CD16+CD56+, Week 8, n=30, 31, 33, 38, 27, 26 | 0.002 (0.0699) | 0.011 (0.1312) | 0.009 (0.0867) | -0.002 (0.0713) | -0.000 (0.1800) | 0.013 (0.1339)
  CD16+CD56+, Week 12, n=27, 29, 32, 36, 26, 24: number analyzed (Participants) | 27 | 29 | 32 | 36 | 26 | 24
  CD16+CD56+, Week 12, n=27, 29, 32, 36, 26, 24 | -0.010 (0.0861) | -0.001 (0.1283) | -0.015 (0.0861) | -0.022 (0.1082) | -0.035 (0.1168) | 0.024 (0.0792)
  CD3+CD4+CD25+CD127, Week 4, n=27,29,32,36,28,26: number analyzed (Participants) | 27 | 29 | 32 | 36 | 28 | 26
  CD3+CD4+CD25+CD127, Week 4, n=27,29,32,36,28,26 | 0.0016 (0.0109) | 0.0021 (0.0195) | 0.0019 (0.0147) | -0.0036 (0.0218) | -0.0016 (0.0172) | -0.0008 (0.0097)
  CD3+CD4+CD25+CD127, Week 8, n=29,27,31,34,25,22: number analyzed (Participants) | 29 | 27 | 31 | 34 | 25 | 22
  CD3+CD4+CD25+CD127, Week 8, n=29,27,31,34,25,22 | 0.0002 (0.0141) | 0.0040 (0.0228) | 0.0027 (0.0133) | -0.0019 (0.0200) | -0.0034 (0.0205) | 0.0020 (0.0122)
  CD3+CD4+CD25+CD127, Week 12, n=25,24,30,34,24,24: number analyzed (Participants) | 25 | 24 | 30 | 34 | 24 | 24
  CD3+CD4+CD25+CD127, Week 12, n=25,24,30,34,24,24 | 0.0060 (0.0121) | 0.0035 (0.0279) | 0.0029 (0.0164) | -0.0035 (0.0229) | -0.0037 (0.0141) | -0.0010 (0.0106)
  CD3+CD4+fP3+CD25+CD127, Week4,n=27,29,32,36,28,26: number analyzed (Participants) | 27 | 29 | 32 | 36 | 28 | 26
  CD3+CD4+fP3+CD25+CD127, Week4,n=27,29,32,36,28,26 | -0.0019 (0.0118) | 0.0057 (0.0110) | 0.0018 (0.0107) | -0.0024 (0.0130) | -0.0005 (0.0115) | -0.0003 (0.0104)
  CD3+CD4+fP3+CD25+CD127, Week 8,n=29,27,31,34,25,22: number analyzed (Participants) | 29 | 27 | 31 | 34 | 25 | 22
  CD3+CD4+fP3+CD25+CD127, Week 8,n=29,27,31,34,25,22 | -0.0006 (0.0170) | 0.0055 (0.0121) | 0.0004 (0.0118) | 0.0055 (0.0134) | 0.0003 (0.0107) | -0.0000 (0.0100)
  CD3+CD4+fP3+CD25+CD127 Week12,n=25,24,30,34,24,24: number analyzed (Participants) | 25 | 24 | 30 | 34 | 24 | 24
  CD3+CD4+fP3+CD25+CD127 Week12,n=25,24,30,34,24,24 | 0.0063 (0.0115) | 0.0041 (0.0147) | 0.0005 (0.0127) | -0.0001 (0.0125) | 0.0001 (0.0099) | 0.0001 (0.0124)
  T-B cell NKL, Week 4, n=30,32,35,38,29,30: number analyzed (Participants) | 30 | 32 | 35 | 38 | 29 | 30
  T-B cell NKL, Week 4, n=30,32,35,38,29,30 | -0.157 (0.5537) | 0.152 (0.5655) | -0.051 (0.4505) | -0.009 (0.4837) | -0.137 (0.4446) | -0.083 (0.4134)
  T-B cell NKL, Week 8, n=30,31,33,38,27,26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  T-B cell NKL, Week 8, n=30,31,33,38,27,26 | 0.057 (0.5699) | 0.195 (0.5345) | -0.028 (0.4384) | -0.064 (0.4563) | -0.186 (0.4999) | 0.006 (0.4809)
  T-B cell NKL, Week 12, n=27,29,32,36,26,24: number analyzed (Participants) | 27 | 29 | 32 | 36 | 26 | 24
  T-B cell NKL, Week 12, n=27,29,32,36,26,24 | -0.063 (0.5793) | 0.163 (0.6093) | -0.081 (0.4282) | -0.094 (0.5229) | -0.193 (0.4038) | 0.008 (0.4342)

30. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in semi-supine position after at least 5 minutes of rest. Baseline was defined as the latest assessment prior to the first dose and change from Baseline was defined as the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
Millimeter of mercury (mmHg)
  SBP, Week 1, n=36, 38, 37, 38, 35, 37: number analyzed (Participants) | 36 | 38 | 37 | 38 | 35 | 37
  SBP, Week 1, n=36, 38, 37, 38, 35, 37 | -1.4 (10.54) | -0.8 (10.54) | 1.6 (10.08) | 2.1 (6.97) | 1.4 (11.18) | 1.1 (11.16)
  SBP, Week 2, n=36, 36, 36, 38, 31, 35: number analyzed (Participants) | 36 | 36 | 36 | 38 | 31 | 35
  SBP, Week 2, n=36, 36, 36, 38, 31, 35 | -2.0 (11.61) | -1.0 (11.45) | 3.0 (10.73) | -0.1 (9.79) | 0.6 (13.73) | -1.1 (13.15)
  SBP, Week 4, n=32, 34, 35, 38, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 38 | 29 | 31
  SBP, Week 4, n=32, 34, 35, 38, 29, 31 | 0.4 (12.40) | -2.0 (12.68) | 2.6 (11.54) | -1.4 (8.35) | -0.3 (13.35) | -0.3 (13.22)
  SBP, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  SBP, Week 8, n=30, 31, 33, 38, 27, 26 | 4.0 (12.11) | -1.6 (14.25) | 4.0 (14.69) | 0.3 (13.42) | 0.4 (13.34) | 2.4 (13.81)
  SBP, Week 12, n=26, 30, 32, 36, 26, 25: number analyzed (Participants) | 26 | 30 | 32 | 36 | 26 | 25
  SBP, Week 12, n=26, 30, 32, 36, 26, 25 | 3.4 (14.09) | -1.5 (14.88) | 1.1 (12.97) | -0.6 (9.51) | 2.0 (11.16) | 1.2 (12.02)
  SBP, Week 14, n=29, 31, 33, 34, 27, 26: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 26
  SBP, Week 14, n=29, 31, 33, 34, 27, 26 | -0.3 (13.10) | -0.9 (14.44) | 2.6 (11.66) | -1.1 (9.70) | -2.4 (15.05) | 2.2 (10.97)
  SBP, EW, n=10, 7, 4, 2, 10, 9: number analyzed (Participants) | 10 | 7 | 4 | 2 | 10 | 9
  SBP, EW, n=10, 7, 4, 2, 10, 9 | 5.3 (14.73) | 0.4 (17.22) | 1.3 (8.73) | -10.5 (2.12) | -1.3 (16.15) | -4.0 (13.19)
  DBP, Week 1, n=36, 38, 37, 38, 35, 37: number analyzed (Participants) | 36 | 38 | 37 | 38 | 35 | 37
  DBP, Week 1, n=36, 38, 37, 38, 35, 37 | 0.9 (7.70) | -0.2 (7.64) | 0.4 (6.61) | 1.5 (7.48) | 1.5 (10.14) | -0.8 (8.27)
  DBP, Week 2, n=36, 36, 36, 38, 31, 35: number analyzed (Participants) | 36 | 36 | 36 | 38 | 31 | 35
  DBP, Week 2, n=36, 36, 36, 38, 31, 35 | 0.5 (8.13) | 0.3 (7.55) | 2.3 (6.52) | 0.3 (7.11) | 1.2 (9.51) | 0.0 (7.94)
  DBP, Week 4, n=32, 34, 35, 38, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 38 | 29 | 31
  DBP, Week 4, n=32, 34, 35, 38, 29, 31 | 1.0 (8.04) | 0.7 (7.53) | 1.2 (6.79) | -0.2 (5.77) | -1.8 (9.32) | -0.2 (7.54)
  DBP, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  DBP, Week 8, n=30, 31, 33, 38, 27, 26 | 0.1 (6.44) | 1.4 (9.17) | 2.1 (7.26) | 0.9 (9.66) | 0.6 (8.42) | 0.6 (8.18)
  DBP, Week 12, n=26, 30, 32, 36, 26, 25: number analyzed (Participants) | 26 | 30 | 32 | 36 | 26 | 25
  DBP, Week 12, n=26, 30, 32, 36, 26, 25 | 2.4 (9.98) | 1.3 (9.00) | 1.0 (8.28) | 0.3 (8.02) | 0.1 (8.60) | -0.1 (7.98)
  DBP, Week 14, n=29, 31, 33, 34, 27, 26: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 26
  DBP, Week 14, n=29, 31, 33, 34, 27, 26 | 0.3 (8.80) | 2.5 (8.27) | 2.2 (5.56) | -0.1 (7.64) | -1.1 (9.45) | 0.2 (9.85)
  DBP, EW, n=10, 7, 4, 2, 10, 9: number analyzed (Participants) | 10 | 7 | 4 | 2 | 10 | 9
  DBP, EW, n=10, 7, 4, 2, 10, 9 | 3.4 (6.22) | 1.4 (7.32) | 3.5 (5.97) | 3.5 (16.26) | 1.2 (11.49) | -1.1 (6.13)

31. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in semi-supine position after at least 5 minutes of rest. Baseline was defined as the latest assessment prior to the first dose and change from Baseline was defined as the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
beats per minute
  Week 1, n=36, 38, 37, 38, 35, 37: number analyzed (Participants) | 36 | 38 | 37 | 38 | 35 | 37
  Week 1, n=36, 38, 37, 38, 35, 37 | 0.5 (8.82) | -0.4 (9.40) | 1.7 (7.07) | -0.1 (9.18) | -0.0 (7.65) | -0.6 (9.96)
  Week 2, n=36, 36, 36, 38, 31, 35: number analyzed (Participants) | 36 | 36 | 36 | 38 | 31 | 35
  Week 2, n=36, 36, 36, 38, 31, 35 | 0.9 (10.33) | -3.2 (9.77) | 1.4 (7.73) | 1.7 (9.76) | -1.5 (11.51) | 1.6 (10.40)
  Week 4, n=32, 34, 35, 38, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 38 | 29 | 31
  Week 4, n=32, 34, 35, 38, 29, 31 | 1.2 (8.08) | -0.9 (8.08) | 0.8 (7.13) | 1.5 (9.78) | 2.4 (11.14) | -1.7 (7.59)
  Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  Week 8, n=30, 31, 33, 38, 27, 26 | -0.4 (8.06) | -0.9 (7.59) | 0.2 (8.02) | 1.3 (9.38) | 2.8 (10.54) | 0.2 (10.28)
  Week 12, n=26, 30, 32, 36, 26, 25: number analyzed (Participants) | 26 | 30 | 32 | 36 | 26 | 25
  Week 12, n=26, 30, 32, 36, 26, 25 | 0.1 (9.16) | -2.2 (10.18) | 1.4 (8.18) | 0.6 (9.80) | 1.2 (11.75) | 2.6 (8.04)
  Week 14, n=29, 31, 33, 34, 27, 26: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 26
  Week 14, n=29, 31, 33, 34, 27, 26 | -0.6 (8.52) | -0.8 (8.27) | 0.2 (9.20) | -0.1 (8.48) | -0.1 (11.14) | 1.3 (6.24)
  EW, n=10, 7, 4, 2, 10, 9: number analyzed (Participants) | 10 | 7 | 4 | 2 | 10 | 9
  EW, n=10, 7, 4, 2, 10, 9 | -2.2 (4.54) | -2.7 (9.25) | -2.5 (5.80) | -4.5 (3.54) | 2.4 (11.99) | -2.1 (7.36)

32. Secondary Outcome: Change From Baseline in Temperature
Description: Temperature was measured in semi-supine position after at least 5 minutes of rest. Baseline was defined as the latest assessment prior to the first dose and change from Baseline was defined as the value at post dose visit minus the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to Week 14
Population: Safety Population
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
degree Celsius
  Week 1, n=36, 38, 37, 38, 35, 37: number analyzed (Participants) | 36 | 38 | 37 | 38 | 35 | 37
  Week 1, n=36, 38, 37, 38, 35, 37 | 0.01 (0.356) | -0.00 (0.336) | -0.03 (0.271) | 0.07 (0.401) | -0.03 (0.548) | -0.03 (0.468)
  Week 2, n=36, 36, 36, 38, 31, 35: number analyzed (Participants) | 36 | 36 | 36 | 38 | 31 | 35
  Week 2, n=36, 36, 36, 38, 31, 35 | 0.03 (0.395) | -0.01 (0.410) | -0.01 (0.314) | 0.19 (0.442) | -0.17 (0.473) | 0.03 (0.384)
  Week 4, n=31, 34, 35, 38, 29, 31: number analyzed (Participants) | 31 | 34 | 35 | 38 | 29 | 31
  Week 4, n=31, 34, 35, 38, 29, 31 | 0.05 (0.445) | 0.11 (0.385) | 0.06 (0.333) | 0.07 (0.318) | -0.04 (0.405) | 0.03 (0.439)
  Week 8, n=29, 31, 32, 38, 27, 26: number analyzed (Participants) | 29 | 31 | 32 | 38 | 27 | 26
  Week 8, n=29, 31, 32, 38, 27, 26 | -0.02 (0.503) | 0.17 (0.334) | 0.12 (0.345) | 0.17 (0.453) | 0.14 (0.473) | 0.11 (0.473)
  Week 12, n=26, 30, 32, 36, 26, 25: number analyzed (Participants) | 26 | 30 | 32 | 36 | 26 | 25
  Week 12, n=26, 30, 32, 36, 26, 25 | 0.02 (0.343) | 0.14 (0.423) | 0.12 (0.429) | 0.18 (0.520) | 0.02 (0.492) | 0.12 (0.561)
  Week 14, n=29, 31, 33, 34, 27, 26: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 26
  Week 14, n=29, 31, 33, 34, 27, 26 | -0.04 (0.372) | 0.10 (0.364) | 0.01 (0.456) | 0.11 (0.406) | -0.03 (0.522) | 0.00 (0.591)
  EW, n=10, 7, 4, 2, 10, 9: number analyzed (Participants) | 10 | 7 | 4 | 2 | 10 | 9
  EW, n=10, 7, 4, 2, 10, 9 | 0.12 (0.466) | -0.09 (0.339) | 0.22 (0.330) | 0.25 (0.778) | 0.30 (0.533) | -0.27 (0.255)

33. Secondary Outcome: Number of Participants With Vital Signs of Clinical Importance
Description: The vital signs including SBP, DBP and pulse rate were measured from Baseline throughout the study. The number of participants with clinically significant abnormal vital signs were presented. Baseline was defined as the latest assessment prior to the first dose. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Up to Week 14
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
Participants
  SBP, Baseline, n=38, 38, 38, 38, 37, 38 | 0 | 2 | 0 | 1 | 1 | 0
  SBP, Week 1, n=36, 38, 37, 38, 35, 37: number analyzed (Participants) | 36 | 38 | 37 | 38 | 35 | 37
  SBP, Week 1, n=36, 38, 37, 38, 35, 37 | 0 | 1 | 0 | 1 | 0 | 0
  SBP, Week 2, n=36, 36, 36, 38, 31, 35: number analyzed (Participants) | 36 | 36 | 36 | 38 | 31 | 35
  SBP, Week 2, n=36, 36, 36, 38, 31, 35 | 0 | 1 | 0 | 0 | 0 | 1
  SBP, Week 4, n=32, 34, 35, 38, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 38 | 29 | 31
  SBP, Week 4, n=32, 34, 35, 38, 29, 31 | 0 | 1 | 0 | 1 | 1 | 0
  SBP, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  SBP, Week 8, n=30, 31, 33, 38, 27, 26 | 0 | 0 | 0 | 2 | 0 | 0
  SBP, Week 12, n=26, 30, 32, 36, 26, 25: number analyzed (Participants) | 26 | 30 | 32 | 36 | 26 | 25
  SBP, Week 12, n=26, 30, 32, 36, 26, 25 | 1 | 0 | 0 | 1 | 0 | 0
  SBP, Week 14, n=29, 31, 33, 34, 27, 26: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 26
  SBP, Week 14, n=29, 31, 33, 34, 27, 26 | 0 | 0 | 0 | 0 | 0 | 0
  SBP, EW, n=10, 7, 4, 2, 10, 9: number analyzed (Participants) | 10 | 7 | 4 | 2 | 10 | 9
  SBP, EW, n=10, 7, 4, 2, 10, 9 | 1 | 1 | 0 | 0 | 0 | 0
  SBP, PS, n=n=38, 38, 38, 38, 37, 38 | 2 | 3 | 0 | 2 | 1 | 1
  DBP, Baseline, n=38, 38, 38, 38, 37, 38 | 0 | 0 | 0 | 1 | 0 | 0
  DBP, Week 1, n=36, 38, 37, 38, 35, 37: number analyzed (Participants) | 36 | 38 | 37 | 38 | 35 | 37
  DBP, Week 1, n=36, 38, 37, 38, 35, 37 | 0 | 0 | 0 | 1 | 0 | 1
  DBP, Week 2, n=36, 36, 36, 38, 31, 35: number analyzed (Participants) | 36 | 36 | 36 | 38 | 31 | 35
  DBP, Week 2, n=36, 36, 36, 38, 31, 35 | 2 | 1 | 1 | 0 | 0 | 1
  DBP, Week 4, n=32, 34, 35, 38, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 38 | 29 | 31
  DBP, Week 4, n=32, 34, 35, 38, 29, 31 | 0 | 0 | 1 | 0 | 0 | 1
  DBP, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  DBP, Week 8, n=30, 31, 33, 38, 27, 26 | 0 | 1 | 1 | 0 | 0 | 1
  DBP, Week 12, n=26, 30, 32, 36, 26, 25: number analyzed (Participants) | 26 | 30 | 32 | 36 | 26 | 25
  DBP, Week 12, n=26, 30, 32, 36, 26, 25 | 1 | 0 | 1 | 2 | 0 | 1
  DBP, Week 14, n=29, 31, 33, 34, 27, 26: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 26
  DBP, Week 14, n=29, 31, 33, 34, 27, 26 | 0 | 0 | 0 | 0 | 0 | 0
  DBP, EW, n=10, 7, 4, 2, 10, 9: number analyzed (Participants) | 10 | 7 | 4 | 2 | 10 | 9
  DBP, EW, n=10, 7, 4, 2, 10, 9 | 0 | 1 | 0 | 0 | 0 | 0
  DBP, PS, n=38, 38, 38, 38, 37, 38 | 2 | 2 | 1 | 3 | 0 | 1
  Pulse rate, Baseline, n=38, 38, 38, 38, 37, 38 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate, Week 1, n=36, 38, 37, 38, 35, 37: number analyzed (Participants) | 36 | 38 | 37 | 38 | 35 | 37
  Pulse rate, Week 1, n=36, 38, 37, 38, 35, 37 | 0 | 0 | 0 | 0 | 1 | 0
  Pulse rate, Week 2, n=36, 36, 36, 38, 31, 35: number analyzed (Participants) | 36 | 36 | 36 | 38 | 31 | 35
  Pulse rate, Week 2, n=36, 36, 36, 38, 31, 35 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate, Week 4, n=32, 34, 35, 38, 29, 31: number analyzed (Participants) | 32 | 34 | 35 | 38 | 29 | 31
  Pulse rate, Week 4, n=32, 34, 35, 38, 29, 31 | 0 | 0 | 0 | 0 | 1 | 0
  Pulse rate, Week 8, n=30, 31, 33, 38, 27, 26: number analyzed (Participants) | 30 | 31 | 33 | 38 | 27 | 26
  Pulse rate, Week 8, n=30, 31, 33, 38, 27, 26 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate, Week 12, n=26, 30, 32, 36, 26, 25: number analyzed (Participants) | 26 | 30 | 32 | 36 | 26 | 25
  Pulse rate, Week 12, n=26, 30, 32, 36, 26, 25 | 0 | 0 | 0 | 0 | 1 | 0
  Pulse rate, Week 14, n=29, 31, 33, 34, 27, 26: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 26
  Pulse rate, Week 14, n=29, 31, 33, 34, 27, 26 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate, EW, n=10, 7, 4, 2, 10, 9: number analyzed (Participants) | 10 | 7 | 4 | 2 | 10 | 9
  Pulse rate, EW, n=10, 7, 4, 2, 10, 9 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate, PS, n=38, 38, 38, 38, 37, 38 | 0 | 1 | 1 | 0 | 1 | 0

34. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Single 12-lead ECGs were obtained over a brief recording period at each specified time point during the study using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, and corrected QT (QTc) intervals. Baseline was defined as the latest assessment (including unscheduled visits) prior to the first dose. For multiple ECGs at one visit, or "Any time post-screen", a participant is categorized as "Abnormal" if >=1 assessment is abnormal. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Up to Week 14
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
Number analyzed (Participants) | 38 | 38 | 38 | 38 | 37 | 38
Participants
  Baseline, n=38, 38, 38, 38, 37, 38 | 5 | 8 | 6 | 4 | 6 | 5
  Week 1, n=36, 38, 37, 37, 34, 37: number analyzed (Participants) | 36 | 38 | 37 | 37 | 34 | 37
  Week 1, n=36, 38, 37, 37, 34, 37 | 4 | 8 | 7 | 4 | 5 | 4
  Week 12, n=26, 30, 32, 36, 26, 25: number analyzed (Participants) | 26 | 30 | 32 | 36 | 26 | 25
  Week 12, n=26, 30, 32, 36, 26, 25 | 2 | 6 | 7 | 4 | 4 | 4
  Week 14, n=29, 31, 33, 34, 27, 25: number analyzed (Participants) | 29 | 31 | 33 | 34 | 27 | 25
  Week 14, n=29, 31, 33, 34, 27, 25 | 2 | 5 | 10 | 5 | 2 | 3
  EW, n=10, 6, 4, 2, 10, 9: number analyzed (Participants) | 10 | 6 | 4 | 2 | 10 | 9
  EW, n=10, 6, 4, 2, 10, 9 | 1 | 3 | 0 | 0 | 0 | 1
  PS, n=38, 38, 38, 38, 36, 37: number analyzed (Participants) | 38 | 38 | 38 | 38 | 36 | 37
  PS, n=38, 38, 38, 38, 36, 37 | 7 | 11 | 10 | 7 | 7 | 7

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study treatment until the Follow up Visit 2 at Week 16.
Description: Safety Population which comprised of all participants who received at least one dose of study treatment
Arm/Group | GSK2894512 1% BID | GSK2894512 1% QD | GSK2894512 0.5% BID | GSK2894512 0.5% QD | Vehicle BID | Vehicle QD
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38 | 0/38 | 0/38 | 0/37 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/38 | 3/38 | 3/38 | 0/38 | 0/37 | 0/38
Other Adverse Events (participants affected / at risk) | 17/38 | 12/38 | 11/38 | 11/38 | 3/37 | 3/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2894512 1% BID (N=38) | GSK2894512 1% QD (N=38) | GSK2894512 0.5% BID (N=38) | GSK2894512 0.5% QD (N=38) | Vehicle BID (N=37) | Vehicle QD (N=38)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enlarged uvula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2894512 1% BID (N=38) | GSK2894512 1% QD (N=38) | GSK2894512 0.5% BID (N=38) | GSK2894512 0.5% QD (N=38) | Vehicle BID (N=37) | Vehicle QD (N=38)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Application site dermatitis (General disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 8 (8) | 2 (2) | 4 (4) | 5 (5) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.